Thomas J. Stephens & Associates, Inc. Stephens Study Number: C16-CD020 Galderma Laboratories, L.P. Study Number: GLI.04.SPR.US10354 Final Report 02 Jan 2018

# VIII. Sample Forms

Informed Consent Form Case Report Forms Questionnaires Daily Diary

## INFORMED CONSENT DOCUMENT AGREEMENT TO BE IN A RESEARCH STUDY

NAME OF TESTING COMPANY: Thomas J. Stephens & Associates, Inc.

NUMBER AND TITLE OF STUDY: C16-CD020 (GLI.04.SPR.US10354); "A Multi-

Center Clinical Trial to Evaluate the Efficacy of

Two Acne Treatments"

NAME OF PERSON IN CHARGE OF

THE RESEARCH STUDY

(STUDY DOCTOR/INVESTIGATOR): Lily Jiang, Ph.D.

**TELEPHONE NUMBER(S), DAYTIME:** 972-392-1529 **AFTER HOURS:** 469-766-4781

## INTRODUCTION

You are being invited to volunteer for a clinical research study. You must read and sign this form before you agree to take part in this study. This form will give you more information about this study. Please ask as many questions as you need to before you decide if you want to be in the study. You should not sign this form if you have any questions that have not been answered.

Thomas J. Stephens & Associates, Inc., a contract research organization, is being paid by the sponsor (the company paying for this study) to conduct this research study.

You must be honest with the Investigator about your health history or it may not be safe for you to be in this study.

### PURPOSE OF THE STUDY

The purpose of this study is to evaluate the efficiency of 2 acne treatments for 24 weeks of use in adult men and women with mild to moderate facial acne, at least 5 inflammatory lesions, and at least 10 - 100 non-inflammatory lesions.

## HOW LONG THE STUDY WILL LAST AND HOW MANY PEOPLE WILL BE IN THE STUDY

This study will last 24 weeks and have up to 8 visits. At least 100 subjects, men and women between the ages of 21-45, are expected to complete this study, with at least 50 subjects completed per cell. Each site is to enroll no more than 40 subjects, with at least 100 subjects expected to complete when combined.

## TO BE IN THIS STUDY

### You must:

- Be a man or woman age 21 to 45 years at the time of enrollment.
- Have mild to moderate acne on the face as determined by the Investigator or designee.
- Have at least 5 inflammatory lesions as determined by the Investigator or designee.
- Have 10 100 non-inflammatory lesions as determined by the Investigator or designee.
- Be willing to use the test products as instructed for 24 weeks.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Be willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol.
- Be willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and be able to read, speak, write, understand English and be willing to share personal information and data, as verified by signing a written authorization at the screening.
- Be willing to withhold all facial treatments during the course of the study including botulinum toxin, injectable fillers, microdermabrasion, IPL, peels, facials, laser treatments and tightening treatments. Waxing and threading is allowed but not facial laser hair removal.
- Males must be regular shavers and willing to shave on the day of the study visits (prior to clinic visits).
- Women of child bearing potential must be willing to take a urine pregnancy test prior to study enrollment, at week 24, and when deemed appropriate by the Investigator and/or Sponsor.
- Individuals of child bearing potential must use an acceptable method of contraception throughout the study. Acceptable methods of birth control include:
  - Oral and other system contraceptives. Individuals must be on a stable use for 3 months prior to study enrollment. Individuals on oral contraceptives must not alter their use, including dose or regimen for the duration of the study
  - Double barrier
  - o Bilateral tubal ligation (tubes tied)
  - Partner vasectomy
  - Abstinence
- Be willing to follow study requirements and report any changes in health status or medications, side effect symptoms, or reactions immediately.
- Be stable on any medication you are taking for at least 30 days

#### YOU CANNOT BE ON THE STUDY

## If you:

- Have been diagnosed with allergies to topical acne products.
- Have a condition and/or disease of the skin that the Investigator deems inappropriate for participation.
- Are a woman who is breastfeeding, pregnant, or planning to become pregnant during the study.
- Have pre-existing or dormant dermatologic conditions on the face (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, severe excoriations etc.) which in the opinion of the Investigator could interfere with the outcome of the study.
- Have a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.).
- Have an uncontrolled disease such as asthma, diabetes, hypertension, hyperthyroidism, or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc. at the Investigator's discretion.
- Are currently participating in another facial usage study or have participated in a clinical trial within 4 weeks prior to inclusion into the study.
- Have a history of skin cancer on the face within the past 5 years.
- Have any planned surgeries and/or invasive medical procedures during the course of the study.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Have started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to study entry or plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study.
- Have facial sunburn or excessive tanned facial skin or are not willing to avoid daily sun exposure on the face and the use of tanning beds or sunless tanning products for the duration of the study.
- Have severe acne, acne conglobata, multiple nodules or cysts (more than 2).
- Are currently taking a natural or prescription testosterone blocker (e.g. saw palmetto, blask cohosh, chaste tree, chasteberry, spironolactone, drospirenone, progestins).
- Are currently on a testosterone booster or prescription testosterone (e.g. DHEA, tribulus, testosterone cypionate, testosterone enanthate, Sustanon, testosterone propionate, testosterone phenylpropriate, Omnadren etc.).
- Are currently taking or have taken within the last 30 days oral or topical prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin (Retin A, Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo.
- Have used oral isotretinoin (Accutane) within the past 6-months.
- Are routinely using (3x a week or more) topical over-the-counter (OTC) acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 14 days of the study entry.
- Are using or have used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study.
- Have excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations as determined by the Investigator or designee.

## WHAT WILL HAPPEN DURING THE STUDY

## \*Visit 1: Screening (\* Visit 1 {Screening} AND Visit 2 {Baseline} may be combined into 1 Visit)

#### You will:

- Be given an IRB-approved Informed Consent Form (ICF), to read and sign. You will be given enough time to read the informed consent, and ask questions about the study, and sign 2 copies of this consent form. (1 for clinic records, 1 for your records)
- Be given an eligibility and health questionnaire to complete, and assigned a screening number.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Will be screened by the Investigator or designee to see if you qualify for the study.
- If you do qualify for the study, you will:
  - o Take a urine pregnancy test (females of child-bearing potential)
  - Have a dermatologist confirm your eligibility
  - Schedule your next appointment.

#### \*Visit 2: Baseline

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Be screened by the Investigator or designee to see if you still qualify for the study.
- Have your health and eligibility re-reviewed.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- If you still qualify for the study you will:
  - o Be assigned a subject number
  - o Have photos taken of your face
  - o Be randomly assigned to receive one of the test products & supporting facial cleanser, moisturizer & facial SPF 30
  - o Be provided verbal and written usage instructions, and a daily diary to record product use
  - Schedule your next appointment

## **Visits 3, 4 (Week 1, Week 2)**

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and returned to you. At week 2, your diary will be retained by the testing facility and you will be given a new diary
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

## Visits 5, 6 (Week 6, Week 12)

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and retained. New products will be dispensed as necessary.
- Schedule your next appointment

## <u>Visit 7</u> (Week 18)

- Be asked if you have experienced any changes in your health since the previous visit.
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

## Visit 8 (Week 24)

- Be asked if you have experienced any changes in your health since the previous visit.
- Take a urine pregnancy test (females of child-bearing potential).
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility.
- Have your product collected, weighed, and retained by the testing facility.

Do not give the study product to other people and keep it out of the reach of children.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

### RISKS OR DISCOMFORTS

If you do not understand what any of these side effects mean, please ask the investigator or study staff to explain these terms to you.

Because the study products are investigational, all of their side effects may not be known. There may be rare and unknown side effects. Some of these may be life threatening.

Possible risks associated with the product are, as with any other cosmetic and OTC products, signs of irritation including:

- Itching
- Burning
- Stinging
- Rash or other allergic reaction

- Tingling
- Scaling/Dryness
- Redness

In some cases, it is possible for a subject to develop allergic reactions to the test material(s). This risk is increased for individuals with a history of allergies, and individuals with asthma and/or a history of hives may also be affected. Symptoms include rash, hives, and itching.

You must tell the Investigator or study staff about all side effects that you have. If you are not honest about your side effects, it may not be safe for you to stay in the study.

## BIRTH CONTROL, DANGERS OF PREGNANCY AND BREASTFEEDING

If you are a female, you must not get pregnant while in this study. The only certain way to not get pregnant is to not have sex. If you are a female and choose to have sex, you must use a type of birth control.

Even if you use birth control during the study, there is a chance you could become pregnant. If you are pregnant or become pregnant during the study, test products or procedures may involve unforeseeable risks to the unborn baby.

A pregnancy test can be wrong. If you become pregnant during the study, stop using the test products and call/inform the Investigator at once.

You cannot be in the study if you are breastfeeding. It is not known whether the test products are safe for breast fed babies. Therefore if you are breastfeeding a child then it may not be safe for you to participate in the study.

## POSSIBLE BENEFITS OF THE STUDY

You will not get any medical benefit from being in this study, and there is no promise that your condition (acne) will get better. It might stay the same or it might get worse. Your participation will provide information that may help others. There may be other marketed products that claim to have similar benefits.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

## OTHER OPTIONS TO PARTICIPATING IN THE STUDY

Since this study is for research only, the only other choice would be not to be in the study.

#### STUDY AND TEST PRODUCT CONFIDENTIALITY

To participate in this study, you must agree to keep any information relating to the design, identity or use of these test product samples confidential.

On rare occasions, the sponsor may allow the testing company to disclose to you the name of the test products if you are not given this information during the study. This information is typically not provided until the end of the study or after the test products have been released for sale to the public. The study doctor or study staff will notify you if the sponsor allows us to give you this information.

#### DISCLOSURE AGREEMENT

This section explains how personal health information collected about you for the study may be used. Your personal health information includes, but is not limited to, information that was collected for your entry into the study and information that is collected during the study. The purpose of collecting this information is to allow the study staff and the Investigator to conduct the study, to evaluate the sponsor's study products and to analyze the study results.

You may decide not to give permission for the release of your personal health information for the study. In that case, you will not be able to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the sponsor's study products.

People who may inspect your personal and health information includes the Investigator, the Institutional Review Board, IntegReview IRB, FDA and other regulatory authorities from the United States or other countries, the study sponsor and people that work with the sponsor which includes, monitoring committees, contract research organizations, and consultants who have contracts with the company to do the study and review the study results. These reviews are done to check on the quality of the study and also for other purposes allowed by law.

The results of the study may be published in a medical book or journal, or presented at meetings for educational purposes. Neither your name, nor any other personal health information that specifically identifies you, will be used in those materials or presentations.

You may ask the Investigator to see and copy your personal health information related to the study. You may also ask the Investigator to correct any study related information about you that is wrong. You may have to wait until the end of the study to see your study records, so that the study can be organized properly.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the Investigator at the address below:

Thomas J. Stephens & Associates, Inc. 1801 North Glenville Drive, Suite 200 Richardson, TX 75081

If you cancel your permission after you have started in the study, the study staff and the Investigator will stop collecting your personal health information. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the study.

Thomas J. Stephens & Associates and the sponsor will make every effort to keep your personal health information private. But after the study staff or the Investigator share your personal health information from the study, federal privacy laws may not keep it private. There might be laws in your state or other federal laws that would protect the privacy of this information.

### **CONFIDENTIALITY**

Your records of being in this study will be kept private except when ordered by law. The following people will have access to your study records:

- The Investigator
- Sponsor company or research institution [including monitor(s) and auditor(s)]
- Other country, state or federal regulatory agencies
- IntegReview IRB

The Institutional Review Board (IRB), IntegReview, and accrediting agencies may inspect and copy your records, which may have your name on them. Therefore, total confidentiality cannot be guaranteed. If the study results are presented at meetings or printed in publications, your name will not be used.

## IN CASE OF STUDY RELATED INJURY

Side effects or complications, both foreseeable and unforeseeable, are possible in any research study without any fault to you, the Investigator, the study site, or the study sponsor. If you get hurt or sick as a direct result of being in this study, the sponsor will pay the costs of reasonable medical treatment. To ask questions about this, talk to the Investigator or study staff.

The sponsor's policy does not offer compensation for other expenses. Be aware that your health care payer/insurer might not cover the costs of study-related injuries or illnesses.

Unreimbursed medical expenses not covered by insurance or other third party coverage will be reimbursed by the sponsor for medical treatment for any injury that, in the opinion of the study doctor and the sponsor, is directly caused by the investigational product or by procedures required by the study protocol which would not have been performed as part of your regular medical care.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

### **LEGAL RIGHTS**

You will not lose any of your legal rights by signing this consent form.

### **CONTACT INFORMATION**

If you have questions, concerns, or complaints about this study or to report a study related injury, contact:

Lily Jiang, Ph.D. 972-392-1529 daytime telephone number 469-766-4781 after hours number

If you are unable to reach anyone at the number(s) listed above and you need medical attention, please go to the nearest emergency room.

If you do not want to talk to the Investigator or study staff, if you have concerns or complaints about the research, or to ask questions about your rights as a study subject you may contact IntegReview. IntegReview's policy indicates that all concerns/complaints are to be submitted in writing for review at a convened IRB meeting to:

| Mailing Address: | OR | Email Address: |
|----------------------------------|----|-----------------------------|
| Chairperson | | integreview@integreview.com |
| IntegReview IRB | | |
| 3815 S. Capital of Texas Highway | | |
| Suite 320 | | |
| Austin, TX 78704 | | |

If you are unable to provide your concerns/complaints in writing or if this is an emergency situation regarding subject safety, contact our office at:

512-326-3001 or toll free at 1-877-562-1589 between 8 a.m. and 5 p.m. Central Time

IntegReview has approved the information in this consent form and has given approval for the Investigator to do the study. This does not mean IntegReview has approved your being in the study. You must consider the information in this consent form for yourself and decide if you want to be in this study.

## PAYMENT FOR BEING IN THE STUDY

You may receive up to \$575.00 for being in the study. You will be paid per completed visit as follows:

| Visit | Compensation (amount) |
|------------------------------|-----------------------|
| Screening/Baseline (Visit 1) | \$40.00 |
| Week 1 (Visit 2) | \$60.00 |
| Week 2 (Visit 3) | \$65.00 |
| Week 6 (Visit 4) | \$75.00 |
| Week 12 (Visit 5) | \$90.00 |

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

VERSION CONTROL

clw/master: 2-17-16 snb/site: 2-20-16

| Week 18 (Visit 6) | \$95.00 |
|-------------------|----------|
| Week 24 (Visit 7) | \$150.00 |

If you choose to leave or are withdrawn from the study for any reason before finishing all visits you will be paid for each completed visit. You will receive payment within 2 weeks of final study visit.

If you do not qualify for any reason, you will be paid \$20.00, which will be mailed to you within 2 weeks of the baseline study visit.

If you are paid \$600.00 or more by Thomas J. Stephens & Associates, Inc. in a calendar year, those payments will be reported to the Internal Revenue Service via form 1099-MISC. As required by tax laws, if you withhold your social security number, Thomas J. Stephens & Associates, Inc. is required to withhold 28% of your payment for tax purposes. In this case a form 1099-MISC will be sent to you reporting your withholding.

## **VOLUNTEERING TO BE IN THE STUDY**

It is your choice if you want to be in the study. No one can force you to be in the study. You may not want to be in this study or you may leave the study at any time without penalty or loss of benefits to which you are otherwise entitled.

The Investigator, the sponsor company, or IntegReview may take you out of the study without your permission, at any time, for the following reasons:

- If you do not follow the Investigator's instructions
- If we find out you should not be in the study
- If the study is stopped
- If it becomes harmful to your health

If you leave the study or if you are taken out of the study, you may be asked to return for a final visit to have some end of study evaluations or tests. If information generated from this study is published or presented, your identity will not be revealed. If you leave the study, no more information about you will be collected for this study. However, all of the information you gave us before you left the study will still be used.

#### **NEW FINDINGS**

If there is new information or any significant new findings that could relate to your willingness to continue participation we will tell you. You can then decide if you still want to be in the study.

## THE REASON FOR INSTITUTIONAL REVIEW BOARDS AND INFORMED CONSENT

## What is a consent form?

The informed consent document contains information required by federal regulations. The informed consent document must be approved by an Institutional Review Board (IRB).

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

## What is an Institutional Review Board (IRB)?

An Institutional Review Board (IRB) is a group of people that reviews research studies. The main goal of this review is to protect the rights and well being of the human subjects participating in research studies.

## IntegReview, the IRB for this study

IntegReview is an IRB whose board members provide IRB services across the United States, Canada, Japan and Latin America.

To meet requirements of the law, the IntegReview Boards currently include:

- Doctors
- Pharmacists
- Nurses
- Toxicologists (people who study the harmful effects of chemicals)
- Other specialists
- Others who do not have a background in science/medicine

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

## AGREEMENT TO BE IN THE STUDY

This consent form contains important information to help you decide if you want to be in the study. If you have any questions that are not answered in this consent form, ask one of the study staff.

| Pleas | se answer YES or NO to the following questions: | |
|---|---|---|
| A. | Is this document in a language you understand? | |
| B. | B. Do you understand the information in this consent form? | |
| C. | C. Have you been given enough time to ask questions and talk about the study? | |
| D. | D. Have all of your questions been answered to your satisfaction? | |
| E. | Do you think you received enough information about the study? | |
| F. | Do you volunteer to be in this study of your own free will and without being pressured by the Investigator or study staff? | |
| G. | Do you know that you can leave the study at any time without giving a reason and without affecting your health care? | |
| Н. | Do you know that your health records from this study may be reviewed by the sponsor company and by government authorities? | |
| I. | Do you know that you cannot be in another study while you are in this study | y? |
| | IF YOU ANSWERED "NO" TO ANY OF THE ABOVE QUEST OR YOU ARE UNABLE TO ANSWER ANY OF THE ABOVE QUEST YOU SHOULD NOT SIGN THIS CONSENT FORM. | |
| Print | ed Name of Adult Study Subject | |
| Signa | nture of Adult Study Subject | Date |
| Print | ed Name of Person Explaining Consent Form | |
| Signa | ature of Person Explaining Consent Form | Date |
| You | will be given a signed and dated copy of this consent form to keep. | |

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

## **Authorization and Release Form**

I hereby for good and valuable consideration grant to Thomas J. Stephens & Associates, the study sponsor and their respective affiliates, agencies, agents, employees, and assigns (collectively, "Authorized Entities"), the unrestricted, royalty free, irrevocable and perpetual right and permission to reproduce, distribute, broadcast and/or otherwise use for advertising and other commercial/noncommercial purposes: (i) my name, likeness, image, video, and any other biographical or personal information ("Personal Content"); and (ii) any statement or endorsement, or any portions thereof ("Testimonial(s)"), made by me relating to the study sponsor's products ("Products"), in any and all media now known or later developed, worldwide in perpetuity, without further compensation or approval by me.

I hereby assign to the Authorized Entities all of my world-wide right, title and interest, including my copyright interests and all renewals, reissues and extensions thereof, in and to the Personal Content and Testimonial(s), including without limitation, any photographic portraits, sound recordings and video performances of and/or by me in connection with the Personal Content and/or Testimonial(s).

I am at least 21 years of age, and competent to contract in my own name. I have read and understand this

| Authorization and Release. | | |
|---|---|---|
| Printed Name of Adult Study Subject | | |
| Signature of Adult Study Subject | | Date |
| Printed Name of Person Explaining Release Form | | |
| Signature of Person Explaining Release Form | | Date |
| Copy of consent form given to subject on | (date) by | (initials) |
| You will be given a signed and dated copy of this con | nsent form to keep | |

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

# AUTHORIZATION TO USE AND DISCLOSE PERSONAL HEALTH INFORMATION FOR RESEARCH

THIS SECTION DESCRIBES YOUR RIGHTS AND HOW PERSONAL HEALTH INFORMATION COLLECTED ABOUT YOU DURING THIS STUDY MAY BE USED AND DISCLOSED AND HOW YOU CAN GET ACCESS TO THIS INFORMATION. PLEASE REVIEW IT CAREFULLY.

The United States government has issued a privacy rule to protect the privacy rights of patients. This rule was issued under a law called the Health Insurance Portability and Accountability Act of 1996 (HIPAA). The Privacy Rule is designed to protect the confidentiality of your personal health information. The document you are reading, called an "Authorization," describes your rights and explains how your health information will be used and disclosed (shared).

Federal law requires hospitals, researchers and health care providers to protect the privacy of information that identifies you and relates to your past, present and future physical and mental health or conditions.

All information collected during the study will be retained by the study doctor and the Study Sponsor, except as required by law. Information from this study will be given to the sponsor. "Sponsor" includes any persons or companies, which are contracted by the sponsor to have access to the research information during and after the study. The information will also be given to the U.S. Food and Drug Administration (FDA). Study records which identify you and the consent form signed by you will be inspected and/or copied for research or regulatory purposes by:

- Sponsor
- Agents for the sponsor
- The US Food and Drug Administration (FDA)
- Department of Health and Human Services (DHHS) agencies
- IntegReview IRB

Because of the need to release information to these parties, absolute confidentiality cannot be guaranteed. The results of this research study may be presented at meetings or in publications; however, your identity will not be disclosed in those presentations.

For purposes of study reporting, you will be identified by your initials and code numbers only. However, your name, date of birth, address, and phone number will be kept on record by the study doctor in case you need to be contacted in the future about this study.

After your personal health information is disclosed to the Study Sponsor, the results of the study may be reanalyzed at a later date and may be combined with the results of other studies. The Study Sponsor and people who work with the Study Sponsor may use the results of this study for other research purposes, including:

- Developing a better understanding of the disease;
- Improving the design of future actual use trials

After the study staff or the study doctor discloses your personal health information to others, it could be re-disclosed and no longer protected by federal privacy laws.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you do not withdraw this Authorization in writing, it will remain in effect indefinitely. Your study doctor will keep this Authorization for at least 6 years. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the study doctor at the address below:

Thomas J. Stephens & Associates, Inc. 1801 North Glenville Drive, Suite 200 Richardson, TX 75081

You have the right to see and get a copy of your records related to the study for as long as the study doctor has this information. However, by signing this Authorization you agree that you might not be able to review or receive some of your records related to the study until after the study has been completed.

If you cancel your permission after you have started in the study, the study staff and the study doctor will stop collecting your personal health information unless the information concerns an adverse event (a bad effect) related to the study. If an adverse event occurs, your entire medical record may be reviewed. All information that has already been collected for study purposes, and any new information about an adverse event related to the study, will be sent to the study sponsor. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the study doctor would not be able to collect the information needed to evaluate the study results.

If you withdraw from the study but do not withdraw your Authorization, new personal health information may be collected until this study ends.

You may decide not to give permission for the release of your personal health information for this study. In that case, you will not be able to participate. This is because the study staff and study doctor would not be able to collect the information needed to evaluate the study results.

At the completion of the study, you have the right to access your protected health information that is created during this research study that relates to your treatment or to payment, provided such information is not exempted under certain laws and regulations. To request this information, please contact the study doctor at the address listed above.

## **Your Right to Access Health Information**

Subject to certain exceptions prescribed by law, you have a right to request access to the health information that we hold about you and to request changes if your health information is incorrect or incomplete. Any request for access or corrections should be made to the principal doctor conducting this study.

Your records obtained while you are in this trial, as well as related health records, will remain strictly confidential at all times. However, these will need to be made available to others working on the Sponsor's behalf, the Independent Ethics Committee members and Medicines Regulatory Authorities.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

By signing the consent form you agree to this access for the current trial and any further research that may be done. However, the Sponsor will take steps to protect your personal information and will not include your name on any sponsor forms, reports, publications, or in any future disclosures. If you withdraw from the study, we will no longer collect your personal information, but we may need to continue to use information already collected.

Personal data which may be sensitive (e.g., date of birth) will be collected and processed, but only for research purposes in connection with this trial.

The trial data will be sent around the world, but you will not be referred to by name or identified in any report or publication nor could the data be traced back to you. Your data may be transferred to a country that does not have the same level of personal data protection as within the United States. However, The Sponsor maintains high standards of confidentiality and protection.

The Sponsor (who will control the use of the data) will take steps to ensure your personal data is protected.

By taking part in this trial you agree not to restrict the use of any data even if you withdraw from the trial and agree to the transfer of your personal data to other Sponsor companies and to Medicines Regulatory Authorities both within and outside of Europe.

| Printed Name of Adult Study Subject | |
|-------------------------------------|------|
| Signature of Adult Study Subject | Date |

THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

# INFORMED CONSENT DOCUMENT AGREEMENT TO BE IN A RESEARCH STUDY

**NAME OF TESTING COMPANY:** Thomas J. Stephens & Associates, Inc.

NUMBER AND TITLE OF STUDY: C16-CD020 (GLI.04.SPR.US10354); "A Multi-

Center Clinical Trial to Evaluate the Efficacy of

Two Acne Treatments"

NAME OF PERSON IN CHARGE OF

THE RESEARCH STUDY

(STUDY DOCTOR/INVESTIGATOR): Lily Jiang, Ph.D.

**TELEPHONE NUMBER(S), DAYTIME:** 972-392-1529 **AFTER HOURS:** 469-766-4781

### INTRODUCTION

You are being invited to volunteer for a clinical research study. You must read and sign this form before you agree to take part in this study. This form will give you more information about this study. Please ask as many questions as you need to before you decide if you want to be in the study. You should not sign this form if you have any questions that have not been answered.

Thomas J. Stephens & Associates, Inc., a contract research organization, is being paid by the sponsor (the company paying for this study) to conduct this research study.

You must be honest with the Investigator about your health history or it may not be safe for you to be in this study.

## **PURPOSE OF THE STUDY**

The purpose of this study is to evaluate the efficiency of 2 acne treatments for 24 weeks of use in adult men and women with mild to moderate facial acne, at least 5 inflammatory lesions, and at least 10 - 100 non-inflammatory lesions.

## HOW LONG THE STUDY WILL LAST AND HOW MANY PEOPLE WILL BE IN THE STUDY

This study will last 24 weeks and have up to 8 visits. At least 100 subjects, men and women between the ages of 21-45, are expected to complete this study, with at least 50 subjects completed per cell.

## TO BE IN THIS STUDY

### You must:

- Be a man or woman age 21 to 45 years at the time of enrollment.
- Have mild to moderate acne on the face as determined by the Investigator or designee.
- Have at least 5 inflammatory lesions as determined by the Investigator or designee.
- Have 10 100 non-inflammatory lesions as determined by the Investigator or designee.
- Be willing to use the test products as instructed for 24 weeks.
- Be willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Be willing to provide written informed consent including photo release, Health Insurance Portability
  and Accountability Act (HIPAA), and be able to read, speak, write, understand English and be willing
  to share personal information and data, as verified by signing a written authorization at the screening.
- Be willing to withhold all facial treatments during the course of the study including botulinum toxin, injectable fillers, microdermabrasion, IPL, peels, facials, laser treatments and tightening treatments. Waxing and threading is allowed but not facial laser hair removal.
- Males must be regular shavers and willing to shave on the day of the study visits (prior to clinic visits).
- Women of child bearing potential must be willing to take a urine pregnancy test prior to study enrollment, at week 24, and when deemed appropriate by the Investigator and/or Sponsor.
- Individuals of child bearing potential must use an acceptable method of contraception throughout the study. Acceptable methods of birth control include:
  - Oral and other system contraceptives. Individuals must be on a stable use for 3 months prior to study enrollment. Individuals on oral contraceptives must not alter their use, including dose or regimen for the duration of the study
  - o Double barrier
  - o Bilateral tubal ligation (tubes tied)
  - o Partner vasectomy
  - Abstinence
- Be willing to follow study requirements and report any changes in health status or medications, side effect symptoms, or reactions immediately.
- Be stable on any medication you are taking for at least 30 days

### YOU CANNOT BE ON THE STUDY

## If you:

- Have been diagnosed with allergies to topical acne products.
- Have a condition and/or disease of the skin that the Investigator deems inappropriate for participation.
- Are a woman who is breastfeeding, pregnant, or planning to become pregnant during the study.
- Have pre-existing or dormant dermatologic conditions on the face (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, severe excoriations etc.) which in the opinion of the Investigator could interfere with the outcome of the study.
- Have a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.).
- Have an uncontrolled disease such as asthma, diabetes, hypertension, hyperthyroidism, or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc. at the Investigator's discretion.
- Are currently participating in another facial usage study or have participated in a clinical trial within 4 weeks prior to inclusion into the study.
- Have a history of skin cancer on the face within the past 5 years.
- Have any planned surgeries and/or invasive medical procedures during the course of the study.
- Have started hormone replacement therapies (HRT) or hormones for birth control less than 3 months
  prior to study entry or plan on starting, stopping, or changing doses of HRT or hormones for birth
  control during the study.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Have facial sunburn or excessive tanned facial skin or are not willing to avoid daily sun exposure on the face and the use of tanning beds or sunless tanning products for the duration of the study.
- Have severe acne, acne conglobata, multiple nodules or cysts (more than 2).
- Are currently taking a natural or prescription testosterone blocker (e.g. saw palmetto, blask cohosh, chaste tree, chasteberry, spironolactone, drospirenone, progestins).
- Are currently on a testosterone booster or prescription testosterone (e.g. DHEA, tribulus, testosterone cypionate, testosterone enanthate, Sustanon, testosterone propionate, testosterone phenylpropriate, Omnadren etc.).
- Are currently taking or have taken within the last 30 days oral or topical prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin (Retin A, Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo.
- Have used oral isotretinoin (Accutane) within the past 6-months.
- Are routinely using (3x a week or more) topical over-the-counter (OTC) acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 14 days of the study entry.
- Are using or have used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study.
- Have excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations as determined by the Investigator or designee.

### WHAT WILL HAPPEN DURING THE STUDY

## \*Visit 1: Screening (\* Visit 1 {Screening} AND Visit 2 {Baseline} may be combined into 1 Visit)

## You will:

- Be given an IRB-approved Informed Consent Form (ICF), to read and sign. You will be given enough time to read the informed consent, and ask questions about the study, and sign 2 copies of this consent form. (1 for clinic records, 1 for your records)
- Be given an eligibility and health questionnaire to complete, and assigned a screening number.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Will be screened by the Investigator or designee to see if you qualify for the study.
- If you do qualify for the study, you will:
  - o Take a urine pregnancy test (females of child-bearing potential)
  - Have a dermatologist confirm your eligibility
  - o Schedule your next appointment.

## \*Visit 2: Baseline

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Be screened by the Investigator or designee to see if you still qualify for the study.
- Have your health and eligibility re-reviewed.
- If you still qualify for the study you will:
  - o Be assigned a subject number
  - Have photos taken of your face

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Be randomly assigned to receive one of the test products & supporting facial cleanser, moisturizer & facial SPF 30
- o Be provided verbal and written usage instructions, and a daily diary to record product use
- Schedule your next appointment

## **Visits 3, 4 (Week 1, Week 2)**

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and returned to you. At week 2, your diary
  will be retained by the testing facility and you will be given a new diary
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

## Visits 5, 6 (Week 6, Week 12)

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and retained. New products will be dispensed as necessary.
- Schedule your next appointment

## Visit 7 (Week 18)

- Be asked if you have experienced any changes in your health since the previous visit.
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

## <u>Visit 8 (Week 24)</u>

- Be asked if you have experienced any changes in your health since the previous visit.
- Take a urine pregnancy test (females of child-bearing potential).
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility.
- Have your product collected, weighed, and retained by the testing facility.

Do not give the study product to other people and keep it out of the reach of children.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

### RISKS OR DISCOMFORTS

If you do not understand what any of these side effects mean, please ask the investigator or study staff to explain these terms to you.

Because the study products are investigational, all of their side effects may not be known. There may be rare and unknown side effects. Some of these may be life threatening.

Possible risks associated with the product are, as with any other cosmetic and OTC products, signs of irritation including:

- Itching
- Burning
- Stinging
- Rash or other allergic reaction

- Tingling
- Scaling/Dryness
- Redness

In some cases, it is possible for a subject to develop allergic reactions to the test material(s). This risk is increased for individuals with a history of allergies, and individuals with asthma and/or a history of hives may also be affected. Symptoms include rash, hives, and itching.

You must tell the Investigator or study staff about all side effects that you have. If you are not honest about your side effects, it may not be safe for you to stay in the study.

## BIRTH CONTROL, DANGERS OF PREGNANCY AND BREASTFEEDING

If you are a female, you must not get pregnant while in this study. The only certain way to not get pregnant is to not have sex. If you are a female and choose to have sex, you must use a type of birth control.

Even if you use birth control during the study, there is a chance you could become pregnant. If you are pregnant or become pregnant during the study, test products or procedures may involve unforeseeable risks to the unborn baby.

A pregnancy test can be wrong. If you become pregnant during the study, stop using the test products and call/inform the Investigator at once.

You cannot be in the study if you are breastfeeding. It is not known whether the test products are safe for breast fed babies. Therefore if you are breastfeeding a child then it may not be safe for you to participate in the study.

## POSSIBLE BENEFITS OF THE STUDY

You will not get any medical benefit from being in this study, and there is no promise that your condition (acne) will get better. It might stay the same or it might get worse. Your participation will provide information that may help others. There may be other marketed products that claim to have similar benefits.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

### OTHER OPTIONS TO PARTICIPATING IN THE STUDY

Since this study is for research only, the only other choice would be not to be in the study.


To participate in this study, you must agree to keep any information relating to the design, identity or use of these test product samples confidential.

On rare occasions, the sponsor may allow the testing company to disclose to you the name of the test products if you are not given this information during the study. This information is typically not provided until the end of the study or after the test products have been released for sale to the public. The study doctor or study staff will notify you if the sponsor allows us to give you this information.

#### DISCLOSURE AGREEMENT

This section explains how personal health information collected about you for the study may be used. Your personal health information includes, but is not limited to, information that was collected for your entry into the study and information that is collected during the study. The purpose of collecting this information is to allow the study staff and the Investigator to conduct the study, to evaluate the sponsor's study products and to analyze the study results.

You may decide not to give permission for the release of your personal health information for the study. In that case, you will not be able to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the sponsor's study products.

People who may inspect your personal and health information includes the Investigator, the Institutional Review Board, IntegReview IRB, FDA and other regulatory authorities from the United States or other countries, the study sponsor and people that work with the sponsor which includes, monitoring committees, contract research organizations, and consultants who have contracts with the company to do the study and review the study results. These reviews are done to check on the quality of the study and also for other purposes allowed by law.

The results of the study may be published in a medical book or journal, or presented at meetings for educational purposes. Neither your name, nor any other personal health information that specifically identifies you, will be used in those materials or presentations.

You may ask the Investigator to see and copy your personal health information related to the study. You may also ask the Investigator to correct any study related information about you that is wrong. You may have to wait until the end of the study to see your study records, so that the study can be organized properly.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the Investigator at the address below:

Thomas J. Stephens & Associates, Inc. 1801 North Glenville Drive, Suite 200 Richardson, TX 75081

If you cancel your permission after you have started in the study, the study staff and the Investigator will stop collecting your personal health information. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the study.

Thomas J. Stephens & Associates and the sponsor will make every effort to keep your personal health information private. But after the study staff or the Investigator share your personal health information from the study, federal privacy laws may not keep it private. There might be laws in your state or other federal laws that would protect the privacy of this information.

### **CONFIDENTIALITY**

Your records of being in this study will be kept private except when ordered by law. The following people will have access to your study records:

- The Investigator
- Sponsor company or research institution [including monitor(s) and auditor(s)]
- Other country, state or federal regulatory agencies
- IntegReview IRB

The Institutional Review Board (IRB), IntegReview, and accrediting agencies may inspect and copy your records, which may have your name on them. Therefore, total confidentiality cannot be guaranteed. If the study results are presented at meetings or printed in publications, your name will not be used.

## IN CASE OF STUDY RELATED INJURY

Side effects or complications, both foreseeable and unforeseeable, are possible in any research study without any fault to you, the Investigator, the study site, or the study sponsor. If you get hurt or sick as a direct result of being in this study, the sponsor will pay the costs of reasonable medical treatment. To ask questions about this, talk to the Investigator or study staff.

The sponsor's policy does not offer compensation for other expenses. Be aware that your health care payer/insurer might not cover the costs of study-related injuries or illnesses.

Unreimbursed medical expenses not covered by insurance or other third party coverage will be reimbursed by the sponsor for medical treatment for any injury that, in the opinion of the study doctor and the sponsor, is directly caused by the investigational product or by procedures required by the study protocol which would not have been performed as part of your regular medical care.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

### **LEGAL RIGHTS**

You will not lose any of your legal rights by signing this consent form.

### **CONTACT INFORMATION**

If you have questions, concerns, or complaints about this study or to report a study related injury, contact:

Lily Jiang, Ph.D. 972-392-1529 daytime telephone number 469-766-4781 after hours number

If you are unable to reach anyone at the number(s) listed above and you need medical attention, please go to the nearest emergency room.

If you do not want to talk to the Investigator or study staff, if you have concerns or complaints about the research, or to ask questions about your rights as a study subject you may contact IntegReview. IntegReview's policy indicates that all concerns/complaints are to be submitted in writing for review at a convened IRB meeting to:

| Mailing Address: | OR | Email Address: |
|----------------------------------|----|-----------------------------|
| Chairperson | | integreview@integreview.com |
| IntegReview IRB | | |
| 3815 S. Capital of Texas Highway | | |
| Suite 320 | | |
| Austin, TX 78704 | | |

If you are unable to provide your concerns/complaints in writing or if this is an emergency situation regarding subject safety, contact our office at:

512-326-3001 or toll free at 1-877-562-1589 between 8 a.m. and 5 p.m. Central Time

IntegReview has approved the information in this consent form and has given approval for the Investigator to do the study. This does not mean IntegReview has approved your being in the study. You must consider the information in this consent form for yourself and decide if you want to be in this study.

## PAYMENT FOR BEING IN THE STUDY

You may receive up to \$575.00 for being in the study. You will be paid per completed visit as follows:

| Visit | Compensation (amount) |
|------------------------------|-----------------------|
| Screening/Baseline (Visit 1) | \$40.00 |
| Week 1 (Visit 2) | \$60.00 |
| Week 2 (Visit 3) | \$65.00 |
| Week 6 (Visit 4) | \$75.00 |
| Week 12 (Visit 5) | \$90.00 |

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

VERSION CONTROL

clw/master: 2-17-16 snb/site: 2-20-16 rss/master: 9-16-16

| Week 18 (Visit 6) | \$95.00 |
|-------------------|----------|
| Week 24 (Visit 7) | \$150.00 |

If you choose to leave or are withdrawn from the study for any reason before finishing all visits you will be paid for each completed visit. You will receive payment within 2 weeks of final study visit.

If you do not qualify for any reason, you will be paid \$20.00, which will be mailed to you within 2 weeks of the baseline study visit.

If you are paid \$600.00 or more by Thomas J. Stephens & Associates, Inc. in a calendar year, those payments will be reported to the Internal Revenue Service via form 1099-MISC. As required by tax laws, if you withhold your social security number, Thomas J. Stephens & Associates, Inc. is required to withhold 28% of your payment for tax purposes. In this case a form 1099-MISC will be sent to you reporting your withholding.

## **VOLUNTEERING TO BE IN THE STUDY**

It is your choice if you want to be in the study. No one can force you to be in the study. You may not want to be in this study or you may leave the study at any time without penalty or loss of benefits to which you are otherwise entitled.

The Investigator, the sponsor company, or IntegReview may take you out of the study without your permission, at any time, for the following reasons:

- If you do not follow the Investigator's instructions
- If we find out you should not be in the study
- If the study is stopped
- If it becomes harmful to your health

If you leave the study or if you are taken out of the study, you may be asked to return for a final visit to have some end of study evaluations or tests. If information generated from this study is published or presented, your identity will not be revealed. If you leave the study, no more information about you will be collected for this study. However, all of the information you gave us before you left the study will still be used.

#### **NEW FINDINGS**

If there is new information or any significant new findings that could relate to your willingness to continue participation we will tell you. You can then decide if you still want to be in the study.

## THE REASON FOR INSTITUTIONAL REVIEW BOARDS AND INFORMED CONSENT

## What is a consent form?

The informed consent document contains information required by federal regulations. The informed consent document must be approved by an Institutional Review Board (IRB).

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

## What is an Institutional Review Board (IRB)?

An Institutional Review Board (IRB) is a group of people that reviews research studies. The main goal of this review is to protect the rights and well being of the human subjects participating in research studies.

## IntegReview, the IRB for this study

IntegReview is an IRB whose board members provide IRB services across the United States, Canada, Japan and Latin America.

To meet requirements of the law, the IntegReview Boards currently include:

- Doctors
- Pharmacists
- Nurses
- Toxicologists (people who study the harmful effects of chemicals)
- Other specialists
- Others who do not have a background in science/medicine

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

## AGREEMENT TO BE IN THE STUDY

This consent form contains important information to help you decide if you want to be in the study. If you have any questions that are not answered in this consent form, ask one of the study staff.

| Pleas | e answer YES or NO to the following questions: | |
|---|---|---|
| A. | Is this document in a language you understand? | |
| B. | Do you understand the information in this consent form? | |
| C. | . Have you been given enough time to ask questions and talk about the study? | |
| D. | Have all of your questions been answered to your satisfaction? | |
| E. | Do you think you received enough information about the study? | |
| F. | Do you volunteer to be in this study of your own free will and without being pressured by the Investigator or study staff? | |
| G. | Do you know that you can leave the study at any time without giving a reason and without affecting your health care? | |
| Н. | Do you know that your health records from this study may be reviewed by the sponsor company and by government authorities? | |
| I. | Do you know that you cannot be in another study while you are in this study? | |
| | IF YOU ANSWERED "NO" TO ANY OF THE ABOVE QUESTIO OR YOU ARE UNABLE TO ANSWER ANY OF THE ABOVE QUES' YOU SHOULD NOT SIGN THIS CONSENT FORM. | |
| Print | ed Name of Adult Study Subject | |
| Signa | nture of Adult Study Subject | Date |
| Print | ed Name of Person Explaining Consent Form | |
| Signa | nture of Person Explaining Consent Form | Date |
| You | will be given a signed and dated copy of this consent form to keep. | |

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

## **Authorization and Release Form**

I hereby for good and valuable consideration grant to Thomas J. Stephens & Associates, the study sponsor and their respective affiliates, agencies, agents, employees, and assigns (collectively, "Authorized Entities"), the unrestricted, royalty free, irrevocable and perpetual right and permission to reproduce, distribute, broadcast and/or otherwise use for advertising and other commercial/noncommercial purposes: (i) my name, likeness, image, video, and any other biographical or personal information ("Personal Content"); and (ii) any statement or endorsement, or any portions thereof ("Testimonial(s)"), made by me relating to the study sponsor's products ("Products"), in any and all media now known or later developed, worldwide in perpetuity, without further compensation or approval by me.

I hereby assign to the Authorized Entities all of my world-wide right, title and interest, including my copyright interests and all renewals, reissues and extensions thereof, in and to the Personal Content and Testimonial(s), including without limitation, any photographic portraits, sound recordings and video performances of and/or by me in connection with the Personal Content and/or Testimonial(s).

I am at least 21 years of age, and competent to contract in my own name. I have read and understand this

| Authorization and Release. | | |
|---|---|---|
| Printed Name of Adult Study Subject | | |
| Signature of Adult Study Subject | | Date |
| Printed Name of Person Explaining Release Form | | |
| Signature of Person Explaining Release Form | | Date |
| Copy of consent form given to subject on | (date) by | (initials) |
| You will be given a signed and dated copy of this con | nsent form to keep | |

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

# AUTHORIZATION TO USE AND DISCLOSE PERSONAL HEALTH INFORMATION FOR RESEARCH

THIS SECTION DESCRIBES YOUR RIGHTS AND HOW PERSONAL HEALTH INFORMATION COLLECTED ABOUT YOU DURING THIS STUDY MAY BE USED AND DISCLOSED AND HOW YOU CAN GET ACCESS TO THIS INFORMATION. PLEASE REVIEW IT CAREFULLY.

The United States government has issued a privacy rule to protect the privacy rights of patients. This rule was issued under a law called the Health Insurance Portability and Accountability Act of 1996 (HIPAA). The Privacy Rule is designed to protect the confidentiality of your personal health information. The document you are reading, called an "Authorization," describes your rights and explains how your health information will be used and disclosed (shared).

Federal law requires hospitals, researchers and health care providers to protect the privacy of information that identifies you and relates to your past, present and future physical and mental health or conditions.

All information collected during the study will be retained by the study doctor and the Study Sponsor, except as required by law. Information from this study will be given to the sponsor. "Sponsor" includes any persons or companies, which are contracted by the sponsor to have access to the research information during and after the study. The information will also be given to the U.S. Food and Drug Administration (FDA). Study records which identify you and the consent form signed by you will be inspected and/or copied for research or regulatory purposes by:

- Sponsor
- Agents for the sponsor
- The US Food and Drug Administration (FDA)
- Department of Health and Human Services (DHHS) agencies
- IntegReview IRB

Because of the need to release information to these parties, absolute confidentiality cannot be guaranteed. The results of this research study may be presented at meetings or in publications; however, your identity will not be disclosed in those presentations.

For purposes of study reporting, you will be identified by your initials and code numbers only. However, your name, date of birth, address, and phone number will be kept on record by the study doctor in case you need to be contacted in the future about this study.

After your personal health information is disclosed to the Study Sponsor, the results of the study may be reanalyzed at a later date and may be combined with the results of other studies. The Study Sponsor and people who work with the Study Sponsor may use the results of this study for other research purposes, including:

- Developing a better understanding of the disease;
- Improving the design of future actual use trials

After the study staff or the study doctor discloses your personal health information to others, it could be re-disclosed and no longer protected by federal privacy laws.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you do not withdraw this Authorization in writing, it will remain in effect indefinitely. Your study doctor will keep this Authorization for at least 6 years. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the study doctor at the address below:

Thomas J. Stephens & Associates, Inc. 1801 North Glenville Drive, Suite 200 Richardson, TX 75081

You have the right to see and get a copy of your records related to the study for as long as the study doctor has this information. However, by signing this Authorization you agree that you might not be able to review or receive some of your records related to the study until after the study has been completed.

If you cancel your permission after you have started in the study, the study staff and the study doctor will stop collecting your personal health information unless the information concerns an adverse event (a bad effect) related to the study. If an adverse event occurs, your entire medical record may be reviewed. All information that has already been collected for study purposes, and any new information about an adverse event related to the study, will be sent to the study sponsor. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the study doctor would not be able to collect the information needed to evaluate the study results.

If you withdraw from the study but do not withdraw your Authorization, new personal health information may be collected until this study ends.

You may decide not to give permission for the release of your personal health information for this study. In that case, you will not be able to participate. This is because the study staff and study doctor would not be able to collect the information needed to evaluate the study results.

At the completion of the study, you have the right to access your protected health information that is created during this research study that relates to your treatment or to payment, provided such information is not exempted under certain laws and regulations. To request this information, please contact the study doctor at the address listed above.

## **Your Right to Access Health Information**

Subject to certain exceptions prescribed by law, you have a right to request access to the health information that we hold about you and to request changes if your health information is incorrect or incomplete. Any request for access or corrections should be made to the principal doctor conducting this study.

Your records obtained while you are in this trial, as well as related health records, will remain strictly confidential at all times. However, these will need to be made available to others working on the Sponsor's behalf, the Independent Ethics Committee members and Medicines Regulatory Authorities.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

By signing the consent form you agree to this access for the current trial and any further research that may be done. However, the Sponsor will take steps to protect your personal information and will not include your name on any sponsor forms, reports, publications, or in any future disclosures. If you withdraw from the study, we will no longer collect your personal information, but we may need to continue to use information already collected.

Personal data which may be sensitive (e.g., date of birth) will be collected and processed, but only for research purposes in connection with this trial.

The trial data will be sent around the world, but you will not be referred to by name or identified in any report or publication nor could the data be traced back to you. Your data may be transferred to a country that does not have the same level of personal data protection as within the United States. However, The Sponsor maintains high standards of confidentiality and protection.

The Sponsor (who will control the use of the data) will take steps to ensure your personal data is protected.

By taking part in this trial you agree not to restrict the use of any data even if you withdraw from the trial and agree to the transfer of your personal data to other Sponsor companies and to Medicines Regulatory Authorities both within and outside of Europe.

| Printed Name of Adult Study Subject | |
|-------------------------------------|------|
| Signature of Adult Study Subject | Date |

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

# INFORMED CONSENT DOCUMENT AGREEMENT TO BE IN A RESEARCH STUDY

**NAME OF TESTING COMPANY:** Thomas J. Stephens & Associates, Inc.

NUMBER AND TITLE OF STUDY: C16-CD020 (GLI.04.SPR.US10354); "A Multi-

Center Clinical Trial to Evaluate the Efficacy of

Two Acne Treatments"

NAME OF PERSON IN CHARGE OF

THE RESEARCH STUDY

(STUDY DOCTOR/INVESTIGATOR): Kun Qian, M.D.

**TELEPHONE NUMBER(S), DAYTIME:** 719-637-2828 **AFTER HOURS:** 719-471-1763

## INTRODUCTION

You are being invited to volunteer for a clinical research study. You must read and sign this form before you agree to take part in this study. This form will give you more information about this study. Please ask as many questions as you need to before you decide if you want to be in the study. You should not sign this form if you have any questions that have not been answered.

Thomas J. Stephens & Associates, Inc., a contract research organization, is being paid by the sponsor (the company paying for this study) to conduct this research study.

You must be honest with the Investigator about your health history or it may not be safe for you to be in this study.

### PURPOSE OF THE STUDY

The purpose of this study is to evaluate the efficiency of 2 acne treatments for 24 weeks of use in adult men and women with mild to moderate facial acne, at least 5 inflammatory lesions, and at least 10 - 100 non-inflammatory lesions.

## HOW LONG THE STUDY WILL LAST AND HOW MANY PEOPLE WILL BE IN THE STUDY

This study will last 24 weeks and have up to 8 visits. At least 100 subjects, men and women between the ages of 21-45, are expected to complete this study, with at least 50 subjects completed per cell. Each site is to enroll no more than 40 subjects, with at least 100 subjects expected to complete when combined.

## TO BE IN THIS STUDY

## You must:

- Be a man or woman age 21 to 45 years at the time of enrollment.
- Have mild to moderate acne on the face as determined by the Investigator or designee.
- Have at least 5 inflammatory lesions as determined by the Investigator or designee.
- Have 10 100 non-inflammatory lesions as determined by the Investigator or designee.
- Be willing to use the test products as instructed for 24 weeks.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Be willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol.
- Be willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and be able to read, speak, write, understand English and be willing to share personal information and data, as verified by signing a written authorization at the screening.
- Be willing to withhold all facial treatments during the course of the study including botulinum toxin, injectable fillers, microdermabrasion, IPL, peels, facials, laser treatments and tightening treatments. Waxing and threading is allowed but not facial laser hair removal.
- Males must be regular shavers and willing to shave on the day of the study visits (prior to clinic visits).
- Women of child bearing potential must be willing to take a urine pregnancy test prior to study enrollment, at week 24, and when deemed appropriate by the Investigator and/or Sponsor.
- Individuals of child bearing potential must use an acceptable method of contraception throughout the study. Acceptable methods of birth control include:
  - Oral and other system contraceptives. Individuals must be on a stable use for 3 months prior to study enrollment. Individuals on oral contraceptives must not alter their use, including dose or regimen for the duration of the study
  - Double barrier
  - Bilateral tubal ligation (tubes tied)
  - Partner vasectomy
  - Abstinence
- Be willing to follow study requirements and report any changes in health status or medications, side effect symptoms, or reactions immediately.
- Be stable on any medication you are taking for at least 30 days

#### YOU CANNOT BE ON THE STUDY

## If you:

- Have been diagnosed with allergies to topical acne products.
- Have a condition and/or disease of the skin that the Investigator deems inappropriate for participation.
- Are a woman who is breastfeeding, pregnant, or planning to become pregnant during the study.
- Have pre-existing or dormant dermatologic conditions on the face (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, severe excoriations etc.) which in the opinion of the Investigator could interfere with the outcome of the study.
- Have a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.).
- Have an uncontrolled disease such as asthma, diabetes, hypertension, hyperthyroidism, or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc. at the Investigator's discretion.
- Are currently participating in another facial usage study or have participated in a clinical trial within 4 weeks prior to inclusion into the study.
- Have a history of skin cancer on the face within the past 5 years.
- Have any planned surgeries and/or invasive medical procedures during the course of the study.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Have started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to study entry or plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study.
- Have facial sunburn or excessive tanned facial skin or are not willing to avoid daily sun exposure on the face and the use of tanning beds or sunless tanning products for the duration of the study.
- Have severe acne, acne conglobata, multiple nodules or cysts (more than 2).
- Are currently taking a natural or prescription testosterone blocker (e.g. saw palmetto, blask cohosh, chaste tree, chasteberry, spironolactone, drospirenone, progestins).
- Are currently on a testosterone booster or prescription testosterone (e.g. DHEA, tribulus, testosterone cypionate, testosterone enanthate, Sustanon, testosterone propionate, testosterone phenylpropriate, Omnadren etc.).
- Are currently taking or have taken within the last 30 days oral or topical prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin (Retin A, Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo.
- Have used oral isotretinoin (Accutane) within the past 6-months.
- Are routinely using (3x a week or more) topical over-the-counter (OTC) acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 14 days of the study entry.
- Are using or have used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study.
- Have excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations as determined by the Investigator or designee.

## WHAT WILL HAPPEN DURING THE STUDY

## \*Visit 1: Screening (\* Visit 1 {Screening} AND Visit 2 {Baseline} may be combined into 1 Visit)

#### You will:

- Be given an IRB-approved Informed Consent Form (ICF), to read and sign. You will be given enough time to read the informed consent, and ask questions about the study, and sign 2 copies of this consent form. (1 for clinic records, 1 for your records)
- Be given an eligibility and health questionnaire to complete, and assigned a screening number.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Will be screened by the Investigator or designee to see if you qualify for the study.
- If you do qualify for the study, you will:
  - o Take a urine pregnancy test (females of child-bearing potential)
  - Have a dermatologist confirm your eligibility
  - Schedule your next appointment.

#### \*Visit 2: Baseline

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Be screened by the Investigator or designee to see if you still qualify for the study.
- Have your health and eligibility re-reviewed.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- If you still qualify for the study you will:
  - o Be assigned a subject number
  - o Have photos taken of your face
  - o Be randomly assigned to receive one of the test products & supporting facial cleanser, moisturizer & facial SPF 30
  - o Be provided verbal and written usage instructions, and a daily diary to record product use
  - Schedule your next appointment

## **Visits 3, 4 (Week 1, Week 2)**

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and returned to you. At week 2, your diary will be retained by the testing facility and you will be given a new diary
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

## Visits 5, 6 (Week 6, Week 12)

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and retained. New products will be dispensed as necessary.
- Schedule your next appointment

## **Visit 7** (Week 18)

- Be asked if you have experienced any changes in your health since the previous visit.
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

## **Visit 8 (Week 24)**

- Be asked if you have experienced any changes in your health since the previous visit.
- Take a urine pregnancy test (females of child-bearing potential).
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility.
- Have your product collected, weighed, and retained by the testing facility.

Do not give the study product to other people and keep it out of the reach of children.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

### RISKS OR DISCOMFORTS

If you do not understand what any of these side effects mean, please ask the investigator or study staff to explain these terms to you.

Because the study products are investigational, all of their side effects may not be known. There may be rare and unknown side effects. Some of these may be life threatening.

Possible risks associated with the product are, as with any other cosmetic and OTC products, signs of irritation including:

- Itching
- Burning
- Stinging
- Rash or other allergic reaction

- Tingling
- Scaling/Dryness
- Redness

In some cases, it is possible for a subject to develop allergic reactions to the test material(s). This risk is increased for individuals with a history of allergies, and individuals with asthma and/or a history of hives may also be affected. Symptoms include rash, hives, and itching.

You must tell the Investigator or study staff about all side effects that you have. If you are not honest about your side effects, it may not be safe for you to stay in the study.

## BIRTH CONTROL, DANGERS OF PREGNANCY AND BREASTFEEDING

If you are a female, you must not get pregnant while in this study. The only certain way to not get pregnant is to not have sex. If you are a female and choose to have sex, you must use a type of birth control.

Even if you use birth control during the study, there is a chance you could become pregnant. If you are pregnant or become pregnant during the study, test products or procedures may involve unforeseeable risks to the unborn baby.

A pregnancy test can be wrong. If you become pregnant during the study, stop using the test products and call/inform the Investigator at once.

You cannot be in the study if you are breastfeeding. It is not known whether the test products are safe for breast fed babies. Therefore if you are breastfeeding a child then it may not be safe for you to participate in the study.

## POSSIBLE BENEFITS OF THE STUDY

You will not get any medical benefit from being in this study, and there is no promise that your condition (acne) will get better. It might stay the same or it might get worse. Your participation will provide information that may help others. There may be other marketed products that claim to have similar benefits.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE
#### OTHER OPTIONS TO PARTICIPATING IN THE STUDY

Since this study is for research only, the only other choice would be not to be in the study.


To participate in this study, you must agree to keep any information relating to the design, identity or use of these test product samples confidential.

On rare occasions, the sponsor may allow the testing company to disclose to you the name of the test products if you are not given this information during the study. This information is typically not provided until the end of the study or after the test products have been released for sale to the public. The study doctor or study staff will notify you if the sponsor allows us to give you this information.

#### DISCLOSURE AGREEMENT

This section explains how personal health information collected about you for the study may be used. Your personal health information includes, but is not limited to, information that was collected for your entry into the study and information that is collected during the study. The purpose of collecting this information is to allow the study staff and the Investigator to conduct the study, to evaluate the sponsor's study products and to analyze the study results.

You may decide not to give permission for the release of your personal health information for the study. In that case, you will not be able to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the sponsor's study products.

People who may inspect your personal and health information includes the Investigator, the Institutional Review Board, IntegReview IRB, FDA and other regulatory authorities from the United States or other countries, the study sponsor and people that work with the sponsor which includes, monitoring committees, contract research organizations, and consultants who have contracts with the company to do the study and review the study results. These reviews are done to check on the quality of the study and also for other purposes allowed by law.

The results of the study may be published in a medical book or journal, or presented at meetings for educational purposes. Neither your name, nor any other personal health information that specifically identifies you, will be used in those materials or presentations.

You may ask the Investigator to see and copy your personal health information related to the study. You may also ask the Investigator to correct any study related information about you that is wrong. You may have to wait until the end of the study to see your study records, so that the study can be organized properly.

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the Investigator at the address below:

Thomas J. Stephens & Associates, Inc. 5050 Edison Ave., Suite 202 Colorado Springs, CO 80915

If you cancel your permission after you have started in the study, the study staff and the Investigator will stop collecting your personal health information. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the study.

Thomas J. Stephens & Associates and the sponsor will make every effort to keep your personal health information private. But after the study staff or the Investigator share your personal health information from the study, federal privacy laws may not keep it private. There might be laws in your state or other federal laws that would protect the privacy of this information.

#### **CONFIDENTIALITY**

Your records of being in this study will be kept private except when ordered by law. The following people will have access to your study records:

- The Investigator
- Sponsor company or research institution [including monitor(s) and auditor(s)]
- Other country, state or federal regulatory agencies
- IntegReview IRB

The Institutional Review Board (IRB), IntegReview, and accrediting agencies may inspect and copy your records, which may have your name on them. Therefore, total confidentiality cannot be guaranteed. If the study results are presented at meetings or printed in publications, your name will not be used.

#### IN CASE OF STUDY RELATED INJURY

Side effects or complications, both foreseeable and unforeseeable, are possible in any research study without any fault to you, the Investigator, the study site, or the study sponsor. If you get hurt or sick as a direct result of being in this study, the sponsor will pay the costs of reasonable medical treatment. To ask questions about this, talk to the Investigator or study staff.

The sponsor's policy does not offer compensation for other expenses. Be aware that your health care payer/insurer might not cover the costs of study-related injuries or illnesses.

Unreimbursed medical expenses not covered by insurance or other third party coverage will be reimbursed by the sponsor for medical treatment for any injury that, in the opinion of the study doctor and the sponsor, is directly caused by the investigational product or by procedures required by the study protocol which would not have been performed as part of your regular medical care.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### **LEGAL RIGHTS**

You will not lose any of your legal rights by signing this consent form.

#### **CONTACT INFORMATION**

If you have questions, concerns, or complaints about this study or to report a study related injury, contact:

Kun Qian, M.D. 719-637-2828 daytime telephone number 719-471-1763 after hours number

If you are unable to reach anyone at the number(s) listed above and you need medical attention, please go to the nearest emergency room.

If you do not want to talk to the Investigator or study staff, if you have concerns or complaints about the research, or to ask questions about your rights as a study subject you may contact IntegReview. IntegReview's policy indicates that all concerns/complaints are to be submitted in writing for review at a convened IRB meeting to:

| Mailing Address: | OR | Email Address: |
|----------------------------------|----|-----------------------------|
| Chairperson | | integreview@integreview.com |
| IntegReview IRB | | |
| 3815 S. Capital of Texas Highway | | |
| Suite 320 | | |
| Austin, TX 78704 | | |

If you are unable to provide your concerns/complaints in writing or if this is an emergency situation regarding subject safety, contact our office at:

512-326-3001 or toll free at 1-877-562-1589 between 8 a.m. and 5 p.m. Central Time

IntegReview has approved the information in this consent form and has given approval for the Investigator to do the study. This does not mean IntegReview has approved your being in the study. You must consider the information in this consent form for yourself and decide if you want to be in this study.

### PAYMENT FOR BEING IN THE STUDY

You may receive up to \$575.00 for being in the study. You will be paid per completed visit as follows:

| Visit | Compensation (amount) |
|---------|-----------------------|
| Visit 1 | \$40.00 |
| Visit 2 | \$60.00 |
| Visit 3 | \$65.00 |
| Visit 4 | \$75.00 |
| Visit 5 | \$90.00 |

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

| Visit 6 | \$95.00 |
|---------|----------|
| Visit 7 | \$150.00 |

If you choose to leave or are withdrawn from the study for any reason before finishing all visits you will be paid for each completed visit. You will receive payment within 2 weeks of final study visit.

If you do not qualify for any reason, you will be paid \$20.00, which will be mailed to you within 2 weeks of the baseline study visit.

If you are paid \$600.00 or more by Thomas J. Stephens & Associates, Inc. in a calendar year, those payments will be reported to the Internal Revenue Service via form 1099-MISC. As required by tax laws, if you withhold your social security number, Thomas J. Stephens & Associates, Inc. is required to withhold 28% of your payment for tax purposes. In this case a form 1099-MISC will be sent to you reporting your withholding.

#### **VOLUNTEERING TO BE IN THE STUDY**

It is your choice if you want to be in the study. No one can force you to be in the study. You may not want to be in this study or you may leave the study at any time without penalty or loss of benefits to which you are otherwise entitled.

The Investigator, the sponsor company, or IntegReview may take you out of the study without your permission, at any time, for the following reasons:

- If you do not follow the Investigator's instructions
- If we find out you should not be in the study
- If the study is stopped
- If it becomes harmful to your health

If you leave the study or if you are taken out of the study, you may be asked to return for a final visit to have some end of study evaluations or tests. If information generated from this study is published or presented, your identity will not be revealed. If you leave the study, no more information about you will be collected for this study. However, all of the information you gave us before you left the study will still be used.

### **NEW FINDINGS**

If there is new information or any significant new findings that could relate to your willingness to continue participation we will tell you. You can then decide if you still want to be in the study.

#### THE REASON FOR INSTITUTIONAL REVIEW BOARDS AND INFORMED CONSENT

#### What is a consent form?

The informed consent document contains information required by federal regulations. The informed consent document must be approved by an Institutional Review Board (IRB).

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### What is an Institutional Review Board (IRB)?

An Institutional Review Board (IRB) is a group of people that reviews research studies. The main goal of this review is to protect the rights and well being of the human subjects participating in research studies.

### IntegReview, the IRB for this study

IntegReview is an IRB whose board members provide IRB services across the United States, Canada, Japan and Latin America.

To meet requirements of the law, the IntegReview Boards currently include:

- Doctors
- Pharmacists
- Nurses
- Toxicologists (people who study the harmful effects of chemicals)
- Other specialists
- Others who do not have a background in science/medicine

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### AGREEMENT TO BE IN THE STUDY

This consent form contains important information to help you decide if you want to be in the study. If you have any questions that are not answered in this consent form, ask one of the study staff.

| Pleas | e answer YES or NO to the following questions: | |
|---|---|---|
| A. | Is this document in a language you understand? | |
| B. | Do you understand the information in this consent form? | |
| C. | . Have you been given enough time to ask questions and talk about the study? | |
| D. | Have all of your questions been answered to your satisfaction? | |
| E. | Do you think you received enough information about the study? | |
| F. | Do you volunteer to be in this study of your own free will and without being pressured by the Investigator or study staff? | |
| G. | Do you know that you can leave the study at any time without giving a reason and without affecting your health care? | |
| Н. | Do you know that your health records from this study may be reviewed by the sponsor company and by government authorities? | |
| I. | Do you know that you cannot be in another study while you are in this stud | y? |
| | IF YOU ANSWERED "NO" TO ANY OF THE ABOVE QUES OR YOU ARE UNABLE TO ANSWER ANY OF THE ABOVE QUES YOU SHOULD NOT SIGN THIS CONSENT FORM. | |
| Printe | ed Name of Adult Study Subject | |
| Signa | ture of Adult Study Subject | Date |
| Printe | ed Name of Person Explaining Consent Form | |
| Signa | ature of Person Explaining Consent Form | Date |
| You | will be given a signed and dated copy of this consent form to keep. | |

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### **Authorization and Release Form**

I hereby for good and valuable consideration grant to Thomas J. Stephens & Associates, the study sponsor and their respective affiliates, agencies, agents, employees, and assigns (collectively, "Authorized Entities"), the unrestricted, royalty free, irrevocable and perpetual right and permission to reproduce, distribute, broadcast and/or otherwise use for advertising and other commercial/noncommercial purposes: (i) my name, likeness, image, video, and any other biographical or personal information ("Personal Content"); and (ii) any statement or endorsement, or any portions thereof ("Testimonial(s)"), made by me relating to the study sponsor's products ("Products"), in any and all media now known or later developed, worldwide in perpetuity, without further compensation or approval by me.

I hereby assign to the Authorized Entities all of my world-wide right, title and interest, including my copyright interests and all renewals, reissues and extensions thereof, in and to the Personal Content and Testimonial(s), including without limitation, any photographic portraits, sound recordings and video performances of and/or by me in connection with the Personal Content and/or Testimonial(s).

I am at least 21 years of age, and competent to contract in my own name. I have read and understand this

| Authorization and Release. | | |
|---|---|---|
| Printed Name of Adult Study Subject | | |
| Signature of Adult Study Subject | | Date |
| Printed Name of Person Explaining Release Form | | |
| Signature of Person Explaining Release Form | | Date |
| Copy of consent form given to subject on | (date) by | (initials) |
| You will be given a signed and dated copy of this cor | isent form to keep | ı <b>.</b> |

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

# AUTHORIZATION TO USE AND DISCLOSE PERSONAL HEALTH INFORMATION FOR RESEARCH

THIS SECTION DESCRIBES YOUR RIGHTS AND HOW PERSONAL HEALTH INFORMATION COLLECTED ABOUT YOU DURING THIS STUDY MAY BE USED AND DISCLOSED AND HOW YOU CAN GET ACCESS TO THIS INFORMATION. PLEASE REVIEW IT CAREFULLY.

The United States government has issued a privacy rule to protect the privacy rights of patients. This rule was issued under a law called the Health Insurance Portability and Accountability Act of 1996 (HIPAA). The Privacy Rule is designed to protect the confidentiality of your personal health information. The document you are reading, called an "Authorization," describes your rights and explains how your health information will be used and disclosed (shared).

Federal law requires hospitals, researchers and health care providers to protect the privacy of information that identifies you and relates to your past, present and future physical and mental health or conditions.

All information collected during the study will be retained by the study doctor and the Study Sponsor, except as required by law. Information from this study will be given to the sponsor. "Sponsor" includes any persons or companies, which are contracted by the sponsor to have access to the research information during and after the study. The information will also be given to the U.S. Food and Drug Administration (FDA). Study records which identify you and the consent form signed by you will be inspected and/or copied for research or regulatory purposes by:

- Sponsor
- Agents for the sponsor
- The US Food and Drug Administration (FDA)
- Department of Health and Human Services (DHHS) agencies
- IntegReview IRB

Because of the need to release information to these parties, absolute confidentiality cannot be guaranteed. The results of this research study may be presented at meetings or in publications; however, your identity will not be disclosed in those presentations.

For purposes of study reporting, you will be identified by your initials and code numbers only. However, your name, date of birth, address, and phone number will be kept on record by the study doctor in case you need to be contacted in the future about this study.

After your personal health information is disclosed to the Study Sponsor, the results of the study may be reanalyzed at a later date and may be combined with the results of other studies. The Study Sponsor and people who work with the Study Sponsor may use the results of this study for other research purposes, including:

- Developing a better understanding of the disease;
- Improving the design of future actual use trials

After the study staff or the study doctor discloses your personal health information to others, it could be re-disclosed and no longer protected by federal privacy laws.

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you do not withdraw this Authorization in writing, it will remain in effect indefinitely. Your study doctor will keep this Authorization for at least 6 years. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the study doctor at the address below:

Thomas J. Stephens & Associates, Inc. 5050 Edison Ave., Suite 202 Colorado Springs, CO 80915

You have the right to see and get a copy of your records related to the study for as long as the study doctor has this information. However, by signing this Authorization you agree that you might not be able to review or receive some of your records related to the study until after the study has been completed.

If you cancel your permission after you have started in the study, the study staff and the study doctor will stop collecting your personal health information unless the information concerns an adverse event (a bad effect) related to the study. If an adverse event occurs, your entire medical record may be reviewed. All information that has already been collected for study purposes, and any new information about an adverse event related to the study, will be sent to the study sponsor. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the study doctor would not be able to collect the information needed to evaluate the study results.

If you withdraw from the study but do not withdraw your Authorization, new personal health information may be collected until this study ends.

You may decide not to give permission for the release of your personal health information for this study. In that case, you will not be able to participate. This is because the study staff and study doctor would not be able to collect the information needed to evaluate the study results.

At the completion of the study, you have the right to access your protected health information that is created during this research study that relates to your treatment or to payment, provided such information is not exempted under certain laws and regulations. To request this information, please contact the study doctor at the address listed above.

### **Your Right to Access Health Information**

Subject to certain exceptions prescribed by law, you have a right to request access to the health information that we hold about you and to request changes if your health information is incorrect or incomplete. Any request for access or corrections should be made to the principal doctor conducting this study.

Your records obtained while you are in this trial, as well as related health records, will remain strictly confidential at all times. However, these will need to be made available to others working on the Sponsor's behalf, the Independent Ethics Committee members and Medicines Regulatory Authorities.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

By signing the consent form you agree to this access for the current trial and any further research that may be done. However, the Sponsor will take steps to protect your personal information and will not include your name on any sponsor forms, reports, publications, or in any future disclosures. If you withdraw from the study, we will no longer collect your personal information, but we may need to continue to use information already collected.

Personal data which may be sensitive (e.g., date of birth) will be collected and processed, but only for research purposes in connection with this trial.

The trial data will be sent around the world, but you will not be referred to by name or identified in any report or publication nor could the data be traced back to you. Your data may be transferred to a country that does not have the same level of personal data protection as within the United States. However, The Sponsor maintains high standards of confidentiality and protection.

The Sponsor (who will control the use of the data) will take steps to ensure your personal data is protected.

By taking part in this trial you agree not to restrict the use of any data even if you withdraw from the trial and agree to the transfer of your personal data to other Sponsor companies and to Medicines Regulatory Authorities both within and outside of Europe.

| Printed Name of Adult Study Subject | |
|-------------------------------------|------|
| Signature of Adult Study Subject | Date |

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

# INFORMED CONSENT DOCUMENT AGREEMENT TO BE IN A RESEARCH STUDY

NAME OF TESTING COMPANY: Thomas J. Stephens & Associates, Inc.

NUMBER AND TITLE OF STUDY: C16-CD020 (GLI.04.SPR.US10354); "A Multi-

Center Clinical Trial to Evaluate the Efficacy of

Two Acne Treatments"

NAME OF PERSON IN CHARGE OF

THE RESEARCH STUDY

(STUDY DOCTOR/INVESTIGATOR): Kun Qian, M.D.

**TELEPHONE NUMBER(S), DAYTIME:** 719-637-2828 **AFTER HOURS:** 719-471-1763

#### INTRODUCTION

You are being invited to volunteer for a clinical research study. You must read and sign this form before you agree to take part in this study. This form will give you more information about this study. Please ask as many questions as you need to before you decide if you want to be in the study. You should not sign this form if you have any questions that have not been answered.

Thomas J. Stephens & Associates, Inc., a contract research organization, is being paid by the sponsor (the company paying for this study) to conduct this research study.

You must be honest with the Investigator about your health history or it may not be safe for you to be in this study.

#### PURPOSE OF THE STUDY

The purpose of this study is to evaluate the efficiency of 2 acne treatments for 24 weeks of use in adult men and women with mild to moderate facial acne, at least 5 inflammatory lesions, and at least 10 - 100 non-inflammatory lesions.

#### HOW LONG THE STUDY WILL LAST AND HOW MANY PEOPLE WILL BE IN THE STUDY

This study will last 24 weeks and have up to 8 visits. At least 100 subjects, men and women between the ages of 21-45, are expected to complete this study, with at least 50 subjects completed per cell.

#### TO BE IN THIS STUDY

#### You must:

- Be a man or woman age 21 to 45 years at the time of enrollment.
- Have mild to moderate acne on the face as determined by the Investigator or designee.
- Have at least 5 inflammatory lesions as determined by the Investigator or designee.
- Have 10 100 non-inflammatory lesions as determined by the Investigator or designee.
- Be willing to use the test products as instructed for 24 weeks.
- Be willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol.

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Be willing to provide written informed consent including photo release, Health Insurance Portability
  and Accountability Act (HIPAA), and be able to read, speak, write, understand English and be willing
  to share personal information and data, as verified by signing a written authorization at the screening.
- Be willing to withhold all facial treatments during the course of the study including botulinum toxin, injectable fillers, microdermabrasion, IPL, peels, facials, laser treatments and tightening treatments. Waxing and threading is allowed but not facial laser hair removal.
- Males must be regular shavers and willing to shave on the day of the study visits (prior to clinic visits).
- Women of child bearing potential must be willing to take a urine pregnancy test prior to study enrollment, at week 24, and when deemed appropriate by the Investigator and/or Sponsor.
- Individuals of child bearing potential must use an acceptable method of contraception throughout the study. Acceptable methods of birth control include:
  - Oral and other system contraceptives. Individuals must be on a stable use for 3 months prior to study enrollment. Individuals on oral contraceptives must not alter their use, including dose or regimen for the duration of the study
  - Double barrier
  - o Bilateral tubal ligation (tubes tied)
  - o Partner vasectomy
  - Abstinence
- Be willing to follow study requirements and report any changes in health status or medications, side effect symptoms, or reactions immediately.
- Be stable on any medication you are taking for at least 30 days

#### YOU CANNOT BE ON THE STUDY

### If you:

- Have been diagnosed with allergies to topical acne products.
- Have a condition and/or disease of the skin that the Investigator deems inappropriate for participation.
- Are a woman who is breastfeeding, pregnant, or planning to become pregnant during the study.
- Have pre-existing or dormant dermatologic conditions on the face (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, severe excoriations etc.) which in the opinion of the Investigator could interfere with the outcome of the study.
- Have a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.).
- Have an uncontrolled disease such as asthma, diabetes, hypertension, hyperthyroidism, or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc. at the Investigator's discretion.
- Are currently participating in another facial usage study or have participated in a clinical trial within 4 weeks prior to inclusion into the study.
- Have a history of skin cancer on the face within the past 5 years.
- Have any planned surgeries and/or invasive medical procedures during the course of the study.
- Have started hormone replacement therapies (HRT) or hormones for birth control less than 3 months
  prior to study entry or plan on starting, stopping, or changing doses of HRT or hormones for birth
  control during the study.

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Have facial sunburn or excessive tanned facial skin or are not willing to avoid daily sun exposure on the face and the use of tanning beds or sunless tanning products for the duration of the study.
- Have severe acne, acne conglobata, multiple nodules or cysts (more than 2).
- Are currently taking a natural or prescription testosterone blocker (e.g. saw palmetto, blask cohosh, chaste tree, chasteberry, spironolactone, drospirenone, progestins).
- Are currently on a testosterone booster or prescription testosterone (e.g. DHEA, tribulus, testosterone cypionate, testosterone enanthate, Sustanon, testosterone propionate, testosterone phenylpropriate, Omnadren etc.).
- Are currently taking or have taken within the last 30 days oral or topical prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin (Retin A, Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo.
- Have used oral isotretinoin (Accutane) within the past 6-months.
- Are routinely using (3x a week or more) topical over-the-counter (OTC) acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 14 days of the study entry.
- Are using or have used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study.
- Have excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations as determined by the Investigator or designee.

#### WHAT WILL HAPPEN DURING THE STUDY

### \*Visit 1: Screening (\* Visit 1 {Screening} AND Visit 2 {Baseline} may be combined into 1 Visit)

### You will:

- Be given an IRB-approved Informed Consent Form (ICF), to read and sign. You will be given enough time to read the informed consent, and ask questions about the study, and sign 2 copies of this consent form. (1 for clinic records, 1 for your records)
- Be given an eligibility and health questionnaire to complete, and assigned a screening number.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Will be screened by the Investigator or designee to see if you qualify for the study.
- If you do qualify for the study, you will:
  - o Take a urine pregnancy test (females of child-bearing potential)
  - Have a dermatologist confirm your eligibility
  - o Schedule your next appointment.

#### \*Visit 2: Baseline

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Be screened by the Investigator or designee to see if you still qualify for the study.
- Have your health and eligibility re-reviewed.
- If you still qualify for the study you will:
  - o Be assigned a subject number
  - Have photos taken of your face

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Be randomly assigned to receive one of the test products & supporting facial cleanser, moisturizer & facial SPF 30
- o Be provided verbal and written usage instructions, and a daily diary to record product use
- o Schedule your next appointment

#### **Visits 3, 4 (Week 1, Week 2)**

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and returned to you. At week 2, your diary
  will be retained by the testing facility and you will be given a new diary
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

### Visits 5, 6 (Week 6, Week 12)

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you
  will be given a new diary.
- Have your product collected, weighed, and retained. New products will be dispensed as necessary.
- Schedule your next appointment

#### Visit 7 (Week 18)

- Be asked if you have experienced any changes in your health since the previous visit.
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

### **Visit 8 (Week 24)**

- Be asked if you have experienced any changes in your health since the previous visit.
- Take a urine pregnancy test (females of child-bearing potential).
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility.
- Have your product collected, weighed, and retained by the testing facility.

Do not give the study product to other people and keep it out of the reach of children.

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### RISKS OR DISCOMFORTS

If you do not understand what any of these side effects mean, please ask the investigator or study staff to explain these terms to you.

Because the study products are investigational, all of their side effects may not be known. There may be rare and unknown side effects. Some of these may be life threatening.

Possible risks associated with the product are, as with any other cosmetic and OTC products, signs of irritation including:

- Itching
- Burning
- Stinging
- Rash or other allergic reaction

- Tingling
- Scaling/Dryness
- Redness

In some cases, it is possible for a subject to develop allergic reactions to the test material(s). This risk is increased for individuals with a history of allergies, and individuals with asthma and/or a history of hives may also be affected. Symptoms include rash, hives, and itching.

You must tell the Investigator or study staff about all side effects that you have. If you are not honest about your side effects, it may not be safe for you to stay in the study.

#### BIRTH CONTROL, DANGERS OF PREGNANCY AND BREASTFEEDING

If you are a female, you must not get pregnant while in this study. The only certain way to not get pregnant is to not have sex. If you are a female and choose to have sex, you must use a type of birth control.

Even if you use birth control during the study, there is a chance you could become pregnant. If you are pregnant or become pregnant during the study, test products or procedures may involve unforeseeable risks to the unborn baby.

A pregnancy test can be wrong. If you become pregnant during the study, stop using the test products and call/inform the Investigator at once.

You cannot be in the study if you are breastfeeding. It is not known whether the test products are safe for breast fed babies. Therefore if you are breastfeeding a child then it may not be safe for you to participate in the study.

#### POSSIBLE BENEFITS OF THE STUDY

You will not get any medical benefit from being in this study, and there is no promise that your condition (acne) will get better. It might stay the same or it might get worse. Your participation will provide information that may help others. There may be other marketed products that claim to have similar benefits.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### OTHER OPTIONS TO PARTICIPATING IN THE STUDY

Since this study is for research only, the only other choice would be not to be in the study.


To participate in this study, you must agree to keep any information relating to the design, identity or use of these test product samples confidential.

On rare occasions, the sponsor may allow the testing company to disclose to you the name of the test products if you are not given this information during the study. This information is typically not provided until the end of the study or after the test products have been released for sale to the public. The study doctor or study staff will notify you if the sponsor allows us to give you this information.

#### DISCLOSURE AGREEMENT

This section explains how personal health information collected about you for the study may be used. Your personal health information includes, but is not limited to, information that was collected for your entry into the study and information that is collected during the study. The purpose of collecting this information is to allow the study staff and the Investigator to conduct the study, to evaluate the sponsor's study products and to analyze the study results.

You may decide not to give permission for the release of your personal health information for the study. In that case, you will not be able to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the sponsor's study products.

People who may inspect your personal and health information includes the Investigator, the Institutional Review Board, IntegReview IRB, FDA and other regulatory authorities from the United States or other countries, the study sponsor and people that work with the sponsor which includes, monitoring committees, contract research organizations, and consultants who have contracts with the company to do the study and review the study results. These reviews are done to check on the quality of the study and also for other purposes allowed by law.

The results of the study may be published in a medical book or journal, or presented at meetings for educational purposes. Neither your name, nor any other personal health information that specifically identifies you, will be used in those materials or presentations.

You may ask the Investigator to see and copy your personal health information related to the study. You may also ask the Investigator to correct any study related information about you that is wrong. You may have to wait until the end of the study to see your study records, so that the study can be organized properly.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the Investigator at the address below:

Thomas J. Stephens & Associates, Inc. 5050 Edison Ave., Suite 202 Colorado Springs, CO 80915

If you cancel your permission after you have started in the study, the study staff and the Investigator will stop collecting your personal health information. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the study.

Thomas J. Stephens & Associates and the sponsor will make every effort to keep your personal health information private. But after the study staff or the Investigator share your personal health information from the study, federal privacy laws may not keep it private. There might be laws in your state or other federal laws that would protect the privacy of this information.

#### **CONFIDENTIALITY**

Your records of being in this study will be kept private except when ordered by law. The following people will have access to your study records:

- The Investigator
- Sponsor company or research institution [including monitor(s) and auditor(s)]
- Other country, state or federal regulatory agencies
- IntegReview IRB

The Institutional Review Board (IRB), IntegReview, and accrediting agencies may inspect and copy your records, which may have your name on them. Therefore, total confidentiality cannot be guaranteed. If the study results are presented at meetings or printed in publications, your name will not be used.

#### IN CASE OF STUDY RELATED INJURY

Side effects or complications, both foreseeable and unforeseeable, are possible in any research study without any fault to you, the Investigator, the study site, or the study sponsor. If you get hurt or sick as a direct result of being in this study, the sponsor will pay the costs of reasonable medical treatment. To ask questions about this, talk to the Investigator or study staff.

The sponsor's policy does not offer compensation for other expenses. Be aware that your health care payer/insurer might not cover the costs of study-related injuries or illnesses.

Unreimbursed medical expenses not covered by insurance or other third party coverage will be reimbursed by the sponsor for medical treatment for any injury that, in the opinion of the study doctor and the sponsor, is directly caused by the investigational product or by procedures required by the study protocol which would not have been performed as part of your regular medical care.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### **LEGAL RIGHTS**

You will not lose any of your legal rights by signing this consent form.

#### **CONTACT INFORMATION**

If you have questions, concerns, or complaints about this study or to report a study related injury, contact:

Kun Qian, M.D. 719-637-2828 daytime telephone number 719-471-1763 after hours number

If you are unable to reach anyone at the number(s) listed above and you need medical attention, please go to the nearest emergency room.

If you do not want to talk to the Investigator or study staff, if you have concerns or complaints about the research, or to ask questions about your rights as a study subject you may contact IntegReview. IntegReview's policy indicates that all concerns/complaints are to be submitted in writing for review at a convened IRB meeting to:

| Mailing Address: | OR | Email Address: |
|----------------------------------|----|-----------------------------|
| Chairperson | | integreview@integreview.com |
| IntegReview IRB | | |
| 3815 S. Capital of Texas Highway | | |
| Suite 320 | | |
| Austin, TX 78704 | | |

If you are unable to provide your concerns/complaints in writing or if this is an emergency situation regarding subject safety, contact our office at:

512-326-3001 or toll free at 1-877-562-1589 between 8 a.m. and 5 p.m. Central Time

IntegReview has approved the information in this consent form and has given approval for the Investigator to do the study. This does not mean IntegReview has approved your being in the study. You must consider the information in this consent form for yourself and decide if you want to be in this study.

### PAYMENT FOR BEING IN THE STUDY

You may receive up to \$575.00 for being in the study. You will be paid per completed visit as follows:

| Visit | Compensation (amount) |
|---------|-----------------------|
| Visit 1 | \$40.00 |
| Visit 2 | \$60.00 |
| Visit 3 | \$65.00 |
| Visit 4 | \$75.00 |
| Visit 5 | \$90.00 |

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

VERSION CONTROL

clw/master: 2-17-16 snb/site: 2-29-16 rss/master: 9-16-16

| Visit 6 | \$95.00 |
|---------|----------|
| Visit 7 | \$150.00 |

If you choose to leave or are withdrawn from the study for any reason before finishing all visits you will be paid for each completed visit. You will receive payment within 2 weeks of final study visit.

If you do not qualify for any reason, you will be paid \$20.00, which will be mailed to you within 2 weeks of the baseline study visit.

If you are paid \$600.00 or more by Thomas J. Stephens & Associates, Inc. in a calendar year, those payments will be reported to the Internal Revenue Service via form 1099-MISC. As required by tax laws, if you withhold your social security number, Thomas J. Stephens & Associates, Inc. is required to withhold 28% of your payment for tax purposes. In this case a form 1099-MISC will be sent to you reporting your withholding.

#### **VOLUNTEERING TO BE IN THE STUDY**

It is your choice if you want to be in the study. No one can force you to be in the study. You may not want to be in this study or you may leave the study at any time without penalty or loss of benefits to which you are otherwise entitled.

The Investigator, the sponsor company, or IntegReview may take you out of the study without your permission, at any time, for the following reasons:

- If you do not follow the Investigator's instructions
- If we find out you should not be in the study
- If the study is stopped
- If it becomes harmful to your health

If you leave the study or if you are taken out of the study, you may be asked to return for a final visit to have some end of study evaluations or tests. If information generated from this study is published or presented, your identity will not be revealed. If you leave the study, no more information about you will be collected for this study. However, all of the information you gave us before you left the study will still be used.

#### **NEW FINDINGS**

If there is new information or any significant new findings that could relate to your willingness to continue participation we will tell you. You can then decide if you still want to be in the study.

#### THE REASON FOR INSTITUTIONAL REVIEW BOARDS AND INFORMED CONSENT

#### What is a consent form?

The informed consent document contains information required by federal regulations. The informed consent document must be approved by an Institutional Review Board (IRB).

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### What is an Institutional Review Board (IRB)?

An Institutional Review Board (IRB) is a group of people that reviews research studies. The main goal of this review is to protect the rights and well being of the human subjects participating in research studies.

### IntegReview, the IRB for this study

IntegReview is an IRB whose board members provide IRB services across the United States, Canada, Japan and Latin America.

To meet requirements of the law, the IntegReview Boards currently include:

- Doctors
- Pharmacists
- Nurses
- Toxicologists (people who study the harmful effects of chemicals)
- Other specialists
- Others who do not have a background in science/medicine

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### AGREEMENT TO BE IN THE STUDY

This consent form contains important information to help you decide if you want to be in the study. If you have any questions that are not answered in this consent form, ask one of the study staff.

| Pleas | e answer YES or NO to the following questions: | |
|---|---|---|
| A. | Is this document in a language you understand? | |
| B. | Do you understand the information in this consent form? | |
| C. | Have you been given enough time to ask questions and talk about the study? | |
| D. | Have all of your questions been answered to your satisfaction? | |
| E. | Do you think you received enough information about the study? | |
| F. | Do you volunteer to be in this study of your own free will and without being pressured by the Investigator or study staff? | |
| G. | Do you know that you can leave the study at any time without giving a reason and without affecting your health care? | |
| Н. | Do you know that your health records from this study may be reviewed by the sponsor company and by government authorities? | |
| I. | Do you know that you cannot be in another study while you are in this study? | |
| | IF YOU ANSWERED "NO" TO ANY OF THE ABOVE QUESTIO OR YOU ARE UNABLE TO ANSWER ANY OF THE ABOVE QUES' YOU SHOULD NOT SIGN THIS CONSENT FORM. | |
| Print | ed Name of Adult Study Subject | |
| Signa | ture of Adult Study Subject | Date |
| Print | ed Name of Person Explaining Consent Form | |
| Signa | ature of Person Explaining Consent Form | Date |
| You | will be given a signed and dated copy of this consent form to keep. | |

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### **Authorization and Release Form**

I hereby for good and valuable consideration grant to Thomas J. Stephens & Associates, the study sponsor and their respective affiliates, agencies, agents, employees, and assigns (collectively, "Authorized Entities"), the unrestricted, royalty free, irrevocable and perpetual right and permission to reproduce, distribute, broadcast and/or otherwise use for advertising and other commercial/noncommercial purposes: (i) my name, likeness, image, video, and any other biographical or personal information ("Personal Content"); and (ii) any statement or endorsement, or any portions thereof ("Testimonial(s)"), made by me relating to the study sponsor's products ("Products"), in any and all media now known or later developed, worldwide in perpetuity, without further compensation or approval by me.

I hereby assign to the Authorized Entities all of my world-wide right, title and interest, including my copyright interests and all renewals, reissues and extensions thereof, in and to the Personal Content and Testimonial(s), including without limitation, any photographic portraits, sound recordings and video performances of and/or by me in connection with the Personal Content and/or Testimonial(s).

I am at least 21 years of age, and competent to contract in my own name. I have read and understand this

| Authorization and Release. | |
|---|---|
| Printed Name of Adult Study Subject | |
| Signature of Adult Study Subject | Date |
| Printed Name of Person Explaining Release Form | |
| Signature of Person Explaining Release Form | Date |
| Copy of consent form given to subject on (date) | by (initials) |
| You will be given a signed and dated copy of this consent form | to keep. |

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

# AUTHORIZATION TO USE AND DISCLOSE PERSONAL HEALTH INFORMATION FOR RESEARCH

THIS SECTION DESCRIBES YOUR RIGHTS AND HOW PERSONAL HEALTH INFORMATION COLLECTED ABOUT YOU DURING THIS STUDY MAY BE USED AND DISCLOSED AND HOW YOU CAN GET ACCESS TO THIS INFORMATION. PLEASE REVIEW IT CAREFULLY.

The United States government has issued a privacy rule to protect the privacy rights of patients. This rule was issued under a law called the Health Insurance Portability and Accountability Act of 1996 (HIPAA). The Privacy Rule is designed to protect the confidentiality of your personal health information. The document you are reading, called an "Authorization," describes your rights and explains how your health information will be used and disclosed (shared).

Federal law requires hospitals, researchers and health care providers to protect the privacy of information that identifies you and relates to your past, present and future physical and mental health or conditions.

All information collected during the study will be retained by the study doctor and the Study Sponsor, except as required by law. Information from this study will be given to the sponsor. "Sponsor" includes any persons or companies, which are contracted by the sponsor to have access to the research information during and after the study. The information will also be given to the U.S. Food and Drug Administration (FDA). Study records which identify you and the consent form signed by you will be inspected and/or copied for research or regulatory purposes by:

- Sponsor
- Agents for the sponsor
- The US Food and Drug Administration (FDA)
- Department of Health and Human Services (DHHS) agencies
- IntegReview IRB

Because of the need to release information to these parties, absolute confidentiality cannot be guaranteed. The results of this research study may be presented at meetings or in publications; however, your identity will not be disclosed in those presentations.

For purposes of study reporting, you will be identified by your initials and code numbers only. However, your name, date of birth, address, and phone number will be kept on record by the study doctor in case you need to be contacted in the future about this study.

After your personal health information is disclosed to the Study Sponsor, the results of the study may be reanalyzed at a later date and may be combined with the results of other studies. The Study Sponsor and people who work with the Study Sponsor may use the results of this study for other research purposes, including:

- Developing a better understanding of the disease;
- Improving the design of future actual use trials

After the study staff or the study doctor discloses your personal health information to others, it could be re-disclosed and no longer protected by federal privacy laws.

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you do not withdraw this Authorization in writing, it will remain in effect indefinitely. Your study doctor will keep this Authorization for at least 6 years. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the study doctor at the address below:

Thomas J. Stephens & Associates, Inc. 5050 Edison Ave., Suite 202 Colorado Springs, CO 80915

You have the right to see and get a copy of your records related to the study for as long as the study doctor has this information. However, by signing this Authorization you agree that you might not be able to review or receive some of your records related to the study until after the study has been completed.

If you cancel your permission after you have started in the study, the study staff and the study doctor will stop collecting your personal health information unless the information concerns an adverse event (a bad effect) related to the study. If an adverse event occurs, your entire medical record may be reviewed. All information that has already been collected for study purposes, and any new information about an adverse event related to the study, will be sent to the study sponsor. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the study doctor would not be able to collect the information needed to evaluate the study results.

If you withdraw from the study but do not withdraw your Authorization, new personal health information may be collected until this study ends.

You may decide not to give permission for the release of your personal health information for this study. In that case, you will not be able to participate. This is because the study staff and study doctor would not be able to collect the information needed to evaluate the study results.

At the completion of the study, you have the right to access your protected health information that is created during this research study that relates to your treatment or to payment, provided such information is not exempted under certain laws and regulations. To request this information, please contact the study doctor at the address listed above.

### **Your Right to Access Health Information**

Subject to certain exceptions prescribed by law, you have a right to request access to the health information that we hold about you and to request changes if your health information is incorrect or incomplete. Any request for access or corrections should be made to the principal doctor conducting this study.

Your records obtained while you are in this trial, as well as related health records, will remain strictly confidential at all times. However, these will need to be made available to others working on the Sponsor's behalf, the Independent Ethics Committee members and Medicines Regulatory Authorities.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

By signing the consent form you agree to this access for the current trial and any further research that may be done. However, the Sponsor will take steps to protect your personal information and will not include your name on any sponsor forms, reports, publications, or in any future disclosures. If you withdraw from the study, we will no longer collect your personal information, but we may need to continue to use information already collected.

Personal data which may be sensitive (e.g., date of birth) will be collected and processed, but only for research purposes in connection with this trial.

The trial data will be sent around the world, but you will not be referred to by name or identified in any report or publication nor could the data be traced back to you. Your data may be transferred to a country that does not have the same level of personal data protection as within the United States. However, The Sponsor maintains high standards of confidentiality and protection.

The Sponsor (who will control the use of the data) will take steps to ensure your personal data is protected.

By taking part in this trial you agree not to restrict the use of any data even if you withdraw from the trial and agree to the transfer of your personal data to other Sponsor companies and to Medicines Regulatory Authorities both within and outside of Europe.

| Printed Name of Adult Study Subject | |
|-------------------------------------|------|
| Signature of Adult Study Subject | Date |

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

### INFORMED CONSENT DOCUMENT AGREEMENT TO BE IN A RESEARCH STUDY

**NAME OF TESTING COMPANY:** Thomas J. Stephens & Associates, Inc.

NUMBER AND TITLE OF STUDY: C16-CD020 (GLI.04.SPR.US10354); "A Multi-

Center Clinical Trial to Evaluate the Efficacy of

Two Acne Treatments"

NAME OF PERSON IN CHARGE OF

THE RESEARCH STUDY

(STUDY DOCTOR/INVESTIGATOR): Edward Lain, MD

**TELEPHONE NUMBER(S), DAYTIME:** 512-279-2545 **AFTER HOURS:** 512-844-4500

#### INTRODUCTION

You are being invited to volunteer for a clinical research study. You must read and sign this form before you agree to take part in this study. This form will give you more information about this study. Please ask as many questions as you need to before you decide if you want to be in the study. You should not sign this form if you have any questions that have not been answered.

Thomas J. Stephens & Associates, Inc., a contract research organization, is being paid by the sponsor (the company paying for this study) to conduct this research study.

You must be honest with the Investigator about your health history or it may not be safe for you to be in this study.

#### PURPOSE OF THE STUDY

The purpose of this study is to evaluate the efficiency of 2 acne treatments for 24 weeks of use in adult men and women with mild to moderate facial acne, at least 5 inflammatory lesions, and at least 10 - 100 non-inflammatory lesions.

### HOW LONG THE STUDY WILL LAST AND HOW MANY PEOPLE WILL BE IN THE STUDY

This study will last 24 weeks and have up to 8 visits. At least 100 subjects, men and women between the ages of 21-45, are expected to complete this study, with at least 50 subjects completed per cell. Each site is to enroll no more than 40 subjects, with at least 100 subjects expected to complete when combined.

#### TO BE IN THIS STUDY

#### You must:

- Be a man or woman age 21 to 45 years at the time of enrollment.
- Have mild to moderate acne on the face as determined by the Investigator or designee.
- Have at least 5 inflammatory lesions as determined by the Investigator or designee.
- Have 10 100 non-inflammatory lesions as determined by the Investigator or designee.
- Be willing to use the test products as instructed for 24 weeks.

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Be willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol.
- Be willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and be able to read, speak, write, understand English and be willing to share personal information and data, as verified by signing a written authorization at the screening.
- Be willing to withhold all facial treatments during the course of the study including botulinum toxin, injectable fillers, microdermabrasion, IPL, peels, facials, laser treatments and tightening treatments. Waxing and threading is allowed but not facial laser hair removal.
- Males must be regular shavers and willing to shave on the day of the study visits (prior to clinic visits).
- Women of child bearing potential must be willing to take a urine pregnancy test prior to study enrollment, at week 24, and when deemed appropriate by the Investigator and/or Sponsor.
- Individuals of child bearing potential must use an acceptable method of contraception throughout the study. Acceptable methods of birth control include:
  - Oral and other system contraceptives. Individuals must be on a stable use for 3 months prior to study enrollment. Individuals on oral contraceptives must not alter their use, including dose or regimen for the duration of the study
  - Double barrier
  - Bilateral tubal ligation (tubes tied)
  - Partner vasectomy
  - Abstinence
- Be willing to follow study requirements and report any changes in health status or medications, side effect symptoms, or reactions immediately.
- Be stable on any medication you are taking for at least 30 days

#### YOU CANNOT BE ON THE STUDY

#### If you:

- Have been diagnosed with allergies to topical acne products.
- Have a condition and/or disease of the skin that the Investigator deems inappropriate for participation.
- Are a woman who is breastfeeding, pregnant, or planning to become pregnant during the study.
- Have pre-existing or dormant dermatologic conditions on the face (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, severe excoriations etc.) which in the opinion of the Investigator could interfere with the outcome of the study.
- Have a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.).
- Have an uncontrolled disease such as asthma, diabetes, hypertension, hyperthyroidism, or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc. at the Investigator's discretion.
- Are currently participating in another facial usage study or have participated in a clinical trial within 4 weeks prior to inclusion into the study.
- Have a history of skin cancer on the face within the past 5 years.
- Have any planned surgeries and/or invasive medical procedures during the course of the study.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Have started hormone replacement therapies (HRT) or hormones for birth control less than 3 months
  prior to study entry or plan on starting, stopping, or changing doses of HRT or hormones for birth
  control during the study.
- Have facial sunburn or excessive tanned facial skin or are not willing to avoid daily sun exposure on the face and the use of tanning beds or sunless tanning products for the duration of the study.
- Have severe acne, acne conglobata, multiple nodules or cysts (more than 2).
- Are currently taking a natural or prescription testosterone blocker (e.g. saw palmetto, blask cohosh, chaste tree, chasteberry, spironolactone, drospirenone, progestins).
- Are currently on a testosterone booster or prescription testosterone (e.g. DHEA, tribulus, testosterone cypionate, testosterone enanthate, Sustanon, testosterone propionate, testosterone phenylpropriate, Omnadren etc.).
- Are currently taking or have taken within the last 30 days oral or topical prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin (Retin A, Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo.
- Have used oral isotretinoin (Accutane) within the past 6-months.
- Are routinely using (3x a week or more) topical over-the-counter (OTC) acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 14 days of the study entry.
- Are using or have used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study.
- Have excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations as determined by the Investigator or designee.

#### WHAT WILL HAPPEN DURING THE STUDY

#### \*Visit 1: Screening (\* Visit 1 {Screening} AND Visit 2 {Baseline} may be combined into 1 Visit)

#### You will:

- Be given an IRB-approved Informed Consent Form (ICF), to read and sign. You will be given enough time to read the informed consent, and ask questions about the study, and sign 2 copies of this consent form. (1 for clinic records, 1 for your records)
- Be given an eligibility and health questionnaire to complete, and assigned a screening number.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Will be screened by the Investigator or designee to see if you qualify for the study.
- If you do qualify for the study, you will:
  - Take a urine pregnancy test (females of child-bearing potential)
  - o Have a dermatologist confirm your eligibility
  - Schedule your next appointment.

#### \*Visit 2: Baseline

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Be screened by the Investigator or designee to see if you still qualify for the study.
- Have your health and eligibility re-reviewed.

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- If you still qualify for the study you will:
  - o Be assigned a subject number
  - o Have photos taken of your face
  - o Be randomly assigned to receive one of the test products & supporting facial cleanser, moisturizer & facial SPF 30
  - o Be provided verbal and written usage instructions, and a daily diary to record product use
  - Schedule your next appointment

### **Visits 3, 4 (Week 1, Week 2)**

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and returned to you. At week 2, your diary will be retained by the testing facility and you will be given a new diary
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

### Visits 5, 6 (Week 6, Week 12)

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and retained. New products will be dispensed as necessary.
- Schedule your next appointment

### <u>Visit 7</u> (Week 18)

- Be asked if you have experienced any changes in your health since the previous visit.
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

### Visit 8 (Week 24)

- Be asked if you have experienced any changes in your health since the previous visit.
- Take a urine pregnancy test (females of child-bearing potential).
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility.
- Have your product collected, weighed, and retained by the testing facility.

Do not give the study product to other people and keep it out of the reach of children.

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### RISKS OR DISCOMFORTS

If you do not understand what any of these side effects mean, please ask the investigator or study staff to explain these terms to you.

Because the study products are investigational, all of their side effects may not be known. There may be rare and unknown side effects. Some of these may be life threatening.

Possible risks associated with the product are, as with any other cosmetic and OTC products, signs of irritation including:

- Itching
- Burning
- Stinging
- Rash or other allergic reaction

- Tingling
- Scaling/Dryness
- Redness

In some cases, it is possible for a subject to develop allergic reactions to the test material(s). This risk is increased for individuals with a history of allergies, and individuals with asthma and/or a history of hives may also be affected. Symptoms include rash, hives, and itching.

You must tell the Investigator or study staff about all side effects that you have. If you are not honest about your side effects, it may not be safe for you to stay in the study.

#### BIRTH CONTROL, DANGERS OF PREGNANCY AND BREASTFEEDING

If you are a female, you must not get pregnant while in this study. The only certain way to not get pregnant is to not have sex. If you are a female and choose to have sex, you must use a type of birth control.

Even if you use birth control during the study, there is a chance you could become pregnant. If you are pregnant or become pregnant during the study, test products or procedures may involve unforeseeable risks to the unborn baby.

A pregnancy test can be wrong. If you become pregnant during the study, stop using the test products and call/inform the Investigator at once.

You cannot be in the study if you are breastfeeding. It is not known whether the test products are safe for breast fed babies. Therefore if you are breastfeeding a child then it may not be safe for you to participate in the study.

#### POSSIBLE BENEFITS OF THE STUDY

You will not get any medical benefit from being in this study, and there is no promise that your condition (acne) will get better. It might stay the same or it might get worse. Your participation will provide information that may help others. There may be other marketed products that claim to have similar benefits.

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### OTHER OPTIONS TO PARTICIPATING IN THE STUDY

Since this study is for research only, the only other choice would be not to be in the study.


To participate in this study, you must agree to keep any information relating to the design, identity or use of these test product samples confidential.

On rare occasions, the sponsor may allow the testing company to disclose to you the name of the test products if you are not given this information during the study. This information is typically not provided until the end of the study or after the test products have been released for sale to the public. The study doctor or study staff will notify you if the sponsor allows us to give you this information.

#### DISCLOSURE AGREEMENT

This section explains how personal health information collected about you for the study may be used. Your personal health information includes, but is not limited to, information that was collected for your entry into the study and information that is collected during the study. The purpose of collecting this information is to allow the study staff and the Investigator to conduct the study, to evaluate the sponsor's study products and to analyze the study results.

You may decide not to give permission for the release of your personal health information for the study. In that case, you will not be able to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the sponsor's study products.

People who may inspect your personal and health information includes the Investigator, the Institutional Review Board, IntegReview IRB, FDA and other regulatory authorities from the United States or other countries, the study sponsor and people that work with the sponsor which includes, monitoring committees, contract research organizations, and consultants who have contracts with the company to do the study and review the study results. These reviews are done to check on the quality of the study and also for other purposes allowed by law.

The results of the study may be published in a medical book or journal, or presented at meetings for educational purposes. Neither your name, nor any other personal health information that specifically identifies you, will be used in those materials or presentations.

You may ask the Investigator to see and copy your personal health information related to the study. You may also ask the Investigator to correct any study related information about you that is wrong. You may have to wait until the end of the study to see your study records, so that the study can be organized properly.

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the Investigator at the address below:

Austin Institute for Clinical Research, Inc. 302 N. Heatherwilde Blvd., Suite 300 Pflugerville, TX 78660

If you cancel your permission after you have started in the study, the study staff and the Investigator will stop collecting your personal health information. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the study.

Thomas J. Stephens & Associates and the sponsor will make every effort to keep your personal health information private. But after the study staff or the Investigator share your personal health information from the study, federal privacy laws may not keep it private. There might be laws in your state or other federal laws that would protect the privacy of this information.

#### **CONFIDENTIALITY**

Your records of being in this study will be kept private except when ordered by law. The following people will have access to your study records:

- The Investigator
- Sponsor company or research institution [including monitor(s) and auditor(s)]
- Other country, state or federal regulatory agencies
- IntegReview IRB

The Institutional Review Board (IRB), IntegReview, and accrediting agencies may inspect and copy your records, which may have your name on them. Therefore, total confidentiality cannot be guaranteed. If the study results are presented at meetings or printed in publications, your name will not be used.

#### IN CASE OF STUDY RELATED INJURY

Side effects or complications, both foreseeable and unforeseeable, are possible in any research study without any fault to you, the Investigator, the study site, or the study sponsor. If you get hurt or sick as a direct result of being in this study, the sponsor will pay the costs of reasonable medical treatment. To ask questions about this, talk to the Investigator or study staff.

The sponsor's policy does not offer compensation for other expenses. Be aware that your health care payer/insurer might not cover the costs of study-related injuries or illnesses.

Unreimbursed medical expenses not covered by insurance or other third party coverage will be reimbursed by the sponsor for medical treatment for any injury that, in the opinion of the study doctor and the sponsor, is directly caused by the investigational product or by procedures required by the study protocol which would not have been performed as part of your regular medical care.

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### **LEGAL RIGHTS**

You will not lose any of your legal rights by signing this consent form.

#### **CONTACT INFORMATION**

If you have questions, concerns, or complaints about this study or to report a study related injury, contact:

Edward Lain, MD 512-279-2545 daytime telephone number 512-844-4500 after hours number

If you are unable to reach anyone at the number(s) listed above and you need medical attention, please go to the nearest emergency room.

If you do not want to talk to the Investigator or study staff, if you have concerns or complaints about the research, or to ask questions about your rights as a study subject you may contact IntegReview. IntegReview's policy indicates that all concerns/complaints are to be submitted in writing for review at a convened IRB meeting to:

| Mailing Address: | OR | Email Address: |
|----------------------------------|----|-----------------------------|
| Chairperson | | integreview@integreview.com |
| IntegReview IRB | | |
| 3815 S. Capital of Texas Highway | | |
| Suite 320 | | |
| Austin, TX 78704 | | |

If you are unable to provide your concerns/complaints in writing or if this is an emergency situation regarding subject safety, contact our office at:

512-326-3001 or toll free at 1-877-562-1589 between 8 a.m. and 5 p.m. Central Time

IntegReview has approved the information in this consent form and has given approval for the Investigator to do the study. This does not mean IntegReview has approved your being in the study. You must consider the information in this consent form for yourself and decide if you want to be in this study.

### PAYMENT FOR BEING IN THE STUDY

You may receive up to \$575.00 for being in the study. You will be paid per completed visit as follows:

| Visit | Compensation (amount) |
|---------------------------------|-----------------------|
| Screening/Baseline (Visit 1, 2) | \$40.00 |
| Visit 3 | \$60.00 |
| Visit 4 | \$65.00 |
| Visit 5 | \$75.00 |
| Visit 6 | \$90.00 |

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

VERSION CONTROL

clw/master: 2-17-16 snb/site: 2-25-16

| Visit 7 | \$95.00 |
|---------|----------|
| Visit 8 | \$150.00 |

If you choose to leave or are withdrawn from the study for any reason before finishing all visits you will be paid for each completed visit. You will receive payment at the end of each study visit.

If you do not qualify for any reason, you will be paid \$20.00, which will be mailed to you within 2 weeks of the baseline study visit.

If you are paid \$600.00 or more by Thomas J. Stephens & Associates, Inc. in a calendar year, those payments will be reported to the Internal Revenue Service via form 1099-MISC. As required by tax laws, if you withhold your social security number, Thomas J. Stephens & Associates, Inc. is required to withhold 28% of your payment for tax purposes. In this case a form 1099-MISC will be sent to you reporting your withholding.

#### **VOLUNTEERING TO BE IN THE STUDY**

It is your choice if you want to be in the study. No one can force you to be in the study. You may not want to be in this study or you may leave the study at any time without penalty or loss of benefits to which you are otherwise entitled.

The Investigator, the sponsor company, or IntegReview may take you out of the study without your permission, at any time, for the following reasons:

- If you do not follow the Investigator's instructions
- If we find out you should not be in the study
- If the study is stopped
- If it becomes harmful to your health

If you leave the study or if you are taken out of the study, you may be asked to return for a final visit to have some end of study evaluations or tests. If information generated from this study is published or presented, your identity will not be revealed. If you leave the study, no more information about you will be collected for this study. However, all of the information you gave us before you left the study will still be used.

#### **NEW FINDINGS**

If there is new information or any significant new findings that could relate to your willingness to continue participation we will tell you. You can then decide if you still want to be in the study.

#### THE REASON FOR INSTITUTIONAL REVIEW BOARDS AND INFORMED CONSENT

#### What is a consent form?

The informed consent document contains information required by federal regulations. The informed consent document must be approved by an Institutional Review Board (IRB).

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### What is an Institutional Review Board (IRB)?

An Institutional Review Board (IRB) is a group of people that reviews research studies. The main goal of this review is to protect the rights and well being of the human subjects participating in research studies.

### IntegReview, the IRB for this study

IntegReview is an IRB whose board members provide IRB services across the United States, Canada, Japan and Latin America.

To meet requirements of the law, the IntegReview Boards currently include:

- Doctors
- Pharmacists
- Nurses
- Toxicologists (people who study the harmful effects of chemicals)
- Other specialists
- Others who do not have a background in science/medicine

THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### AGREEMENT TO BE IN THE STUDY

This consent form contains important information to help you decide if you want to be in the study. If you have any questions that are not answered in this consent form, ask one of the study staff.

| Please | answer YES or NO to the following questions: | |
|---|---|---|
| A. | Is this document in a language you understand? | |
| B. | Do you understand the information in this consent form? | |
| C. | Have you been given enough time to ask questions and talk about the study? | |
| D. | Have all of your questions been answered to your satisfaction? | |
| E. | Do you think you received enough information about the study? | |
| F. | Do you volunteer to be in this study of your own free will and without being pressured by the Investigator or study staff? | |
| G. | Do you know that you can leave the study at any time without giving a reason and without affecting your health care? | |
| Н. | Do you know that your health records from this study may be reviewed by the sponsor company and by government authorities? | |
| I. | Do you know that you cannot be in another study while you are in this study? | |
| | IF YOU ANSWERED "NO" TO ANY OF THE ABOVE QUESTION OR YOU ARE UNABLE TO ANSWER ANY OF THE ABOVE QUESTI YOU SHOULD NOT SIGN THIS CONSENT FORM. | |
| Printe | d Name of Adult Study Subject | |
| Signat | ure of Adult Study Subject | Date |
| Printe | d Name of Person Explaining Consent Form | |
| Signat | ure of Person Explaining Consent Form | Date |
| You w | rill be given a signed and dated copy of this consent form to keep. | |

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE
## **Authorization and Release Form**

I hereby for good and valuable consideration grant to Thomas J. Stephens & Associates, the study sponsor and their respective affiliates, agencies, agents, employees, and assigns (collectively, "Authorized Entities"), the unrestricted, royalty free, irrevocable and perpetual right and permission to reproduce, distribute, broadcast and/or otherwise use for advertising and other commercial/noncommercial purposes: (i) my name, likeness, image, video, and any other biographical or personal information ("Personal Content"); and (ii) any statement or endorsement, or any portions thereof ("Testimonial(s)"), made by me relating to the study sponsor's products ("Products"), in any and all media now known or later developed, worldwide in perpetuity, without further compensation or approval by me.

I hereby assign to the Authorized Entities all of my world-wide right, title and interest, including my copyright interests and all renewals, reissues and extensions thereof, in and to the Personal Content and Testimonial(s), including without limitation, any photographic portraits, sound recordings and video performances of and/or by me in connection with the Personal Content and/or Testimonial(s).

I am at least 21 years of age, and competent to contract in my own name. I have read and understand this

| Authorization and Release. | | |
|---|---|---|
| Printed Name of Adult Study Subject | | |
| Signature of Adult Study Subject | | Date |
| Printed Name of Person Explaining Release Form | | |
| Signature of Person Explaining Release Form | | Date |
| Copy of consent form given to subject on | (date) by | (initials) |
| You will be given a signed and dated copy of this co | nsent form to keep. | |

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

# AUTHORIZATION TO USE AND DISCLOSE PERSONAL HEALTH INFORMATION FOR RESEARCH

THIS SECTION DESCRIBES YOUR RIGHTS AND HOW PERSONAL HEALTH INFORMATION COLLECTED ABOUT YOU DURING THIS STUDY MAY BE USED AND DISCLOSED AND HOW YOU CAN GET ACCESS TO THIS INFORMATION. PLEASE REVIEW IT CAREFULLY.

The United States government has issued a privacy rule to protect the privacy rights of patients. This rule was issued under a law called the Health Insurance Portability and Accountability Act of 1996 (HIPAA). The Privacy Rule is designed to protect the confidentiality of your personal health information. The document you are reading, called an "Authorization," describes your rights and explains how your health information will be used and disclosed (shared).

Federal law requires hospitals, researchers and health care providers to protect the privacy of information that identifies you and relates to your past, present and future physical and mental health or conditions.

All information collected during the study will be retained by the study doctor and the Study Sponsor, except as required by law. Information from this study will be given to the sponsor. "Sponsor" includes any persons or companies, which are contracted by the sponsor to have access to the research information during and after the study. The information will also be given to the U.S. Food and Drug Administration (FDA). Study records which identify you and the consent form signed by you will be inspected and/or copied for research or regulatory purposes by:

- Sponsor
- Agents for the sponsor
- The US Food and Drug Administration (FDA)
- Department of Health and Human Services (DHHS) agencies
- IntegReview IRB

Because of the need to release information to these parties, absolute confidentiality cannot be guaranteed. The results of this research study may be presented at meetings or in publications; however, your identity will not be disclosed in those presentations.

For purposes of study reporting, you will be identified by your initials and code numbers only. However, your name, date of birth, address, and phone number will be kept on record by the study doctor in case you need to be contacted in the future about this study.

After your personal health information is disclosed to the Study Sponsor, the results of the study may be reanalyzed at a later date and may be combined with the results of other studies. The Study Sponsor and people who work with the Study Sponsor may use the results of this study for other research purposes, including:

- Developing a better understanding of the disease;
- Improving the design of future actual use trials

After the study staff or the study doctor discloses your personal health information to others, it could be re-disclosed and no longer protected by federal privacy laws.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you do not withdraw this Authorization in writing, it will remain in effect indefinitely. Your study doctor will keep this Authorization for at least 6 years. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the study doctor at the address below:

Austin Institute for Clinical Research, Inc. 302 N. Heatherwilde Blvd., Suite 300 Pflugerville, TX 78660

You have the right to see and get a copy of your records related to the study for as long as the study doctor has this information. However, by signing this Authorization you agree that you might not be able to review or receive some of your records related to the study until after the study has been completed.

If you cancel your permission after you have started in the study, the study staff and the study doctor will stop collecting your personal health information unless the information concerns an adverse event (a bad effect) related to the study. If an adverse event occurs, your entire medical record may be reviewed. All information that has already been collected for study purposes, and any new information about an adverse event related to the study, will be sent to the study sponsor. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the study doctor would not be able to collect the information needed to evaluate the study results.

If you withdraw from the study but do not withdraw your Authorization, new personal health information may be collected until this study ends.

You may decide not to give permission for the release of your personal health information for this study. In that case, you will not be able to participate. This is because the study staff and study doctor would not be able to collect the information needed to evaluate the study results.

At the completion of the study, you have the right to access your protected health information that is created during this research study that relates to your treatment or to payment, provided such information is not exempted under certain laws and regulations. To request this information, please contact the study doctor at the address listed above.

# **Your Right to Access Health Information**

Subject to certain exceptions prescribed by law, you have a right to request access to the health information that we hold about you and to request changes if your health information is incorrect or incomplete. Any request for access or corrections should be made to the principal doctor conducting this study.

Your records obtained while you are in this trial, as well as related health records, will remain strictly confidential at all times. However, these will need to be made available to others working on the Sponsor's behalf, the Independent Ethics Committee members and Medicines Regulatory Authorities.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

By signing the consent form you agree to this access for the current trial and any further research that may be done. However, the Sponsor will take steps to protect your personal information and will not include your name on any sponsor forms, reports, publications, or in any future disclosures. If you withdraw from the study, we will no longer collect your personal information, but we may need to continue to use information already collected.

Personal data which may be sensitive (e.g., date of birth) will be collected and processed, but only for research purposes in connection with this trial.

The trial data will be sent around the world, but you will not be referred to by name or identified in any report or publication nor could the data be traced back to you. Your data may be transferred to a country that does not have the same level of personal data protection as within the United States. However, The Sponsor maintains high standards of confidentiality and protection.

The Sponsor (who will control the use of the data) will take steps to ensure your personal data is protected.

By taking part in this trial you agree not to restrict the use of any data even if you withdraw from the trial and agree to the transfer of your personal data to other Sponsor companies and to Medicines Regulatory Authorities both within and outside of Europe.

| _ |
|------|
| Date |

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

# INFORMED CONSENT DOCUMENT AGREEMENT TO BE IN A RESEARCH STUDY

**NAME OF TESTING COMPANY:** Austin Institute for Clinical Research, Inc.

NUMBER AND TITLE OF STUDY: C16-CD020 (GLI.04.SPR.US10354); "A Multi-

Center Clinical Trial to Evaluate the Efficacy of

Two Acne Treatments"

NAME OF PERSON IN CHARGE OF

THE RESEARCH STUDY

(STUDY DOCTOR/INVESTIGATOR): Edward Lain, MD

**TELEPHONE NUMBER(S), DAYTIME:** 512-279-2545 **AFTER HOURS:** 512-844-4500

#### INTRODUCTION

You are being invited to volunteer for a clinical research study. You must read and sign this form before you agree to take part in this study. This form will give you more information about this study. Please ask as many questions as you need to before you decide if you want to be in the study. You should not sign this form if you have any questions that have not been answered.

Austin Institute for Clinical Research, Inc. is being paid by the sponsor (the company paying for this study) to conduct this research study.

You must be honest with the Investigator about your health history or it may not be safe for you to be in this study.

#### PURPOSE OF THE STUDY

The purpose of this study is to evaluate the efficiency of 2 acne treatments for 24 weeks of use in adult men and women with mild to moderate facial acne, at least 5 inflammatory lesions, and at least 10 - 100 non-inflammatory lesions.

#### HOW LONG THE STUDY WILL LAST AND HOW MANY PEOPLE WILL BE IN THE STUDY

This study will last 24 weeks and have up to 8 visits. At least 100 subjects, men and women between the ages of 21-45, are expected to complete this study, with at least 50 subjects completed per cell. Each site is to enroll no more than 40 subjects, with at least 100 subjects expected to complete when combined.

#### TO BE IN THIS STUDY

#### You must:

- Be a man or woman age 21 to 45 years at the time of enrollment.
- Have mild to moderate acne on the face as determined by the Investigator or designee.
- Have at least 5 inflammatory lesions as determined by the Investigator or designee.
- Have 10 100 non-inflammatory lesions as determined by the Investigator or designee.
- Be willing to use the test products as instructed for 24 weeks.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Be willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol.
- Be willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and be able to read, speak, write, understand English and be willing to share personal information and data, as verified by signing a written authorization at the screening.
- Be willing to withhold all facial treatments during the course of the study including botulinum toxin, injectable fillers, microdermabrasion, IPL, peels, facials, laser treatments and tightening treatments. Waxing and threading is allowed but not facial laser hair removal.
- Males must be regular shavers and willing to shave on the day of the study visits (prior to clinic visits).
- Women of child bearing potential must be willing to take a urine pregnancy test prior to study enrollment, at week 24, and when deemed appropriate by the Investigator and/or Sponsor.
- Individuals of child bearing potential must use an acceptable method of contraception throughout the study. Acceptable methods of birth control include:
  - Oral and other system contraceptives. Individuals must be on a stable use for 3 months prior to study enrollment. Individuals on oral contraceptives must not alter their use, including dose or regimen for the duration of the study
  - Double barrier
  - o Bilateral tubal ligation (tubes tied)
  - Partner vasectomy
  - Abstinence
- Be willing to follow study requirements and report any changes in health status or medications, side effect symptoms, or reactions immediately.
- Be stable on any medication you are taking for at least 30 days

#### YOU CANNOT BE ON THE STUDY

## If you:

- Have been diagnosed with allergies to topical acne products.
- Have a condition and/or disease of the skin that the Investigator deems inappropriate for participation.
- Are a woman who is breastfeeding, pregnant, or planning to become pregnant during the study.
- Have pre-existing or dormant dermatologic conditions on the face (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, severe excoriations etc.) which in the opinion of the Investigator could interfere with the outcome of the study.
- Have a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.).
- Have an uncontrolled disease such as asthma, diabetes, hypertension, hyperthyroidism, or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc. at the Investigator's discretion.
- Are currently participating in another facial usage study or have participated in a clinical trial within 4 weeks prior to inclusion into the study.
- Have a history of skin cancer on the face within the past 5 years.
- Have any planned surgeries and/or invasive medical procedures during the course of the study.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Have started hormone replacement therapies (HRT) or hormones for birth control less than 3 months
  prior to study entry or plan on starting, stopping, or changing doses of HRT or hormones for birth
  control during the study.
- Have facial sunburn or excessive tanned facial skin or are not willing to avoid daily sun exposure on the face and the use of tanning beds or sunless tanning products for the duration of the study.
- Have severe acne, acne conglobata, multiple nodules or cysts (more than 2).
- Are currently taking a natural or prescription testosterone blocker (e.g. saw palmetto, blask cohosh, chaste tree, chasteberry, spironolactone, drospirenone, progestins).
- Are currently on a testosterone booster or prescription testosterone (e.g. DHEA, tribulus, testosterone cypionate, testosterone enanthate, Sustanon, testosterone propionate, testosterone phenylpropriate, Omnadren etc.).
- Are currently taking or have taken within the last 30 days oral or topical prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin (Retin A, Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo.
- Have used oral isotretinoin (Accutane) within the past 6-months.
- Are routinely using (3x a week or more) topical over-the-counter (OTC) acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 14 days of the study entry.
- Are using or have used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study.
- Have excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations as determined by the Investigator or designee.

#### WHAT WILL HAPPEN DURING THE STUDY

## \*Visit 1: Screening (\* Visit 1 {Screening} AND Visit 2 {Baseline} may be combined into 1 Visit)

#### You will:

- Be given an IRB-approved Informed Consent Form (ICF), to read and sign. You will be given enough time to read the informed consent, and ask questions about the study, and sign 2 copies of this consent form. (1 for clinic records, 1 for your records)
- Be given an eligibility and health questionnaire to complete, and assigned a screening number.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Will be screened by the Investigator or designee to see if you qualify for the study.
- If you do qualify for the study, you will:
  - o Take a urine pregnancy test (females of child-bearing potential)
  - Have a dermatologist confirm your eligibility
  - o Schedule your next appointment.

#### \*Visit 2: Baseline

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Be screened by the Investigator or designee to see if you still qualify for the study.
- Have your health and eligibility re-reviewed.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- If you still qualify for the study you will:
  - o Be assigned a subject number
  - Have photos taken of your face
  - o Be randomly assigned to receive one of the test products & supporting facial cleanser, moisturizer & facial SPF 30
  - o Be provided verbal and written usage instructions, and a daily diary to record product use
  - Schedule your next appointment

# **Visits 3, 4 (Week 1, Week 2)**

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and returned to you. At week 2, your diary will be retained by the testing facility and you will be given a new diary
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

# Visits 5, 6 (Week 6, Week 12)

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and retained. New products will be dispensed as necessary.
- Schedule your next appointment

# **Visit 7** (Week 18)

- Be asked if you have experienced any changes in your health since the previous visit.
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

# Visit 8 (Week 24)

- Be asked if you have experienced any changes in your health since the previous visit.
- Take a urine pregnancy test (females of child-bearing potential).
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility.
- Have your product collected, weighed, and retained by the testing facility.

Do not give the study product to other people and keep it out of the reach of children.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### RISKS OR DISCOMFORTS

If you do not understand what any of these side effects mean, please ask the investigator or study staff to explain these terms to you.

Because the study products are investigational, all of their side effects may not be known. There may be rare and unknown side effects. Some of these may be life threatening.

Possible risks associated with the product are, as with any other cosmetic and OTC products, signs of irritation including:

- Itching
- Burning
- Stinging
- Rash or other allergic reaction

- Tingling
- Scaling/Dryness
- Redness

In some cases, it is possible for a subject to develop allergic reactions to the test material(s). This risk is increased for individuals with a history of allergies, and individuals with asthma and/or a history of hives may also be affected. Symptoms include rash, hives, and itching.

You must tell the Investigator or study staff about all side effects that you have. If you are not honest about your side effects, it may not be safe for you to stay in the study.

## BIRTH CONTROL, DANGERS OF PREGNANCY AND BREASTFEEDING

If you are a female, you must not get pregnant while in this study. The only certain way to not get pregnant is to not have sex. If you are a female and choose to have sex, you must use a type of birth control.

Even if you use birth control during the study, there is a chance you could become pregnant. If you are pregnant or become pregnant during the study, test products or procedures may involve unforeseeable risks to the unborn baby.

A pregnancy test can be wrong. If you become pregnant during the study, stop using the test products and call/inform the Investigator at once.

You cannot be in the study if you are breastfeeding. It is not known whether the test products are safe for breast fed babies. Therefore if you are breastfeeding a child then it may not be safe for you to participate in the study.

#### POSSIBLE BENEFITS OF THE STUDY

You will not get any medical benefit from being in this study, and there is no promise that your condition (acne) will get better. It might stay the same or it might get worse. Your participation will provide information that may help others. There may be other marketed products that claim to have similar benefits.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

## OTHER OPTIONS TO PARTICIPATING IN THE STUDY

Since this study is for research only, the only other choice would be not to be in the study.


To participate in this study, you must agree to keep any information relating to the design, identity or use of these test product samples confidential.

On rare occasions, the sponsor may allow the testing company to disclose to you the name of the test products if you are not given this information during the study. This information is typically not provided until the end of the study or after the test products have been released for sale to the public. The study doctor or study staff will notify you if the sponsor allows us to give you this information.

#### DISCLOSURE AGREEMENT

This section explains how personal health information collected about you for the study may be used. Your personal health information includes, but is not limited to, information that was collected for your entry into the study and information that is collected during the study. The purpose of collecting this information is to allow the study staff and the Investigator to conduct the study, to evaluate the sponsor's study products and to analyze the study results.

You may decide not to give permission for the release of your personal health information for the study. In that case, you will not be able to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the sponsor's study products.

People who may inspect your personal and health information includes the Investigator, the Institutional Review Board, IntegReview IRB, FDA and other regulatory authorities from the United States or other countries, the study sponsor and people that work with the sponsor which includes, monitoring committees, contract research organizations, and consultants who have contracts with the company to do the study and review the study results. These reviews are done to check on the quality of the study and also for other purposes allowed by law.

The results of the study may be published in a medical book or journal, or presented at meetings for educational purposes. Neither your name, nor any other personal health information that specifically identifies you, will be used in those materials or presentations.

You may ask the Investigator to see and copy your personal health information related to the study. You may also ask the Investigator to correct any study related information about you that is wrong. You may have to wait until the end of the study to see your study records, so that the study can be organized properly.

This permission to share your personal health information for this study does not have an expiration date. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the Investigator at the address below:

Austin Institute for Clinical Research, Inc. 302 N. Heatherwilde Blvd., Suite 300 Pflugerville, TX 78660

If you cancel your permission after you have started in the study, the study staff and the Investigator will stop collecting your personal health information. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the study.

Austin Institute for Clinical Research, Inc. and the sponsor will make every effort to keep your personal health information private. But after the study staff or the Investigator share your personal health information from the study, federal privacy laws may not keep it private. There might be laws in your state or other federal laws that would protect the privacy of this information.

#### **CONFIDENTIALITY**

Your records of being in this study will be kept private except when ordered by law. The following people will have access to your study records:

- The Investigator
- Sponsor company or research institution [including monitor(s) and auditor(s)]
- Other country, state or federal regulatory agencies
- IntegReview IRB

The Institutional Review Board (IRB), IntegReview, and accrediting agencies may inspect and copy your records, which may have your name on them. Therefore, total confidentiality cannot be guaranteed. If the study results are presented at meetings or printed in publications, your name will not be used.

#### IN CASE OF STUDY RELATED INJURY

Side effects or complications, both foreseeable and unforeseeable, are possible in any research study without any fault to you, the Investigator, the study site, or the study sponsor. If you get hurt or sick as a direct result of being in this study, the sponsor will pay the costs of reasonable medical treatment. To ask questions about this, talk to the Investigator or study staff.

The sponsor's policy does not offer compensation for other expenses. Be aware that your health care payer/insurer might not cover the costs of study-related injuries or illnesses.

Unreimbursed medical expenses not covered by insurance or other third party coverage will be reimbursed by the sponsor for medical treatment for any injury that, in the opinion of the study doctor and the sponsor, is directly caused by the investigational product or by procedures required by the study protocol which would not have been performed as part of your regular medical care.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### **LEGAL RIGHTS**

You will not lose any of your legal rights by signing this consent form.

#### **CONTACT INFORMATION**

If you have questions, concerns, or complaints about this study or to report a study related injury, contact:

Edward Lain, MD 512-279-2545 daytime telephone number 512-844-4500 after hours number

If you are unable to reach anyone at the number(s) listed above and you need medical attention, please go to the nearest emergency room.

If you do not want to talk to the Investigator or study staff, if you have concerns or complaints about the research, or to ask questions about your rights as a study subject you may contact IntegReview. IntegReview's policy indicates that all concerns/complaints are to be submitted in writing for review at a convened IRB meeting to:

| Mailing Address: | OR | Email Address: |
|----------------------------------|----|-----------------------------|
| Chairperson | | integreview@integreview.com |
| IntegReview IRB | | |
| 3815 S. Capital of Texas Highway | | |
| Suite 320 | | |
| Austin, TX 78704 | | |

If you are unable to provide your concerns/complaints in writing or if this is an emergency situation regarding subject safety, contact our office at:

512-326-3001 or toll free at 1-877-562-1589 between 8 a.m. and 5 p.m. Central Time

IntegReview has approved the information in this consent form and has given approval for the Investigator to do the study. This does not mean IntegReview has approved your being in the study. You must consider the information in this consent form for yourself and decide if you want to be in this study.

## PAYMENT FOR BEING IN THE STUDY

You may receive up to \$575.00 for being in the study. You will be paid per completed visit as follows:

| Visit | Compensation (amount) |
|---------------------------------|-----------------------|
| Screening/Baseline (Visit 1, 2) | \$40.00 |
| Visit 3 | \$60.00 |
| Visit 4 | \$65.00 |
| Visit 5 | \$75.00 |
| Visit 6 | \$90.00 |

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

VERSION CONTROL

clw/master: 2-17-16 snb/site: 2-25-16 clw/site: 2-29-16

| Visit 7 | \$95.00 |
|---------|----------|
| Visit 8 | \$150.00 |

If you choose to leave or are withdrawn from the study for any reason before finishing all visits you will be paid for each completed visit. You will receive payment at the end of each study visit.

If you do not qualify for any reason, you will be paid \$20.00, which will be mailed to you within 2 weeks of the baseline study visit.

If you are paid \$600.00 or more by Austin Institute for Clinical Research, Inc. in a calendar year, those payments will be reported to the Internal Revenue Service via form 1099-MISC. As required by tax laws, if you withhold your social security number, Austin Institute for Clinical Research, Inc. is required to withhold 28% of your payment for tax purposes. In this case a form 1099-MISC will be sent to you reporting your withholding.

## **VOLUNTEERING TO BE IN THE STUDY**

It is your choice if you want to be in the study. No one can force you to be in the study. You may not want to be in this study or you may leave the study at any time without penalty or loss of benefits to which you are otherwise entitled.

The Investigator, the sponsor company, or IntegReview may take you out of the study without your permission, at any time, for the following reasons:

- If you do not follow the Investigator's instructions
- If we find out you should not be in the study
- If the study is stopped
- If it becomes harmful to your health

If you leave the study or if you are taken out of the study, you may be asked to return for a final visit to have some end of study evaluations or tests. If information generated from this study is published or presented, your identity will not be revealed. If you leave the study, no more information about you will be collected for this study. However, all of the information you gave us before you left the study will still be used.

#### **NEW FINDINGS**

If there is new information or any significant new findings that could relate to your willingness to continue participation we will tell you. You can then decide if you still want to be in the study.

#### THE REASON FOR INSTITUTIONAL REVIEW BOARDS AND INFORMED CONSENT

#### What is a consent form?

The informed consent document contains information required by federal regulations. The informed consent document must be approved by an Institutional Review Board (IRB).

## What is an Institutional Review Board (IRB)?

An Institutional Review Board (IRB) is a group of people that reviews research studies. The main goal of this review is to protect the rights and well being of the human subjects participating in research studies.

# IntegReview, the IRB for this study

IntegReview is an IRB whose board members provide IRB services across the United States, Canada, Japan and Latin America.

To meet requirements of the law, the IntegReview Boards currently include:

- Doctors
- Pharmacists
- Nurses
- Toxicologists (people who study the harmful effects of chemicals)
- Other specialists
- Others who do not have a background in science/medicine

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

## AGREEMENT TO BE IN THE STUDY

This consent form contains important information to help you decide if you want to be in the study. If you have any questions that are not answered in this consent form, ask one of the study staff.

| Pleas | e answer YES or NO to the following questions: | |
|---|---|---|
| A. | Is this document in a language you understand? | |
| B. | Do you understand the information in this consent form? | |
| C. | Have you been given enough time to ask questions and talk about the study? | |
| D. | Have all of your questions been answered to your satisfaction? | |
| E. | Do you think you received enough information about the study? | |
| F. | Do you volunteer to be in this study of your own free will and without being pressured by the Investigator or study staff? | |
| G. | Do you know that you can leave the study at any time without giving a reason and without affecting your health care? | |
| Н. | Do you know that your health records from this study may be reviewed by the sponsor company and by government authorities? | |
| I. | Do you know that you cannot be in another study while you are in this study? | |
| | IF YOU ANSWERED "NO" TO ANY OF THE ABOVE QUESTION OR YOU ARE UNABLE TO ANSWER ANY OF THE ABOVE QUESTION YOU SHOULD NOT SIGN THIS CONSENT FORM. | |
| Printe | ed Name of Adult Study Subject | |
| Signa | ture of Adult Study Subject | Date |
| Printe | ed Name of Person Explaining Consent Form | |
| Signa | ture of Person Explaining Consent Form | Date |
| You v | will be given a signed and dated copy of this consent form to keep. | |

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

## **Authorization and Release Form**

I hereby for good and valuable consideration grant to Austin Institute for Clinical Research, Inc., the study sponsor and their respective affiliates, agencies, agents, employees, and assigns (collectively, "Authorized Entities"), the unrestricted, royalty free, irrevocable and perpetual right and permission to reproduce, distribute, broadcast and/or otherwise use for advertising and other commercial/noncommercial purposes: (i) my name, likeness, image, video, and any other biographical or personal information ("Personal Content"); and (ii) any statement or endorsement, or any portions thereof ("Testimonial(s)"), made by me relating to the study sponsor's products ("Products"), in any and all media now known or later developed, worldwide in perpetuity, without further compensation or approval by me.

I hereby assign to the Authorized Entities all of my world-wide right, title and interest, including my copyright interests and all renewals, reissues and extensions thereof, in and to the Personal Content and Testimonial(s), including without limitation, any photographic portraits, sound recordings and video performances of and/or by me in connection with the Personal Content and/or Testimonial(s).

I am at least 21 years of age, and competent to contract in my own name. I have read and understand this

| Authorization and Release. | | |
|---|---|---|
| Printed Name of Adult Study Subject | | |
| Signature of Adult Study Subject | | Date |
| Printed Name of Person Explaining Release Form | | |
| Signature of Person Explaining Release Form | | Date |
| Copy of consent form given to subject on | (date) by | (initials) |
| You will be given a signed and dated copy of this | consent form to keep. | |

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

# AUTHORIZATION TO USE AND DISCLOSE PERSONAL HEALTH INFORMATION FOR RESEARCH

THIS SECTION DESCRIBES YOUR RIGHTS AND HOW PERSONAL HEALTH INFORMATION COLLECTED ABOUT YOU DURING THIS STUDY MAY BE USED AND DISCLOSED AND HOW YOU CAN GET ACCESS TO THIS INFORMATION. PLEASE REVIEW IT CAREFULLY.

The United States government has issued a privacy rule to protect the privacy rights of patients. This rule was issued under a law called the Health Insurance Portability and Accountability Act of 1996 (HIPAA). The Privacy Rule is designed to protect the confidentiality of your personal health information. The document you are reading, called an "Authorization," describes your rights and explains how your health information will be used and disclosed (shared).

Federal law requires hospitals, researchers and health care providers to protect the privacy of information that identifies you and relates to your past, present and future physical and mental health or conditions.

All information collected during the study will be retained by the study doctor and the Study Sponsor, except as required by law. Information from this study will be given to the sponsor. "Sponsor" includes any persons or companies, which are contracted by the sponsor to have access to the research information during and after the study. The information will also be given to the U.S. Food and Drug Administration (FDA). Study records which identify you and the consent form signed by you will be inspected and/or copied for research or regulatory purposes by:

- Sponsor
- Agents for the sponsor
- The US Food and Drug Administration (FDA)
- Department of Health and Human Services (DHHS) agencies
- IntegReview IRB

Because of the need to release information to these parties, absolute confidentiality cannot be guaranteed. The results of this research study may be presented at meetings or in publications; however, your identity will not be disclosed in those presentations.

For purposes of study reporting, you will be identified by your initials and code numbers only. However, your name, date of birth, address, and phone number will be kept on record by the study doctor in case you need to be contacted in the future about this study.

After your personal health information is disclosed to the Study Sponsor, the results of the study may be reanalyzed at a later date and may be combined with the results of other studies. The Study Sponsor and people who work with the Study Sponsor may use the results of this study for other research purposes, including:

- Developing a better understanding of the disease;
- Improving the design of future actual use trials

After the study staff or the study doctor discloses your personal health information to others, it could be re-disclosed and no longer protected by federal privacy laws.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you do not withdraw this Authorization in writing, it will remain in effect indefinitely. Your study doctor will keep this Authorization for at least 6 years. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the study doctor at the address below:

Austin Institute for Clinical Research, Inc. 302 N. Heatherwilde Blvd., Suite 300 Pflugerville, TX 78660

You have the right to see and get a copy of your records related to the study for as long as the study doctor has this information. However, by signing this Authorization you agree that you might not be able to review or receive some of your records related to the study until after the study has been completed.

If you cancel your permission after you have started in the study, the study staff and the study doctor will stop collecting your personal health information unless the information concerns an adverse event (a bad effect) related to the study. If an adverse event occurs, your entire medical record may be reviewed. All information that has already been collected for study purposes, and any new information about an adverse event related to the study, will be sent to the study sponsor. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the study doctor would not be able to collect the information needed to evaluate the study results.

If you withdraw from the study but do not withdraw your Authorization, new personal health information may be collected until this study ends.

You may decide not to give permission for the release of your personal health information for this study. In that case, you will not be able to participate. This is because the study staff and study doctor would not be able to collect the information needed to evaluate the study results.

At the completion of the study, you have the right to access your protected health information that is created during this research study that relates to your treatment or to payment, provided such information is not exempted under certain laws and regulations. To request this information, please contact the study doctor at the address listed above.

# **Your Right to Access Health Information**

Subject to certain exceptions prescribed by law, you have a right to request access to the health information that we hold about you and to request changes if your health information is incorrect or incomplete. Any request for access or corrections should be made to the principal doctor conducting this study.

Your records obtained while you are in this trial, as well as related health records, will remain strictly confidential at all times. However, these will need to be made available to others working on the Sponsor's behalf, the Independent Ethics Committee members and Medicines Regulatory Authorities.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

By signing the consent form you agree to this access for the current trial and any further research that may be done. However, the Sponsor will take steps to protect your personal information and will not include your name on any sponsor forms, reports, publications, or in any future disclosures. If you withdraw from the study, we will no longer collect your personal information, but we may need to continue to use information already collected.

Personal data which may be sensitive (e.g., date of birth) will be collected and processed, but only for research purposes in connection with this trial.

The trial data will be sent around the world, but you will not be referred to by name or identified in any report or publication nor could the data be traced back to you. Your data may be transferred to a country that does not have the same level of personal data protection as within the United States. However, The Sponsor maintains high standards of confidentiality and protection.

The Sponsor (who will control the use of the data) will take steps to ensure your personal data is protected.

By taking part in this trial you agree not to restrict the use of any data even if you withdraw from the trial and agree to the transfer of your personal data to other Sponsor companies and to Medicines Regulatory Authorities both within and outside of Europe.

| Printed Name of Adult Study Subject | |
|-------------------------------------|------|
| Signature of Adult Study Subject | Date |

# INFORMED CONSENT DOCUMENT AGREEMENT TO BE IN A RESEARCH STUDY

**NAME OF TESTING COMPANY:** Austin Institute for Clinical Research, Inc.

NUMBER AND TITLE OF STUDY: C16-CD020 (GLI.04.SPR.US10354); "A Multi-

Center Clinical Trial to Evaluate the Efficacy of

Two Acne Treatments"

NAME OF PERSON IN CHARGE OF

THE RESEARCH STUDY

(STUDY DOCTOR/INVESTIGATOR): Edward Lain, MD

**TELEPHONE NUMBER(S), DAYTIME:** 512-279-2545 **AFTER HOURS:** 512-844-4500

#### INTRODUCTION

You are being invited to volunteer for a clinical research study. You must read and sign this form before you agree to take part in this study. This form will give you more information about this study. Please ask as many questions as you need to before you decide if you want to be in the study. You should not sign this form if you have any questions that have not been answered.

Austin Institute for Clinical Research, Inc. is being paid by the sponsor (the company paying for this study) to conduct this research study.

You must be honest with the Investigator about your health history or it may not be safe for you to be in this study.

## PURPOSE OF THE STUDY

The purpose of this study is to evaluate the efficiency of 2 acne treatments for 24 weeks of use in adult men and women with mild to moderate facial acne, at least 5 inflammatory lesions, and at least 10 - 100 non-inflammatory lesions.

#### HOW LONG THE STUDY WILL LAST AND HOW MANY PEOPLE WILL BE IN THE STUDY

This study will last 24 weeks and have up to 8 visits. At least 100 subjects, men and women between the ages of 21-45, are expected to complete this study, with at least 50 subjects completed per cell.

## TO BE IN THIS STUDY

#### You must:

- Be a man or woman age 21 to 45 years at the time of enrollment.
- Have mild to moderate acne on the face as determined by the Investigator or designee.
- Have at least 5 inflammatory lesions as determined by the Investigator or designee.
- Have 10 100 non-inflammatory lesions as determined by the Investigator or designee.
- Be willing to use the test products as instructed for 24 weeks.
- Be willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol.

- Be willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and be able to read, speak, write, understand English and be willing to share personal information and data, as verified by signing a written authorization at the screening.
- Be willing to withhold all facial treatments during the course of the study including botulinum toxin, injectable fillers, microdermabrasion, IPL, peels, facials, laser treatments and tightening treatments. Waxing and threading is allowed but not facial laser hair removal.
- Males must be regular shavers and willing to shave on the day of the study visits (prior to clinic visits).
- Women of child bearing potential must be willing to take a urine pregnancy test prior to study enrollment, at week 24, and when deemed appropriate by the Investigator and/or Sponsor.
- Individuals of child bearing potential must use an acceptable method of contraception throughout the study. Acceptable methods of birth control include:
  - Oral and other system contraceptives. Individuals must be on a stable use for 3 months prior to study enrollment. Individuals on oral contraceptives must not alter their use, including dose or regimen for the duration of the study
  - o Double barrier
  - o Bilateral tubal ligation (tubes tied)
  - o Partner vasectomy
  - Abstinence
- Be willing to follow study requirements and report any changes in health status or medications, side effect symptoms, or reactions immediately.
- Be stable on any medication you are taking for at least 30 days

#### YOU CANNOT BE ON THE STUDY

## If you:

- Have been diagnosed with allergies to topical acne products.
- Have a condition and/or disease of the skin that the Investigator deems inappropriate for participation.
- Are a woman who is breastfeeding, pregnant, or planning to become pregnant during the study.
- Have pre-existing or dormant dermatologic conditions on the face (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, severe excoriations etc.) which in the opinion of the Investigator could interfere with the outcome of the study.
- Have a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.).
- Have an uncontrolled disease such as asthma, diabetes, hypertension, hyperthyroidism, or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc. at the Investigator's discretion.
- Are currently participating in another facial usage study or have participated in a clinical trial within 4 weeks prior to inclusion into the study.
- Have a history of skin cancer on the face within the past 5 years.
- Have any planned surgeries and/or invasive medical procedures during the course of the study.
- Have started hormone replacement therapies (HRT) or hormones for birth control less than 3 months
  prior to study entry or plan on starting, stopping, or changing doses of HRT or hormones for birth
  control during the study.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Have facial sunburn or excessive tanned facial skin or are not willing to avoid daily sun exposure on the face and the use of tanning beds or sunless tanning products for the duration of the study.
- Have severe acne, acne conglobata, multiple nodules or cysts (more than 2).
- Are currently taking a natural or prescription testosterone blocker (e.g. saw palmetto, blask cohosh, chaste tree, chasteberry, spironolactone, drospirenone, progestins).
- Are currently on a testosterone booster or prescription testosterone (e.g. DHEA, tribulus, testosterone cypionate, testosterone enanthate, Sustanon, testosterone propionate, testosterone phenylpropriate, Omnadren etc.).
- Are currently taking or have taken within the last 30 days oral or topical prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin (Retin A, Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo.
- Have used oral isotretinoin (Accutane) within the past 6-months.
- Are routinely using (3x a week or more) topical over-the-counter (OTC) acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 14 days of the study entry.
- Are using or have used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study.
- Have excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations as determined by the Investigator or designee.

#### WHAT WILL HAPPEN DURING THE STUDY

## \*Visit 1: Screening (\* Visit 1 {Screening} AND Visit 2 {Baseline} may be combined into 1 Visit)

## You will:

- Be given an IRB-approved Informed Consent Form (ICF), to read and sign. You will be given enough time to read the informed consent, and ask questions about the study, and sign 2 copies of this consent form. (1 for clinic records, 1 for your records)
- Be given an eligibility and health questionnaire to complete, and assigned a screening number.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Will be screened by the Investigator or designee to see if you qualify for the study.
- If you do qualify for the study, you will:
  - o Take a urine pregnancy test (females of child-bearing potential)
  - Have a dermatologist confirm your eligibility
  - o Schedule your next appointment.

## \*Visit 2: Baseline

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Be screened by the Investigator or designee to see if you still qualify for the study.
- Have your health and eligibility re-reviewed.
- If you still qualify for the study you will:
  - o Be assigned a subject number
  - Have photos taken of your face

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Be randomly assigned to receive one of the test products & supporting facial cleanser, moisturizer & facial SPF 30
- o Be provided verbal and written usage instructions, and a daily diary to record product use
- Schedule your next appointment

## **Visits 3, 4 (Week 1, Week 2)**

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and returned to you. At week 2, your diary
  will be retained by the testing facility and you will be given a new diary
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

## Visits 5, 6 (Week 6, Week 12)

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and retained. New products will be dispensed as necessary.
- Schedule your next appointment

## **Visit 7 (Week 18)**

- Be asked if you have experienced any changes in your health since the previous visit.
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

# <u>Visit 8 (Week 24)</u>

- Be asked if you have experienced any changes in your health since the previous visit.
- Take a urine pregnancy test (females of child-bearing potential).
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility.
- Have your product collected, weighed, and retained by the testing facility.

Do not give the study product to other people and keep it out of the reach of children.

## RISKS OR DISCOMFORTS

If you do not understand what any of these side effects mean, please ask the investigator or study staff to explain these terms to you.

Because the study products are investigational, all of their side effects may not be known. There may be rare and unknown side effects. Some of these may be life threatening.

Possible risks associated with the product are, as with any other cosmetic and OTC products, signs of irritation including:

- Itching
- Burning
- Stinging
- Rash or other allergic reaction

- Tingling
- Scaling/Dryness
- Redness

In some cases, it is possible for a subject to develop allergic reactions to the test material(s). This risk is increased for individuals with a history of allergies, and individuals with asthma and/or a history of hives may also be affected. Symptoms include rash, hives, and itching.

You must tell the Investigator or study staff about all side effects that you have. If you are not honest about your side effects, it may not be safe for you to stay in the study.

## BIRTH CONTROL, DANGERS OF PREGNANCY AND BREASTFEEDING

If you are a female, you must not get pregnant while in this study. The only certain way to not get pregnant is to not have sex. If you are a female and choose to have sex, you must use a type of birth control.

Even if you use birth control during the study, there is a chance you could become pregnant. If you are pregnant or become pregnant during the study, test products or procedures may involve unforeseeable risks to the unborn baby.

A pregnancy test can be wrong. If you become pregnant during the study, stop using the test products and call/inform the Investigator at once.

You cannot be in the study if you are breastfeeding. It is not known whether the test products are safe for breast fed babies. Therefore if you are breastfeeding a child then it may not be safe for you to participate in the study.

#### POSSIBLE BENEFITS OF THE STUDY

You will not get any medical benefit from being in this study, and there is no promise that your condition (acne) will get better. It might stay the same or it might get worse. Your participation will provide information that may help others. There may be other marketed products that claim to have similar benefits.

## OTHER OPTIONS TO PARTICIPATING IN THE STUDY

Since this study is for research only, the only other choice would be not to be in the study.


To participate in this study, you must agree to keep any information relating to the design, identity or use of these test product samples confidential.

On rare occasions, the sponsor may allow the testing company to disclose to you the name of the test products if you are not given this information during the study. This information is typically not provided until the end of the study or after the test products have been released for sale to the public. The study doctor or study staff will notify you if the sponsor allows us to give you this information.

#### DISCLOSURE AGREEMENT

This section explains how personal health information collected about you for the study may be used. Your personal health information includes, but is not limited to, information that was collected for your entry into the study and information that is collected during the study. The purpose of collecting this information is to allow the study staff and the Investigator to conduct the study, to evaluate the sponsor's study products and to analyze the study results.

You may decide not to give permission for the release of your personal health information for the study. In that case, you will not be able to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the sponsor's study products.

People who may inspect your personal and health information includes the Investigator, the Institutional Review Board, IntegReview IRB, FDA and other regulatory authorities from the United States or other countries, the study sponsor and people that work with the sponsor which includes, monitoring committees, contract research organizations, and consultants who have contracts with the company to do the study and review the study results. These reviews are done to check on the quality of the study and also for other purposes allowed by law.

The results of the study may be published in a medical book or journal, or presented at meetings for educational purposes. Neither your name, nor any other personal health information that specifically identifies you, will be used in those materials or presentations.

You may ask the Investigator to see and copy your personal health information related to the study. You may also ask the Investigator to correct any study related information about you that is wrong. You may have to wait until the end of the study to see your study records, so that the study can be organized properly.

This permission to share your personal health information for this study does not have an expiration date. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the Investigator at the address below:

Austin Institute for Clinical Research, Inc. 302 N. Heatherwilde Blvd., Suite 300 Pflugerville, TX 78660

If you cancel your permission after you have started in the study, the study staff and the Investigator will stop collecting your personal health information. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the study.

Austin Institute for Clinical Research, Inc. and the sponsor will make every effort to keep your personal health information private. But after the study staff or the Investigator share your personal health information from the study, federal privacy laws may not keep it private. There might be laws in your state or other federal laws that would protect the privacy of this information.

#### **CONFIDENTIALITY**

Your records of being in this study will be kept private except when ordered by law. The following people will have access to your study records:

- The Investigator
- Sponsor company or research institution [including monitor(s) and auditor(s)]
- Other country, state or federal regulatory agencies
- IntegReview IRB

The Institutional Review Board (IRB), IntegReview, and accrediting agencies may inspect and copy your records, which may have your name on them. Therefore, total confidentiality cannot be guaranteed. If the study results are presented at meetings or printed in publications, your name will not be used.

#### IN CASE OF STUDY RELATED INJURY

Side effects or complications, both foreseeable and unforeseeable, are possible in any research study without any fault to you, the Investigator, the study site, or the study sponsor. If you get hurt or sick as a direct result of being in this study, the sponsor will pay the costs of reasonable medical treatment. To ask questions about this, talk to the Investigator or study staff.

The sponsor's policy does not offer compensation for other expenses. Be aware that your health care payer/insurer might not cover the costs of study-related injuries or illnesses.

Unreimbursed medical expenses not covered by insurance or other third party coverage will be reimbursed by the sponsor for medical treatment for any injury that, in the opinion of the study doctor and the sponsor, is directly caused by the investigational product or by procedures required by the study protocol which would not have been performed as part of your regular medical care.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### **LEGAL RIGHTS**

You will not lose any of your legal rights by signing this consent form.

#### **CONTACT INFORMATION**

If you have questions, concerns, or complaints about this study or to report a study related injury, contact:

Edward Lain, MD 512-279-2545 daytime telephone number 512-844-4500 after hours number

If you are unable to reach anyone at the number(s) listed above and you need medical attention, please go to the nearest emergency room.

If you do not want to talk to the Investigator or study staff, if you have concerns or complaints about the research, or to ask questions about your rights as a study subject you may contact IntegReview. IntegReview's policy indicates that all concerns/complaints are to be submitted in writing for review at a convened IRB meeting to:

| Mailing Address: | OR | Email Address: |
|----------------------------------|----|-----------------------------|
| Chairperson | | integreview@integreview.com |
| IntegReview IRB | | |
| 3815 S. Capital of Texas Highway | | |
| Suite 320 | | |
| Austin, TX 78704 | | |

If you are unable to provide your concerns/complaints in writing or if this is an emergency situation regarding subject safety, contact our office at:

512-326-3001 or toll free at 1-877-562-1589 between 8 a.m. and 5 p.m. Central Time

IntegReview has approved the information in this consent form and has given approval for the Investigator to do the study. This does not mean IntegReview has approved your being in the study. You must consider the information in this consent form for yourself and decide if you want to be in this study.

## PAYMENT FOR BEING IN THE STUDY

You may receive up to \$575.00 for being in the study. You will be paid per completed visit as follows:

| Visit | Compensation (amount) |
|---------------------------------|-----------------------|
| Screening/Baseline (Visit 1, 2) | \$40.00 |
| Visit 3 | \$60.00 |
| Visit 4 | \$65.00 |
| Visit 5 | \$75.00 |
| Visit 6 | \$90.00 |

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

| Visit 7 | \$95.00 |
|---------|----------|
| Visit 8 | \$150.00 |

If you choose to leave or are withdrawn from the study for any reason before finishing all visits you will be paid for each completed visit. You will receive payment at the end of each study visit.

If you do not qualify for any reason, you will be paid \$20.00, which will be mailed to you within 2 weeks of the baseline study visit.

If you are paid \$600.00 or more by Austin Institute for Clinical Research, Inc. in a calendar year, those payments will be reported to the Internal Revenue Service via form 1099-MISC. As required by tax laws, if you withhold your social security number, Austin Institute for Clinical Research, Inc. is required to withhold 28% of your payment for tax purposes. In this case a form 1099-MISC will be sent to you reporting your withholding.

## **VOLUNTEERING TO BE IN THE STUDY**

It is your choice if you want to be in the study. No one can force you to be in the study. You may not want to be in this study or you may leave the study at any time without penalty or loss of benefits to which you are otherwise entitled.

The Investigator, the sponsor company, or IntegReview may take you out of the study without your permission, at any time, for the following reasons:

- If you do not follow the Investigator's instructions
- If we find out you should not be in the study
- If the study is stopped
- If it becomes harmful to your health

If you leave the study or if you are taken out of the study, you may be asked to return for a final visit to have some end of study evaluations or tests. If information generated from this study is published or presented, your identity will not be revealed. If you leave the study, no more information about you will be collected for this study. However, all of the information you gave us before you left the study will still be used.

#### **NEW FINDINGS**

If there is new information or any significant new findings that could relate to your willingness to continue participation we will tell you. You can then decide if you still want to be in the study.

#### THE REASON FOR INSTITUTIONAL REVIEW BOARDS AND INFORMED CONSENT

#### What is a consent form?

The informed consent document contains information required by federal regulations. The informed consent document must be approved by an Institutional Review Board (IRB).

## What is an Institutional Review Board (IRB)?

An Institutional Review Board (IRB) is a group of people that reviews research studies. The main goal of this review is to protect the rights and well being of the human subjects participating in research studies.

# IntegReview, the IRB for this study

IntegReview is an IRB whose board members provide IRB services across the United States, Canada, Japan and Latin America.

To meet requirements of the law, the IntegReview Boards currently include:

- Doctors
- Pharmacists
- Nurses
- Toxicologists (people who study the harmful effects of chemicals)
- Other specialists
- Others who do not have a background in science/medicine

## AGREEMENT TO BE IN THE STUDY

This consent form contains important information to help you decide if you want to be in the study. If you have any questions that are not answered in this consent form, ask one of the study staff.

| Pleas | e answer YES or NO to the following questions: | |
|---|---|---|
| A. | Is this document in a language you understand? | |
| B. | Do you understand the information in this consent form? | |
| C. | Have you been given enough time to ask questions and talk about the study? | |
| D. | Have all of your questions been answered to your satisfaction? | |
| E. | Do you think you received enough information about the study? | |
| F. | Do you volunteer to be in this study of your own free will and without being pressured by the Investigator or study staff? | |
| G. | Do you know that you can leave the study at any time without giving a reason and without affecting your health care? | |
| Н. | Do you know that your health records from this study may be reviewed by the sponsor company and by government authorities? | |
| I. | Do you know that you cannot be in another study while you are in this study? | |
| | IF YOU ANSWERED "NO" TO ANY OF THE ABOVE QUESTIO OR YOU ARE UNABLE TO ANSWER ANY OF THE ABOVE QUES' YOU SHOULD NOT SIGN THIS CONSENT FORM. | |
| Print | ed Name of Adult Study Subject | |
| Signa | nture of Adult Study Subject | Date |
| Print | ed Name of Person Explaining Consent Form | |
| Signa | ature of Person Explaining Consent Form | Date |
| You | will be given a signed and dated copy of this consent form to keep. | |

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

## **Authorization and Release Form**

I hereby for good and valuable consideration grant to Austin Institute for Clinical Research, Inc., the study sponsor and their respective affiliates, agencies, agents, employees, and assigns (collectively, "Authorized Entities"), the unrestricted, royalty free, irrevocable and perpetual right and permission to reproduce, distribute, broadcast and/or otherwise use for advertising and other commercial/noncommercial purposes: (i) my name, likeness, image, video, and any other biographical or personal information ("Personal Content"); and (ii) any statement or endorsement, or any portions thereof ("Testimonial(s)"), made by me relating to the study sponsor's products ("Products"), in any and all media now known or later developed, worldwide in perpetuity, without further compensation or approval by me.

I hereby assign to the Authorized Entities all of my world-wide right, title and interest, including my copyright interests and all renewals, reissues and extensions thereof, in and to the Personal Content and Testimonial(s), including without limitation, any photographic portraits, sound recordings and video performances of and/or by me in connection with the Personal Content and/or Testimonial(s).

I am at least 21 years of age, and competent to contract in my own name. I have read and understand this

| Authorization and Release. | | |
|---|---|---|
| Printed Name of Adult Study Subject | | |
| Signature of Adult Study Subject | | Date |
| Printed Name of Person Explaining Release Form | | |
| Signature of Person Explaining Release Form | | Date |
| Copy of consent form given to subject on | (date) by | (initials) |
| You will be given a signed and dated copy of this | consent form to keep. | |

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

# AUTHORIZATION TO USE AND DISCLOSE PERSONAL HEALTH INFORMATION FOR RESEARCH

THIS SECTION DESCRIBES YOUR RIGHTS AND HOW PERSONAL HEALTH INFORMATION COLLECTED ABOUT YOU DURING THIS STUDY MAY BE USED AND DISCLOSED AND HOW YOU CAN GET ACCESS TO THIS INFORMATION. PLEASE REVIEW IT CAREFULLY.

The United States government has issued a privacy rule to protect the privacy rights of patients. This rule was issued under a law called the Health Insurance Portability and Accountability Act of 1996 (HIPAA). The Privacy Rule is designed to protect the confidentiality of your personal health information. The document you are reading, called an "Authorization," describes your rights and explains how your health information will be used and disclosed (shared).

Federal law requires hospitals, researchers and health care providers to protect the privacy of information that identifies you and relates to your past, present and future physical and mental health or conditions.

All information collected during the study will be retained by the study doctor and the Study Sponsor, except as required by law. Information from this study will be given to the sponsor. "Sponsor" includes any persons or companies, which are contracted by the sponsor to have access to the research information during and after the study. The information will also be given to the U.S. Food and Drug Administration (FDA). Study records which identify you and the consent form signed by you will be inspected and/or copied for research or regulatory purposes by:

- Sponsor
- Agents for the sponsor
- The US Food and Drug Administration (FDA)
- Department of Health and Human Services (DHHS) agencies
- IntegReview IRB

Because of the need to release information to these parties, absolute confidentiality cannot be guaranteed. The results of this research study may be presented at meetings or in publications; however, your identity will not be disclosed in those presentations.

For purposes of study reporting, you will be identified by your initials and code numbers only. However, your name, date of birth, address, and phone number will be kept on record by the study doctor in case you need to be contacted in the future about this study.

After your personal health information is disclosed to the Study Sponsor, the results of the study may be reanalyzed at a later date and may be combined with the results of other studies. The Study Sponsor and people who work with the Study Sponsor may use the results of this study for other research purposes, including:

- Developing a better understanding of the disease;
- Improving the design of future actual use trials

After the study staff or the study doctor discloses your personal health information to others, it could be re-disclosed and no longer protected by federal privacy laws.

This permission to share your personal health information for this study does not have an expiration date. If you do not withdraw this Authorization in writing, it will remain in effect indefinitely. Your study doctor will keep this Authorization for at least 6 years. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the study doctor at the address below:

Austin Institute for Clinical Research, Inc. 302 N. Heatherwilde Blvd., Suite 300 Pflugerville, TX 78660

You have the right to see and get a copy of your records related to the study for as long as the study doctor has this information. However, by signing this Authorization you agree that you might not be able to review or receive some of your records related to the study until after the study has been completed.

If you cancel your permission after you have started in the study, the study staff and the study doctor will stop collecting your personal health information unless the information concerns an adverse event (a bad effect) related to the study. If an adverse event occurs, your entire medical record may be reviewed. All information that has already been collected for study purposes, and any new information about an adverse event related to the study, will be sent to the study sponsor. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the study doctor would not be able to collect the information needed to evaluate the study results.

If you withdraw from the study but do not withdraw your Authorization, new personal health information may be collected until this study ends.

You may decide not to give permission for the release of your personal health information for this study. In that case, you will not be able to participate. This is because the study staff and study doctor would not be able to collect the information needed to evaluate the study results.

At the completion of the study, you have the right to access your protected health information that is created during this research study that relates to your treatment or to payment, provided such information is not exempted under certain laws and regulations. To request this information, please contact the study doctor at the address listed above.

# **Your Right to Access Health Information**

Subject to certain exceptions prescribed by law, you have a right to request access to the health information that we hold about you and to request changes if your health information is incorrect or incomplete. Any request for access or corrections should be made to the principal doctor conducting this study.

Your records obtained while you are in this trial, as well as related health records, will remain strictly confidential at all times. However, these will need to be made available to others working on the Sponsor's behalf, the Independent Ethics Committee members and Medicines Regulatory Authorities.

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

By signing the consent form you agree to this access for the current trial and any further research that may be done. However, the Sponsor will take steps to protect your personal information and will not include your name on any sponsor forms, reports, publications, or in any future disclosures. If you withdraw from the study, we will no longer collect your personal information, but we may need to continue to use information already collected.

Personal data which may be sensitive (e.g., date of birth) will be collected and processed, but only for research purposes in connection with this trial.

The trial data will be sent around the world, but you will not be referred to by name or identified in any report or publication nor could the data be traced back to you. Your data may be transferred to a country that does not have the same level of personal data protection as within the United States. However, The Sponsor maintains high standards of confidentiality and protection.

The Sponsor (who will control the use of the data) will take steps to ensure your personal data is protected.

By taking part in this trial you agree not to restrict the use of any data even if you withdraw from the trial and agree to the transfer of your personal data to other Sponsor companies and to Medicines Regulatory Authorities both within and outside of Europe.

| Printed Name of Adult Study Subject | |
|-------------------------------------|------|
| Signature of Adult Study Subject | Date |

# INFORMED CONSENT DOCUMENT AGREEMENT TO BE IN A RESEARCH STUDY

NAME OF TESTING COMPANY: RCTS, Inc.,

NUMBER AND TITLE OF STUDY: C16-CD020 (GLI.04.SPR.US10354); "A Multi-

Center Clinical Trial to Evaluate the Efficacy of

Two Acne Treatments"

NAME OF PERSON IN CHARGE OF THE

**RESEARCH STUDY (INVESTIGATOR):** Barry T. Reece, M.S., M.B.A.

Principal Investigator

**MEDICAL INVESTIGATORS:** Raymond L. Garcia, M.D.

**Board Certified Dermatologist** 

Gene Ream, M.D.

**Board Certified Dermatologist** 

TELEPHONE NUMBER(S), DAYTIME: 972-871-7578

**AFTER HOURS:** 972-841-2916 (Emergencies Only, Cell Phone

Number)

#### INTRODUCTION

You are being invited to volunteer for a clinical research study. You must read and sign this form before you agree to take part in this study. This form will give you more information about this study. Please ask as many questions as you need to before you decide if you want to be in the study. You should not sign this form if you have any questions that have not been answered.

RCTS, Inc., a contract research organization, is being paid by the sponsor (the company paying for this study) to conduct this research study.

You must be honest with the Investigator about your health history or it may not be safe for you to be in this study.

## **PURPOSE OF THE STUDY**

The purpose of this study is to evaluate the efficiency of 2 acne treatments for 24 weeks of use in adult men and women with mild to moderate facial acne, at least 5 inflammatory lesions, and at least 10 - 100 non-inflammatory lesions.

## HOW LONG THE STUDY WILL LAST AND HOW MANY PEOPLE WILL BE IN THE STUDY

This study will last 24 weeks and have up to 8 visits. At least 100 subjects, men and women between the ages of 21-45, are expected to complete this study, with at least 50 subjects completed per cell. Each site is to enroll no more than 40 subjects, with at least 100 subjects expected to complete when combined.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

**VERSION CONTROL** 

clw/master: 2-17-16 snb/site: 2-25-16

#### TO BE IN THIS STUDY

#### You must:

- Be a man or woman age 21 to 45 years at the time of enrollment.
- Have mild to moderate acne on the face as determined by the Investigator or designee.
- Have at least 5 inflammatory lesions as determined by the Investigator or designee.
- Have 10 100 non-inflammatory lesions as determined by the Investigator or designee.
- Be willing to use the test products as instructed for 24 weeks.
- Be willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol.
- Be willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and be able to read, speak, write, understand English and be willing to share personal information and data, as verified by signing a written authorization at the screening.
- Be willing to withhold all facial treatments during the course of the study including botulinum toxin, injectable fillers, microdermabrasion, IPL, peels, facials, laser treatments and tightening treatments. Waxing and threading is allowed but not facial laser hair removal.
- Males must be regular shavers and willing to shave on the day of the study visits (prior to clinic visits).
- Women of child bearing potential must be willing to take a urine pregnancy test prior to study enrollment, at week 24, and when deemed appropriate by the Investigator and/or Sponsor.
- Individuals of child bearing potential must use an acceptable method of contraception throughout the study. Acceptable methods of birth control include:
  - Oral and other system contraceptives. Individuals must be on a stable use for 3 months prior to study enrollment. Individuals on oral contraceptives must not alter their use, including dose or regimen for the duration of the study
  - Double barrier
  - o Bilateral tubal ligation (tubes tied)
  - o Partner vasectomy
  - o Abstinence
- Be willing to follow study requirements and report any changes in health status or medications, side effect symptoms, or reactions immediately.
- Be stable on any medication you are taking for at least 30 days

## YOU CANNOT BE ON THE STUDY

# If you:

- Have been diagnosed with allergies to topical acne products.
- Have a condition and/or disease of the skin that the Investigator deems inappropriate for participation.
- Are a woman who is breastfeeding, pregnant, or planning to become pregnant during the study.
- Have pre-existing or dormant dermatologic conditions on the face (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, severe excoriations etc.) which in the opinion of the Investigator could interfere with the outcome of the study.
- Have a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab,

# THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE
- cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.).
- Have an uncontrolled disease such as asthma, diabetes, hypertension, hyperthyroidism, or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc. at the Investigator's discretion.
- Are currently participating in another facial usage study or have participated in a clinical trial within 4 weeks prior to inclusion into the study.
- Have a history of skin cancer on the face within the past 5 years.
- Have any planned surgeries and/or invasive medical procedures during the course of the study.
- Have started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to study entry or plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study.
- Have facial sunburn or excessive tanned facial skin or are not willing to avoid daily sun exposure on the face and the use of tanning beds or sunless tanning products for the duration of the study.
- Have severe acne, acne conglobata, multiple nodules or cysts (more than 2).
- Are currently taking a natural or prescription testosterone blocker (e.g. saw palmetto, blask cohosh, chaste tree, chasteberry, spironolactone, drospirenone, progestins).
- Are currently on a testosterone booster or prescription testosterone (e.g. DHEA, tribulus, testosterone cypionate, testosterone enanthate, Sustanon, testosterone propionate, testosterone phenylpropriate, Omnadren etc.).
- Are currently taking or have taken within the last 30 days oral or topical prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin (Retin A, Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo.
- Have used oral isotretinoin (Accutane) within the past 6-months.
- Are routinely using (3x a week or more) topical over-the-counter (OTC) acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 14 days of the study entry.
- Are using or have used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study.
- Have excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations as determined by the Investigator or designee.

#### WHAT WILL HAPPEN DURING THE STUDY

#### \*Visit 1: Screening (\* Visit 1 {Screening} AND Visit 2 {Baseline} may be combined into 1 Visit)

#### You will:

- Be given an IRB-approved Informed Consent Form (ICF), to read and sign. You will be given enough time to read the informed consent, and ask questions about the study, and sign 1 copy of this consent form and be given a signed photocopy to keep for your records.
- Be given an eligibility and health questionnaire to complete, and assigned a screening number.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Will be screened by the Investigator or designee to see if you qualify for the study.
- If you do qualify for the study, you will:
  - Take a urine pregnancy test (females of child-bearing potential)

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Have a trained evaluator confirm your eligibility
- o Schedule your next appointment.

#### \*Visit 2: Baseline

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Be screened by the Investigator or designee to see if you still qualify for the study.
- Have your health and eligibility re-reviewed.
- If you still qualify for the study you will:
  - o Be assigned a subject number
  - Have photos taken of your face
  - o Be randomly assigned to receive one of the test products & supporting facial cleanser, moisturizer & facial SPF 30
  - o Be provided verbal and written usage instructions, and a daily diary to record product use
  - o Schedule your next appointment

### **Visits 3, 4 (Week 1, Week 2)**

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and returned to you. At week 2, your diary will be retained by the testing facility and you will be given a new diary
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

#### Visits 5, 6 (Week 6, Week 12)

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and retained. New products will be dispensed as necessary.
- Schedule your next appointment

#### Visit 7 (Week 18)

- Be asked if you have experienced any changes in your health since the previous visit.
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

### **Visit 8 (Week 24)**

- Be asked if you have experienced any changes in your health since the previous visit.
- Take a urine pregnancy test (females of child-bearing potential).

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility.
- Have your product collected, weighed, and retained by the testing facility.

Do not give the study product to other people and keep it out of the reach of children.

#### RISKS OR DISCOMFORTS

If you do not understand what any of these side effects mean, please ask the investigator or study staff to explain these terms to you.

Because the study products are investigational, all of their side effects may not be known. There may be rare and unknown side effects. Some of these may be life threatening.

Possible risks associated with the product are, as with any other cosmetic and OTC products, signs of irritation including:

- Itching
- Burning
- Stinging
- Rash or other allergic reaction

- Tingling
- Scaling/Dryness
- Redness

In some cases, it is possible for a subject to develop allergic reactions to the test material(s). This risk is increased for individuals with a history of allergies, and individuals with asthma and/or a history of hives may also be affected. Symptoms include rash, hives, and itching.

You must tell the Investigator or study staff about all side effects that you have. If you are not honest about your side effects, it may not be safe for you to stay in the study.

### BIRTH CONTROL, DANGERS OF PREGNANCY AND BREASTFEEDING

If you are a female, you must not get pregnant while in this study. The only certain way to not get pregnant is to not have sex. If you are a female and choose to have sex, you must use a type of birth control.

Even if you use birth control during the study, there is a chance you could become pregnant. If you are pregnant or become pregnant during the study, test products or procedures may involve unforeseeable risks to the unborn baby.

A pregnancy test can be wrong. If you become pregnant during the study, stop using the test products and call/inform the Investigator at once.

You cannot be in the study if you are breastfeeding. It is not known whether the test products are safe for breast fed babies. Therefore if you are breastfeeding a child then it may not be safe for you to participate in the study.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### POSSIBLE BENEFITS OF THE STUDY

You will not get any medical benefit from being in this study, and there is no promise that your condition (acne) will get better. It might stay the same or it might get worse. Your participation will provide information that may help others. There may be other marketed products that claim to have similar benefits.

#### OTHER OPTIONS TO PARTICIPATING IN THE STUDY

Since this study is for research only, the only other choice would be not to be in the study.


To participate in this study, you must agree to keep any information relating to the design, identity or use of these test product samples confidential.

On rare occasions, the sponsor may allow the testing company to disclose to you the name of the test products if you are not given this information during the study. This information is typically not provided until the end of the study or after the test products have been released for sale to the public. The study doctor or study staff will notify you if the sponsor allows us to give you this information.

#### DISCLOSURE AGREEMENT

This section explains how personal health information collected about you for the study may be used. Your personal health information includes, but is not limited to, information that was collected for your entry into the study and information that is collected during the study. The purpose of collecting this information is to allow the study staff and the Investigator to conduct the study, to evaluate the sponsor's study products and to analyze the study results.

You may decide not to give permission for the release of your personal health information for the study. In that case, you will not be able to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the sponsor's study products.

People who may inspect your personal and health information includes the Investigator, the Institutional Review Board, IntegReview IRB, FDA and other regulatory authorities from the United States or other countries, the study sponsor and people that work with the sponsor which includes, monitoring committees, contract research organizations, and consultants who have contracts with the company to do the study and review the study results. These reviews are done to check on the quality of the study and also for other purposes allowed by law.

The results of the study may be published in a medical book or journal, or presented at meetings for educational purposes. Neither your name, nor any other personal health information that specifically identifies you, will be used in those materials or presentations.

You may ask the Investigator to see and copy your personal health information related to the study. You may also ask the Investigator to correct any study related information about you that is wrong. You may have to wait until the end of the study to see your study records, so that the study can be organized properly.

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the Investigator at the address below:

Barry T. Reece 3207 Esters Road Irving, Texas 75062

If you cancel your permission after you have started in the study, the study staff and the Investigator will stop collecting your personal health information. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the study.

RCTS, Inc., and the sponsor will make every effort to keep your personal health information private. But after the study staff or the Investigator share your personal health information from the study, federal privacy laws may not keep it private. There might be laws in your state or other federal laws that would protect the privacy of this information.

#### **CONFIDENTIALITY**

Your records of being in this study will be kept private except when ordered by law. The following people will have access to your study records:

- The Investigator
- Sponsor company or research institution [including monitor(s) and auditor(s)]
- Other country, state or federal regulatory agencies
- IntegReview IRB

The Institutional Review Board (IRB), IntegReview, and accrediting agencies may inspect and copy your records, which may have your name on them. Therefore, total confidentiality cannot be guaranteed. If the study results are presented at meetings or printed in publications, your name will not be used.

#### IN CASE OF STUDY RELATED INJURY

Side effects or complications, both foreseeable and unforeseeable, are possible in any research study without any fault to you, the Investigator, the study site, or the study sponsor. If you get hurt or sick as a direct result of being in this study, the sponsor will pay the costs of reasonable medical treatment. To ask questions about this, talk to the Investigator or study staff.

The sponsor's policy does not offer compensation for other expenses. Be aware that your health care payer/insurer might not cover the costs of study-related injuries or illnesses.

Unreimbursed medical expenses not covered by insurance or other third party coverage will be reimbursed by the sponsor for medical treatment for any injury that, in the opinion of the study doctor and the sponsor, is directly caused by the investigational product or by procedures required by the study protocol which would not have been performed as part of your regular medical care.

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### **LEGAL RIGHTS**

You will not lose any of your legal rights by signing this consent form.

#### **CONTACT INFORMATION**

If you have questions, concerns, or complaints about this study or to report a study related injury, contact:

Barry T. Reece 972-871-7578 daytime telephone number 972-841-2916 after hours number (cell phone)

If you are unable to reach anyone at the number(s) listed above and you need medical attention, please go to the nearest emergency room.

If you do not want to talk to the Investigator or study staff, if you have concerns or complaints about the research, or to ask questions about your rights as a study subject you may contact IntegReview. IntegReview's policy indicates that all concerns/complaints are to be submitted in writing for review at a convened IRB meeting to:

| Mailing Address: | OR | Email Address: |
|----------------------------------|----|-----------------------------|
| Chairperson | | integreview@integreview.com |
| IntegReview IRB | | |
| 3815 S. Capital of Texas Highway | | |
| Suite 320 | | |
| Austin, TX 78704 | | |

If you are unable to provide your concerns/complaints in writing or if this is an emergency situation regarding subject safety, contact our office at:

512-326-3001 or toll free at 1-877-562-1589 between 8 a.m. and 5 p.m. Central Time

IntegReview has approved the information in this consent form and has given approval for the Investigator to do the study. This does not mean IntegReview has approved your being in the study. You must consider the information in this consent form for yourself and decide if you want to be in this study.

### PAYMENT FOR BEING IN THE STUDY

You may receive up to \$600.00 for being in the study. You will be paid per completed visit as follows:

| Visit | Compensation (amount) |
|--------------------|-----------------------|
| Visit 1: Screening | \$25.00 |
| Visit 2: Baseline | \$50.00 |
| Visit 3: Week 1 | \$50.00 |
| Visit 4: Week 2 | \$50.00 |
| Visit 5: Week 6 | \$50.00 |

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

**VERSION CONTROL** 

clw/master: 2-17-16 snb/site: 2-25-16

| Visit 6: Week 12 | \$50.00 |
|----------------------------------|----------|
| Visit 7: Week 18 | \$50.00 |
| Visit 8: Week 24 | \$50.00 |
| Bonus for completing all visits: | \$225.00 |

If you choose to leave or are withdrawn from the study for any reason before finishing all visits you will be paid for each completed visit. You will receive payment on the originally scheduled last day of the study.

If you are paid \$600.00 or more by RCTS, Inc., in a calendar year, those payments will be reported to the Internal Revenue Service via form 1099-MISC. As required by tax laws, if you withhold your social security number, RCTS, Inc. is required to withhold 28% of your payment for tax purposes. In this case a form 1099-MISC will be sent to you reporting your withholding.

#### **VOLUNTEERING TO BE IN THE STUDY**

It is your choice if you want to be in the study. No one can force you to be in the study. You may not want to be in this study or you may leave the study at any time without penalty or loss of benefits to which you are otherwise entitled.

The Investigator, the sponsor company, or IntegReview may take you out of the study without your permission, at any time, for the following reasons:

- If you do not follow the Investigator's instructions
- If we find out you should not be in the study
- If the study is stopped
- If it becomes harmful to your health

If you leave the study or if you are taken out of the study, you may be asked to return for a final visit to have some end of study evaluations or tests. If information generated from this study is published or presented, your identity will not be revealed. If you leave the study, no more information about you will be collected for this study. However, all of the information you gave us before you left the study will still be used.

#### **NEW FINDINGS**

If there is new information or any significant new findings that could relate to your willingness to continue participation we will tell you. You can then decide if you still want to be in the study.

#### THE REASON FOR INSTITUTIONAL REVIEW BOARDS AND INFORMED CONSENT

### What is a consent form?

The informed consent document contains information required by federal regulations. The informed consent document must be approved by an Institutional Review Board (IRB).

#### What is an Institutional Review Board (IRB)?

An Institutional Review Board (IRB) is a group of people that reviews research studies. The main goal of this review is to protect the rights and well being of the human subjects participating in research studies.

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

**VERSION CONTROL** 

clw/master: 2-17-16 snb/site: 2-25-16

### IntegReview, the IRB for this study

IntegReview is an IRB whose board members provide IRB services across the United States, Canada, Japan and Latin America.

To meet requirements of the law, the IntegReview Boards currently include:

- Doctors
- Pharmacists
- Nurses
- Toxicologists (people who study the harmful effects of chemicals)
- Other specialists
- Others who do not have a background in science/medicine

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### AGREEMENT TO BE IN THE STUDY

This consent form contains important information to help you decide if you want to be in the study. If you have any questions that are not answered in this consent form, ask one of the study staff.

| Pleas | e answer <b>YES</b> or <b>NO</b> to the following questions: | |
|---|---|---|
| A. | . Is this document in a language you understand? | |
| B. | Do you understand the information in this consent form? | |
| C. | . Have you been given enough time to ask questions and talk about the study? | |
| D. | D. Have all of your questions been answered to your satisfaction? | |
| E. | . Do you think you received enough information about the study? | |
| F. | Do you volunteer to be in this study of your own free will and without being pressured by the Investigator or study staff? | |
| G. | G. Do you know that you can leave the study at any time without giving a reason and without affecting your health care? | |
| Н. | Do you know that your health records from this study may be reviewed by the sponsor company and by government authorities? | |
| I. | Do you know that you cannot be in another study while you are in this study? | |
| | IF YOU ANSWERED "NO" TO ANY OF THE ABOVE QUESTION OR YOU ARE UNABLE TO ANSWER ANY OF THE ABOVE QUEST YOU SHOULD NOT SIGN THIS CONSENT FORM. | |
| Print | ed Name of Adult Study Subject | |
| Signa | ature of Adult Study Subject | Date |
| Print | ed Name of Person Explaining Consent Form | |
| Signa | ature of Person Explaining Consent Form | Date |
| You | will be given a signed and dated copy of this consent form to keep. | |

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

### **Authorization and Photographic Release Form**

I hereby for good and valuable consideration grant to RCTS, Inc., the study sponsor and their respective affiliates, agencies, agents, employees, and assigns (collectively, "Authorized Entities"), the unrestricted, royalty free, irrevocable and perpetual right and permission to reproduce, distribute, broadcast and/or otherwise use for advertising and other commercial/noncommercial purposes: (i) my name, likeness, image, video, and any other biographical or personal information ("Personal Content"); and (ii) any statement or endorsement, or any portions thereof ("Testimonial(s)"), made by me relating to the study sponsor's products ("Products"), in any and all media now known or later developed, worldwide in perpetuity, without further compensation or approval by me.

I hereby assign to the Authorized Entities all of my world-wide right, title and interest, including my copyright interests and all renewals, reissues and extensions thereof, in and to the Personal Content and Testimonial(s), including without limitation, any photographic portraits, sound recordings and video performances of and/or by me in connection with the Personal Content and/or Testimonial(s).

I am at least 21 years of age, and competent to contract in my own name. I have read and understand this

| Authorization and Release. | |
|---|---|
| Printed Name of Adult Study Subject | |
| Signature of Adult Study Subject | Date |
| Printed Name of Person Explaining Release Form | |
| Signature of Person Explaining Release Form | Date |
| Copy of consent form given to subject on (date) | by (initials) |
| You will be given a signed and dated copy of this consent form | to keep. |

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

# AUTHORIZATION TO USE AND DISCLOSE PERSONAL HEALTH INFORMATION FOR RESEARCH

THIS SECTION DESCRIBES YOUR RIGHTS AND HOW PERSONAL HEALTH INFORMATION COLLECTED ABOUT YOU DURING THIS STUDY MAY BE USED AND DISCLOSED AND HOW YOU CAN GET ACCESS TO THIS INFORMATION. PLEASE REVIEW IT CAREFULLY.

The United States government has issued a privacy rule to protect the privacy rights of patients. This rule was issued under a law called the Health Insurance Portability and Accountability Act of 1996 (HIPAA). The Privacy Rule is designed to protect the confidentiality of your personal health information. The document you are reading, called an "Authorization," describes your rights and explains how your health information will be used and disclosed (shared).

Federal law requires hospitals, researchers and health care providers to protect the privacy of information that identifies you and relates to your past, present and future physical and mental health or conditions.

All information collected during the study will be retained by the study doctor and the Study Sponsor, except as required by law. Information from this study will be given to the sponsor. "Sponsor" includes any persons or companies, which are contracted by the sponsor to have access to the research information during and after the study. The information will also be given to the U.S. Food and Drug Administration (FDA). Study records which identify you and the consent form signed by you will be inspected and/or copied for research or regulatory purposes by:

- Sponsor
- Agents for the sponsor
- The US Food and Drug Administration (FDA)
- Department of Health and Human Services (DHHS) agencies
- IntegReview IRB

Because of the need to release information to these parties, absolute confidentiality cannot be guaranteed. The results of this research study may be presented at meetings or in publications; however, your identity will not be disclosed in those presentations.

For purposes of study reporting, you will be identified by your initials and code numbers only. However, your name, date of birth, address, and phone number will be kept on record by the study doctor in case you need to be contacted in the future about this study.

After your personal health information is disclosed to the Study Sponsor, the results of the study may be reanalyzed at a later date and may be combined with the results of other studies. The Study Sponsor and people who work with the Study Sponsor may use the results of this study for other research purposes, including:

- Developing a better understanding of the disease;
- Improving the design of future actual use trials

After the study staff or the study doctor discloses your personal health information to others, it could be re-disclosed and no longer protected by federal privacy laws.

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you do not withdraw this Authorization in writing, it will remain in effect indefinitely. Your study doctor will keep this Authorization for at least 6 years. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the study doctor at the address below:

RCTS, Inc., 3207 Esters Road Irving, Texas, 75062

You have the right to see and get a copy of your records related to the study for as long as the study doctor has this information. However, by signing this Authorization you agree that you might not be able to review or receive some of your records related to the study until after the study has been completed.

If you cancel your permission after you have started in the study, the study staff and the study doctor will stop collecting your personal health information unless the information concerns an adverse event (a bad effect) related to the study. If an adverse event occurs, your entire medical record may be reviewed. All information that has already been collected for study purposes, and any new information about an adverse event related to the study, will be sent to the study sponsor. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the study doctor would not be able to collect the information needed to evaluate the study results.

If you withdraw from the study but do not withdraw your Authorization, new personal health information may be collected until this study ends.

You may decide not to give permission for the release of your personal health information for this study. In that case, you will not be able to participate. This is because the study staff and study doctor would not be able to collect the information needed to evaluate the study results.

At the completion of the study, you have the right to access your protected health information that is created during this research study that relates to your treatment or to payment, provided such information is not exempted under certain laws and regulations. To request this information, please contact the study doctor at the address listed above.

### **Your Right to Access Health Information**

Subject to certain exceptions prescribed by law, you have a right to request access to the health information that we hold about you and to request changes if your health information is incorrect or incomplete. Any request for access or corrections should be made to the principal doctor conducting this study.

Your records obtained while you are in this trial, as well as related health records, will remain strictly confidential at all times. However, these will need to be made available to others working on the Sponsor's behalf, the Independent Ethics Committee members and Medicines Regulatory Authorities.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

By signing the consent form you agree to this access for the current trial and any further research that may be done. However, the Sponsor will take steps to protect your personal information and will not include your name on any sponsor forms, reports, publications, or in any future disclosures. If you withdraw from the study, we will no longer collect your personal information, but we may need to continue to use information already collected.

Personal data which may be sensitive (e.g., date of birth) will be collected and processed, but only for research purposes in connection with this trial.

The trial data will be sent around the world, but you will not be referred to by name or identified in any report or publication nor could the data be traced back to you. Your data may be transferred to a country that does not have the same level of personal data protection as within the United States. However, The Sponsor maintains high standards of confidentiality and protection.

The Sponsor (who will control the use of the data) will take steps to ensure your personal data is protected.

By taking part in this trial you agree not to restrict the use of any data even if you withdraw from the trial and agree to the transfer of your personal data to other Sponsor companies and to Medicines Regulatory Authorities both within and outside of Europe.

| Printed Name of Adult Study Subject | |
|-------------------------------------|------|
| Signature of Adult Study Subject | Date |

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

# INFORMED CONSENT DOCUMENT AGREEMENT TO BE IN A RESEARCH STUDY

NAME OF TESTING COMPANY: RCTS, Inc.,

NUMBER AND TITLE OF STUDY: C16-CD020 (GLI.04.SPR.US10354); "A Multi-

Center Clinical Trial to Evaluate the Efficacy of

Two Acne Treatments"

NAME OF PERSON IN CHARGE OF THE

**RESEARCH STUDY (INVESTIGATOR):** Barry T. Reece, M.S., M.B.A.

Principal Investigator

**MEDICAL INVESTIGATORS:** Raymond L. Garcia, M.D.

**Board Certified Dermatologist** 

Gene Ream, M.D.

**Board Certified Dermatologist** 

TELEPHONE NUMBER(S), DAYTIME: 972-871-7578

**AFTER HOURS:** 972-841-2916 (Emergencies Only, Cell Phone

Number)

#### INTRODUCTION

You are being invited to volunteer for a clinical research study. You must read and sign this form before you agree to take part in this study. This form will give you more information about this study. Please ask as many questions as you need to before you decide if you want to be in the study. You should not sign this form if you have any questions that have not been answered.

RCTS, Inc., a contract research organization, is being paid by the sponsor (the company paying for this study) to conduct this research study.

You must be honest with the Investigator about your health history or it may not be safe for you to be in this study.

### **PURPOSE OF THE STUDY**

The purpose of this study is to evaluate the efficiency of 2 acne treatments for 24 weeks of use in adult men and women with mild to moderate facial acne, at least 5 inflammatory lesions, and at least 10 - 100 non-inflammatory lesions.

#### HOW LONG THE STUDY WILL LAST AND HOW MANY PEOPLE WILL BE IN THE STUDY

This study will last 24 weeks and have up to 8 visits. At least 100 subjects, men and women between the ages of 21-45, are expected to complete this study, with at least 50 subjects completed per cell.

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### TO BE IN THIS STUDY

#### You must:

- Be a man or woman age 21 to 45 years at the time of enrollment.
- Have mild to moderate acne on the face as determined by the Investigator or designee.
- Have at least 5 inflammatory lesions as determined by the Investigator or designee.
- Have 10 100 non-inflammatory lesions as determined by the Investigator or designee.
- Be willing to use the test products as instructed for 24 weeks.
- Be willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol.
- Be willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and be able to read, speak, write, understand English and be willing to share personal information and data, as verified by signing a written authorization at the screening.
- Be willing to withhold all facial treatments during the course of the study including botulinum toxin, injectable fillers, microdermabrasion, IPL, peels, facials, laser treatments and tightening treatments. Waxing and threading is allowed but not facial laser hair removal.
- Males must be regular shavers and willing to shave on the day of the study visits (prior to clinic visits).
- Women of child bearing potential must be willing to take a urine pregnancy test prior to study enrollment, at week 24, and when deemed appropriate by the Investigator and/or Sponsor.
- Individuals of child bearing potential must use an acceptable method of contraception throughout the study. Acceptable methods of birth control include:
  - Oral and other system contraceptives. Individuals must be on a stable use for 3 months prior to study enrollment. Individuals on oral contraceptives must not alter their use, including dose or regimen for the duration of the study
  - Double barrier
  - o Bilateral tubal ligation (tubes tied)
  - o Partner vasectomy
  - o Abstinence
- Be willing to follow study requirements and report any changes in health status or medications, side effect symptoms, or reactions immediately.
- Be stable on any medication you are taking for at least 30 days

#### YOU CANNOT BE ON THE STUDY

### If you:

- Have been diagnosed with allergies to topical acne products.
- Have a condition and/or disease of the skin that the Investigator deems inappropriate for participation.
- Are a woman who is breastfeeding, pregnant, or planning to become pregnant during the study.
- Have pre-existing or dormant dermatologic conditions on the face (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, severe excoriations etc.) which in the opinion of the Investigator could interfere with the outcome of the study.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- Have a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.).
- Have an uncontrolled disease such as asthma, diabetes, hypertension, hyperthyroidism, or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc. at the Investigator's discretion.
- Are currently participating in another facial usage study or have participated in a clinical trial within 4 weeks prior to inclusion into the study.
- Have a history of skin cancer on the face within the past 5 years.
- Have any planned surgeries and/or invasive medical procedures during the course of the study.
- Have started hormone replacement therapies (HRT) or hormones for birth control less than 3 months
  prior to study entry or plan on starting, stopping, or changing doses of HRT or hormones for birth
  control during the study.
- Have facial sunburn or excessive tanned facial skin or are not willing to avoid daily sun exposure on the face and the use of tanning beds or sunless tanning products for the duration of the study.
- Have severe acne, acne conglobata, multiple nodules or cysts (more than 2).
- Are currently taking a natural or prescription testosterone blocker (e.g. saw palmetto, blask cohosh, chaste tree, chasteberry, spironolactone, drospirenone, progestins).
- Are currently on a testosterone booster or prescription testosterone (e.g. DHEA, tribulus, testosterone cypionate, testosterone enanthate, Sustanon, testosterone propionate, testosterone phenylpropriate, Omnadren etc.).
- Are currently taking or have taken within the last 30 days oral or topical prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin (Retin A, Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo.
- Have used oral isotretinoin (Accutane) within the past 6-months.
- Are routinely using (3x a week or more) topical over-the-counter (OTC) acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 14 days of the study entry.
- Are using or have used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study.
- Have excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations as determined by the Investigator or designee.

#### WHAT WILL HAPPEN DURING THE STUDY

### \*Visit 1: Screening (\* Visit 1 {Screening} AND Visit 2 {Baseline} may be combined into 1 Visit)

#### You will:

- Be given an IRB-approved Informed Consent Form (ICF), to read and sign. You will be given enough time to read the informed consent, and ask questions about the study, and sign 1 copy of this consent form and be given a signed photocopy to keep for your records.
- Be given an eligibility and health questionnaire to complete, and assigned a screening number.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Will be screened by the Investigator or designee to see if you qualify for the study.

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

- If you do qualify for the study, you will:
  - o Take a urine pregnancy test (females of child-bearing potential)
  - o Have a trained evaluator confirm your eligibility
  - o Schedule your next appointment.

#### \*Visit 2: Baseline

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Be screened by the Investigator or designee to see if you still qualify for the study.
- Have your health and eligibility re-reviewed.
- If you still qualify for the study you will:
  - o Be assigned a subject number
  - Have photos taken of your face
  - o Be randomly assigned to receive one of the test products & supporting facial cleanser, moisturizer & facial SPF 30
  - o Be provided verbal and written usage instructions, and a daily diary to record product use
  - Schedule your next appointment

### Visits 3, 4 (Week 1, Week 2)

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and returned to you. At week 2, your diary will be retained by the testing facility and you will be given a new diary
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

#### Visits 5, 6 (Week 6, Week 12)

- Be asked if you have experienced any changes in your health since the previous visit.
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and retained. New products will be dispensed as necessary.
- Schedule your next appointment

### **Visit 7 (Week 18)**

- Be asked if you have experienced any changes in your health since the previous visit.
- Have your diary collected and reviewed for compliance, and retained by the testing facility and you will be given a new diary.
- Have your product collected, weighed, and returned to you
- Schedule your next appointment

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### Visit 8 (Week 24)

- Be asked if you have experienced any changes in your health since the previous visit.
- Take a urine pregnancy test (females of child-bearing potential).
- Will acclimate for 15 minutes in a room at 68-75°F and 35-65% humidity.
- Have your face examined by the Investigator or designee
- Have photos taken of your face
- Complete a self-assessment questionnaire
- Have your diary collected and reviewed for compliance, and retained by the testing facility.
- Have your product collected, weighed, and retained by the testing facility.

Do not give the study product to other people and keep it out of the reach of children.

#### RISKS OR DISCOMFORTS

If you do not understand what any of these side effects mean, please ask the investigator or study staff to explain these terms to you.

Because the study products are investigational, all of their side effects may not be known. There may be rare and unknown side effects. Some of these may be life threatening.

Possible risks associated with the product are, as with any other cosmetic and OTC products, signs of irritation including:

- Itching
- Burning
- Stinging
- Rash or other allergic reaction

- Tingling
- Scaling/Dryness
- Redness

In some cases, it is possible for a subject to develop allergic reactions to the test material(s). This risk is increased for individuals with a history of allergies, and individuals with asthma and/or a history of hives may also be affected. Symptoms include rash, hives, and itching.

You must tell the Investigator or study staff about all side effects that you have. If you are not honest about your side effects, it may not be safe for you to stay in the study.

### BIRTH CONTROL, DANGERS OF PREGNANCY AND BREASTFEEDING

If you are a female, you must not get pregnant while in this study. The only certain way to not get pregnant is to not have sex. If you are a female and choose to have sex, you must use a type of birth control.

Even if you use birth control during the study, there is a chance you could become pregnant. If you are pregnant or become pregnant during the study, test products or procedures may involve unforeseeable risks to the unborn baby.

A pregnancy test can be wrong. If you become pregnant during the study, stop using the test products and call/inform the Investigator at once.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

You cannot be in the study if you are breastfeeding. It is not known whether the test products are safe for breast fed babies. Therefore if you are breastfeeding a child then it may not be safe for you to participate in the study.

#### POSSIBLE BENEFITS OF THE STUDY

You will not get any medical benefit from being in this study, and there is no promise that your condition (acne) will get better. It might stay the same or it might get worse. Your participation will provide information that may help others. There may be other marketed products that claim to have similar benefits.

#### OTHER OPTIONS TO PARTICIPATING IN THE STUDY

Since this study is for research only, the only other choice would be not to be in the study.


To participate in this study, you must agree to keep any information relating to the design, identity or use of these test product samples confidential.

On rare occasions, the sponsor may allow the testing company to disclose to you the name of the test products if you are not given this information during the study. This information is typically not provided until the end of the study or after the test products have been released for sale to the public. The study doctor or study staff will notify you if the sponsor allows us to give you this information.

#### **DISCLOSURE AGREEMENT**

This section explains how personal health information collected about you for the study may be used. Your personal health information includes, but is not limited to, information that was collected for your entry into the study and information that is collected during the study. The purpose of collecting this information is to allow the study staff and the Investigator to conduct the study, to evaluate the sponsor's study products and to analyze the study results.

You may decide not to give permission for the release of your personal health information for the study. In that case, you will not be able to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the sponsor's study products.

People who may inspect your personal and health information includes the Investigator, the Institutional Review Board, IntegReview IRB, FDA and other regulatory authorities from the United States or other countries, the study sponsor and people that work with the sponsor which includes, monitoring committees, contract research organizations, and consultants who have contracts with the company to do the study and review the study results. These reviews are done to check on the quality of the study and also for other purposes allowed by law.

The results of the study may be published in a medical book or journal, or presented at meetings for educational purposes. Neither your name, nor any other personal health information that specifically identifies you, will be used in those materials or presentations.

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

You may ask the Investigator to see and copy your personal health information related to the study. You may also ask the Investigator to correct any study related information about you that is wrong. You may have to wait until the end of the study to see your study records, so that the study can be organized properly.

This permission to share your personal health information for this study does not have an expiration date. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the Investigator at the address below:

Barry T. Reece 3207 Esters Road Irving, Texas 75062

If you cancel your permission after you have started in the study, the study staff and the Investigator will stop collecting your personal health information. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the Investigator would not be able to collect the information needed to evaluate the study.

RCTS, Inc., and the sponsor will make every effort to keep your personal health information private. But after the study staff or the Investigator share your personal health information from the study, federal privacy laws may not keep it private. There might be laws in your state or other federal laws that would protect the privacy of this information.

### **CONFIDENTIALITY**

Your records of being in this study will be kept private except when ordered by law. The following people will have access to your study records:

- The Investigator
- Sponsor company or research institution [including monitor(s) and auditor(s)]
- Other country, state or federal regulatory agencies
- IntegReview IRB

The Institutional Review Board (IRB), IntegReview, and accrediting agencies may inspect and copy your records, which may have your name on them. Therefore, total confidentiality cannot be guaranteed. If the study results are presented at meetings or printed in publications, your name will not be used.

#### IN CASE OF STUDY RELATED INJURY

Side effects or complications, both foreseeable and unforeseeable, are possible in any research study without any fault to you, the Investigator, the study site, or the study sponsor. If you get hurt or sick as a direct result of being in this study, the sponsor will pay the costs of reasonable medical treatment. To ask questions about this, talk to the Investigator or study staff.

The sponsor's policy does not offer compensation for other expenses. Be aware that your health care payer/insurer might not cover the costs of study-related injuries or illnesses.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

Unreimbursed medical expenses not covered by insurance or other third party coverage will be reimbursed by the sponsor for medical treatment for any injury that, in the opinion of the study doctor and the sponsor, is directly caused by the investigational product or by procedures required by the study protocol which would not have been performed as part of your regular medical care.

#### LEGAL RIGHTS

You will not lose any of your legal rights by signing this consent form.

#### **CONTACT INFORMATION**

If you have questions, concerns, or complaints about this study or to report a study related injury, contact:

Barry T. Reece 972-871-7578 daytime telephone number 972-841-2916 after hours number (cell phone)

If you are unable to reach anyone at the number(s) listed above and you need medical attention, please go to the nearest emergency room.

If you do not want to talk to the Investigator or study staff, if you have concerns or complaints about the research, or to ask questions about your rights as a study subject you may contact IntegReview. IntegReview's policy indicates that all concerns/complaints are to be submitted in writing for review at a convened IRB meeting to:

| Mailing Address: | OR | Email Address: |
|----------------------------------|----|-----------------------------|
| Chairperson | | integreview@integreview.com |
| IntegReview IRB | | |
| 3815 S. Capital of Texas Highway | | |
| Suite 320 | | |
| Austin, TX 78704 | | |

If you are unable to provide your concerns/complaints in writing or if this is an emergency situation regarding subject safety, contact our office at:

512-326-3001 or toll free at 1-877-562-1589 between 8 a.m. and 5 p.m. Central Time

IntegReview has approved the information in this consent form and has given approval for the Investigator to do the study. This does not mean IntegReview has approved your being in the study. You must consider the information in this consent form for yourself and decide if you want to be in this study.

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### PAYMENT FOR BEING IN THE STUDY

You may receive up to \$600.00 for being in the study. You will be paid per completed visit as follows:

| Visit | Compensation (amount) |
|----------------------------------|-----------------------|
| Visit 1: Screening | \$25.00 |
| Visit 2: Baseline | \$50.00 |
| Visit 3: Week 1 | \$50.00 |
| Visit 4: Week 2 | \$50.00 |
| Visit 5: Week 6 | \$50.00 |
| Visit 6: Week 12 | \$50.00 |
| Visit 7: Week 18 | \$50.00 |
| Visit 8: Week 24 | \$50.00 |
| Bonus for completing all visits: | \$225.00 |

If you choose to leave or are withdrawn from the study for any reason before finishing all visits you will be paid for each completed visit. You will receive payment on the originally scheduled last day of the study.

If you are paid \$600.00 or more by RCTS, Inc., in a calendar year, those payments will be reported to the Internal Revenue Service via form 1099-MISC. As required by tax laws, if you withhold your social security number, RCTS, Inc. is required to withhold 28% of your payment for tax purposes. In this case a form 1099-MISC will be sent to you reporting your withholding.

#### **VOLUNTEERING TO BE IN THE STUDY**

It is your choice if you want to be in the study. No one can force you to be in the study. You may not want to be in this study or you may leave the study at any time without penalty or loss of benefits to which you are otherwise entitled.

The Investigator, the sponsor company, or IntegReview may take you out of the study without your permission, at any time, for the following reasons:

- If you do not follow the Investigator's instructions
- If we find out you should not be in the study
- If the study is stopped
- If it becomes harmful to your health

If you leave the study or if you are taken out of the study, you may be asked to return for a final visit to have some end of study evaluations or tests. If information generated from this study is published or presented, your identity will not be revealed. If you leave the study, no more information about you will be collected for this study. However, all of the information you gave us before you left the study will still be used.

#### **NEW FINDINGS**

If there is new information or any significant new findings that could relate to your willingness to continue participation we will tell you. You can then decide if you still want to be in the study.

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### THE REASON FOR INSTITUTIONAL REVIEW BOARDS AND INFORMED CONSENT

### What is a consent form?

The informed consent document contains information required by federal regulations. The informed consent document must be approved by an Institutional Review Board (IRB).

#### What is an Institutional Review Board (IRB)?

An Institutional Review Board (IRB) is a group of people that reviews research studies. The main goal of this review is to protect the rights and well being of the human subjects participating in research studies. *IntegReview, the IRB for this study* 

IntegReview is an IRB whose board members provide IRB services across the United States, Canada, Japan and Latin America.

To meet requirements of the law, the IntegReview Boards currently include:

- Doctors
- Pharmacists
- Nurses
- Toxicologists (people who study the harmful effects of chemicals)
- Other specialists
- Others who do not have a background in science/medicine

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

#### AGREEMENT TO BE IN THE STUDY

This consent form contains important information to help you decide if you want to be in the study. If you have any questions that are not answered in this consent form, ask one of the study staff.

| Pleas | se answer YES or NO to the following questions: | |
|---|---|---|
| A. Is this document in a language you understand? | | |
| B. | B. Do you understand the information in this consent form? | |
| C. | C. Have you been given enough time to ask questions and talk about the study? | |
| D. | Have all of your questions been answered to your satisfaction? | |
| E. | Do you think you received enough information about the study? | |
| F. | Do you volunteer to be in this study of your own free will and without being pressured by the Investigator or study staff? | g<br> |
| G. | Do you know that you can leave the study at any time without giving a reason and without affecting your health care? | |
| Н. | Do you know that your health records from this study may be reviewed by the sponsor company and by government authorities? | |
| I. | Do you know that you cannot be in another study while you are in this study | y? |
| | IF YOU ANSWERED "NO" TO ANY OF THE ABOVE QUEST<br>OR YOU ARE UNABLE TO ANSWER ANY OF THE ABOVE QU<br>YOU SHOULD NOT SIGN THIS CONSENT FORM. | |
| Print | ed Name of Adult Study Subject | |
| Signa | ature of Adult Study Subject | Date |
| Print | ed Name of Person Explaining Consent Form | |
| Signa | ature of Person Explaining Consent Form | Date |
| You | will be given a signed and dated copy of this consent form to keep. | |

### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

### **Authorization and Photographic Release Form**

Authorization and Release

I hereby for good and valuable consideration grant to RCTS, Inc., the study sponsor and their respective affiliates, agencies, agents, employees, and assigns (collectively, "Authorized Entities"), the unrestricted, royalty free, irrevocable and perpetual right and permission to reproduce, distribute, broadcast and/or otherwise use for advertising and other commercial/noncommercial purposes: (i) my name, likeness, image, video, and any other biographical or personal information ("Personal Content"); and (ii) any statement or endorsement, or any portions thereof ("Testimonial(s)"), made by me relating to the study sponsor's products ("Products"), in any and all media now known or later developed, worldwide in perpetuity, without further compensation or approval by me.

I hereby assign to the Authorized Entities all of my world-wide right, title and interest, including my copyright interests and all renewals, reissues and extensions thereof, in and to the Personal Content and Testimonial(s), including without limitation, any photographic portraits, sound recordings and video performances of and/or by me in connection with the Personal Content and/or Testimonial(s).

I am at least 21 years of age, and competent to contract in my own name. I have read and understand this

| Printed Name of Adult Study Subject | |
|---------------------------------------------------------|------------|
| Signature of Adult Study Subject | Date |
| Dried I Manage Character Containing Dalacter Containing | |
| Printed Name of Person Explaining Release Form | |
| Signature of Person Explaining Release Form | Date |
| Copy of consent form given to subject on (date) by | (initials) |

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

You will be given a signed and dated copy of this consent form to keep.

# AUTHORIZATION TO USE AND DISCLOSE PERSONAL HEALTH INFORMATION FOR RESEARCH

THIS SECTION DESCRIBES YOUR RIGHTS AND HOW PERSONAL HEALTH INFORMATION COLLECTED ABOUT YOU DURING THIS STUDY MAY BE USED AND DISCLOSED AND HOW YOU CAN GET ACCESS TO THIS INFORMATION. PLEASE REVIEW IT CAREFULLY.

The United States government has issued a privacy rule to protect the privacy rights of patients. This rule was issued under a law called the Health Insurance Portability and Accountability Act of 1996 (HIPAA). The Privacy Rule is designed to protect the confidentiality of your personal health information. The document you are reading, called an "Authorization," describes your rights and explains how your health information will be used and disclosed (shared).

Federal law requires hospitals, researchers and health care providers to protect the privacy of information that identifies you and relates to your past, present and future physical and mental health or conditions.

All information collected during the study will be retained by the study doctor and the Study Sponsor, except as required by law. Information from this study will be given to the sponsor. "Sponsor" includes any persons or companies, which are contracted by the sponsor to have access to the research information during and after the study. The information will also be given to the U.S. Food and Drug Administration (FDA). Study records which identify you and the consent form signed by you will be inspected and/or copied for research or regulatory purposes by:

- Sponsor
- Agents for the sponsor
- The US Food and Drug Administration (FDA)
- Department of Health and Human Services (DHHS) agencies
- IntegReview IRB

Because of the need to release information to these parties, absolute confidentiality cannot be guaranteed. The results of this research study may be presented at meetings or in publications; however, your identity will not be disclosed in those presentations.

For purposes of study reporting, you will be identified by your initials and code numbers only. However, your name, date of birth, address, and phone number will be kept on record by the study doctor in case you need to be contacted in the future about this study.

After your personal health information is disclosed to the Study Sponsor, the results of the study may be reanalyzed at a later date and may be combined with the results of other studies. The Study Sponsor and people who work with the Study Sponsor may use the results of this study for other research purposes, including:

- Developing a better understanding of the disease;
- Improving the design of future actual use trials

After the study staff or the study doctor discloses your personal health information to others, it could be re-disclosed and no longer protected by federal privacy laws.

#### THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

This permission to share your personal health information for this study does not have an expiration date. If you do not withdraw this Authorization in writing, it will remain in effect indefinitely. Your study doctor will keep this Authorization for at least 6 years. If you no longer want to share your personal health information, you may cancel your permission at any time by writing to the study staff and/or the study doctor at the address below:

RCTS, Inc., 3207 Esters Road Irving, Texas, 75062

You have the right to see and get a copy of your records related to the study for as long as the study doctor has this information. However, by signing this Authorization you agree that you might not be able to review or receive some of your records related to the study until after the study has been completed.

If you cancel your permission after you have started in the study, the study staff and the study doctor will stop collecting your personal health information unless the information concerns an adverse event (a bad effect) related to the study. If an adverse event occurs, your entire medical record may be reviewed. All information that has already been collected for study purposes, and any new information about an adverse event related to the study, will be sent to the study sponsor. Although they will stop collecting new information about you, they will need to use the information they have already collected to evaluate the study results. If you start the study and then cancel your permission, you will not be able to continue to participate in the study. This is because the study staff and/or the study doctor would not be able to collect the information needed to evaluate the study results.

If you withdraw from the study but do not withdraw your Authorization, new personal health information may be collected until this study ends.

You may decide not to give permission for the release of your personal health information for this study. In that case, you will not be able to participate. This is because the study staff and study doctor would not be able to collect the information needed to evaluate the study results.

At the completion of the study, you have the right to access your protected health information that is created during this research study that relates to your treatment or to payment, provided such information is not exempted under certain laws and regulations. To request this information, please contact the study doctor at the address listed above.

### **Your Right to Access Health Information**

Subject to certain exceptions prescribed by law, you have a right to request access to the health information that we hold about you and to request changes if your health information is incorrect or incomplete. Any request for access or corrections should be made to the principal doctor conducting this study.

Your records obtained while you are in this trial, as well as related health records, will remain strictly confidential at all times. However, these will need to be made available to others working on the Sponsor's behalf, the Independent Ethics Committee members and Medicines Regulatory Authorities.

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

By signing the consent form you agree to this access for the current trial and any further research that may be done. However, the Sponsor will take steps to protect your personal information and will not include your name on any sponsor forms, reports, publications, or in any future disclosures. If you withdraw from the study, we will no longer collect your personal information, but we may need to continue to use information already collected.

Personal data which may be sensitive (e.g., date of birth) will be collected and processed, but only for research purposes in connection with this trial.

The trial data will be sent around the world, but you will not be referred to by name or identified in any report or publication nor could the data be traced back to you. Your data may be transferred to a country that does not have the same level of personal data protection as within the United States. However, The Sponsor maintains high standards of confidentiality and protection.

The Sponsor (who will control the use of the data) will take steps to ensure your personal data is protected.

By taking part in this trial you agree not to restrict the use of any data even if you withdraw from the trial and agree to the transfer of your personal data to other Sponsor companies and to Medicines Regulatory Authorities both within and outside of Europe.

| Printed Name of Adult Study Subject | |
|-------------------------------------|------|
| Signature of Adult Study Subject | Date |

## THIS IS AN IMPORTANT DOCUMENT - KEEP FOR FUTURE REFERENCE

| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |

# Visit 1 –Baseline (Day 1)

| 2. F<br>2. F<br>4. F<br>5. Is<br>6. F<br>7. Is<br>8. Is | Is a man or woman between the ages of 21 and 45 years of age at the time of enrollment. Has mild to moderate acne (score of 2-3 on FDA Investigator's Global Assessment Scale) on the face. Have at least 5 inflammatory lesions. Have 10 – 100 non-inflammatory lesions. Is willing to use the test products as instructed for 24 weeks. Has a Fitzpatrick skin type I-VI Is willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol. Is willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and is able to read, speak, write, understand English and is willing to share personal | Yes | No |
|---|---|---|---|
| 3. H<br>4. H<br>5. H<br>6. H<br>7. H<br>8. H<br>r | Assessment Scale) on the face. Have at least 5 inflammatory lesions. Have 10 – 100 non-inflammatory lesions. Is willing to use the test products as instructed for 24 weeks. Has a Fitzpatrick skin type I-VI Is willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol. Is willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and is able to | | |
| 4. F<br>5. I:<br>6. F<br>7. I:<br>8. I:<br>F | Have 10 – 100 non-inflammatory lesions. Is willing to use the test products as instructed for 24 weeks. Has a Fitzpatrick skin type I-VI Is willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol. Is willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and is able to | | |
| 5. I: 6. F 7. I: 8. I: | Is willing to use the test products as instructed for 24 weeks. Has a Fitzpatrick skin type I-VI Is willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol. Is willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and is able to | | |
| 6. F<br>7. II<br>8. II<br>6. F<br>7. II | Has a Fitzpatrick skin type I-VI Is willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol. Is willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and is able to | | |
| 7. l: | Is willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol. Is willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and is able to | | |
| 8. I:<br>F<br>r<br>ii | procedural requirements of the clinical trial protocol. Is willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and is able to | | |
| F<br>r<br>ii | Health Insurance Portability and Accountability Act (HIPAA), and is able to | | |
| 5 | information and data, as verified by signing a written authorization at the screening | | |
| iı<br>p | Is willing to withhold all facial treatments during the course of the study including botulinum toxin, injectable fillers, microdermabrasion, IPL, peels, facials, laser treatments and tightening treatments. Waxing and threading is allowed but not facial laser hair removal. | | С |
| | If male, who is a regular shaver and willing to shave on the day of the study visits (prior to clinic visits). | | |
| t | If a woman of child bearing potential, is willing to take a urine pregnancy test prior to study enrollment, at week 24, and when deemed appropriate by the Investigator and/or Sponsor. | | |
| c | Is of child bearing potential who uses an acceptable method of contraception throughout the study. Acceptable methods of birth control include Oral and other system contraceptives. Individuals must be on a stable use for 3 months prior to study enrollment. Individuals on oral contraceptives must not alter their use, including dose or regimen for the duration of the study Double barrier Bilateral tubal ligation Partner vasectomy Abstinence | | С |
| | Is willing to follow study requirements and report any changes in health status or medications, adverse event symptoms, or reactions immediately. | | |
| 14. N | Must be stable on any medication they are taking for at least 30 days | | |

| ĺ | Source Documents | | | | | | |
|---|---|---|---|---|---|---|---|
| | | | | | Subject I | nitials | |
| | | Galderma | Study # C16-CD020 | INVESTIGTOR NAME | | | |
| | | | | To be added per site | <u> </u> | | |
| | | | | | Subject N | lumber | |
| | | | | | | Yes* | No |
| | 1. | Has been diagnose | ed with allergies to topical | l acne products. | | | |
| | 2. | | <u> </u> | hat the Investigator deems | | | |
| | | inappropriate for participation. | | | | | |
| | 3. | Is nursing, pregna | nt, or planning to become | pregnant during the study. | | | |
| | 4. | Have pre-existing | or dormant dermatologic | conditions on the face (e.g. | , | | |
| | | psoriasis, rosacea, eczema, seborrheic dermatitis, severe excoriations etc.) | | | | | |
| | | which in the opinion of the Investigator could interfere with the outcome of the | | | | | |
| | | study. | | | | | |
| | 5. | | | ne deficiency disorders (incl | • | | |
| | | • | | munosuppressive medication | ons (e.g., | | |
| | | · | | e, Enbrel, Imuran, Humira, | | | |
| | <i>C</i> | | | dnisone, Remicade, Stelara.) | i <u>.</u> | | |
| | 6. | | ed disease such as asthma | l, diabetes, hypertension,<br>luals having multiple health | | | |
| | | • | • • • • | ion even if the conditions ar | | | |
| | | • | , medication, etc. at the In | | C | | |
| | 7. | | | sage study or has participate | ed in a | | |
| | | | • | rch facility or doctor's office | | | |
| | | | nclusion into the study. | , | | | |
| | 8. | Has a history of sk | in cancer within the past! | 5 years. | | | |
| | 9. | Has any planned s | urgeries and/or invasive r | nedical procedures during t | he | | |
| | | course of the stud | | | | | |
| | 10. | | | s (HRT) or hormones for bir | | | |
| | | | | try or plans on starting, sto | pping, or | | |
| | | | | h control during the study. | | | |
| | 11. | | | ll skin or is not willing to avo | • | _ | |
| | | • | | ning beds or sunless tannin | g | | |
| | 12 | | uration of the study. | nodulas ar cysts (mara than | 2) | + | |
| | | | | nodules or cysts (more than<br>testosterone blocker (e.g. sa | | | |
| | 13. | | • | berry, spironolactone, drosp | | | |
| | | progestins). | moon, chaste tree, chaster | cerry, spiroriolactoric, arosp | , co., | | |
| | 14. | | estosterone booster or pre | escription testosterone (e.g | . DHEA. | 1 | |
| | | • | one cypionate, testostero | | <b>-</b> / | | |
| | | | | nylpropriate, Omnadren etc | .). | | |
| | | (CONTINUED ON | | • | | | |

| | Source D | ocuments | Subject Ir | nitials | |
|---|---|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME | Judgetti | Treats | |
| | | To be added per site | Subject N | umber | |
| Visit 1 –Baseline | | | | | |
| VISIC 1 DUSCHIIC | | | | | |
| EXCLUSION CRITERIA (CON | NTINUED) | | | 1 | |
| | | | | Yes* | No |
| prescription med<br>Clindamycin, Bac<br>tretinoin.(Retin A | dications for acne suctrim, Tetracycline, Eryth | nromycin, Vibramycin an<br>Tazarotene), Azelaic acid | nocycline,<br>d topical | | |
| | retinoin (Accutane) within | | | | |
| 17. Is routinely using (3x a week or more) topical OTC acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 30 days of the study entry. | | | | | |
| 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. | | | | | |
| 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. | | | | | |
| | · | <b>OT</b> enroll the subject. | 1 | ı | |
| Visit 1 – Baseline INCLUSION/EXCLUSION | | | | | |
| Is the subject eligible per I | | a? | | | |
| ☐ Yes ☐ No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: | | | | | |
| Inclusion # Exclusion # | | | | | |
| Investigators review | | | | | |
| • | | wed by me, deemed accuration and is eligible to be enr | | • | and |

DD

MMM

YYYY

Investigator's Signature

| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |

# Visit 1 –Baseline (Day 1)

| INCLUSI | ION CRITERIA | | |
|---|---|---|---|
| | | Yes | No* |
| 1. | Is a man or woman between the ages of 21 and 45 years of age at the time of enrollment. | | |
| 2. | Has mild to moderate acne (score of 2-3 on FDA Investigator's Global Assessment Scale) on the face. | | |
| 3. | Have at least 5 inflammatory lesions. | | |
| 4. | Have 10 – 100 non-inflammatory lesions. | | |
| 5. | Is willing to use the test products as instructed for 24 weeks. | | |
| 6. | Has a Fitzpatrick skin type I-VI | | |
| 7. | Is willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol. | | |
| 8. | Is willing to provide written informed consent including photo release, Health Insurance Portability and Accountability Act (HIPAA), and is able to read, speak, write, understand English and is willing to share personal information and data, as verified by signing a written authorization at the screening | | |
| 9. | Is willing to withhold all facial treatments during the course of the study including botulinum toxin, injectable fillers, microdermabrasion, IPL, peels, facials, laser treatments and tightening treatments. Waxing and threading is allowed but not facial laser hair removal. | | |
| 10. | If male, who is a regular shaver and willing to shave on the day of the study visits (prior to clinic visits). | | |
| 11. | If a woman of child bearing potential, is willing to take a urine pregnancy test prior to study enrollment, at week 24, and when deemed appropriate by the Investigator and/or Sponsor. | | |
| 12. | Is of child bearing potential who uses an acceptable method of contraception throughout the study. Acceptable methods of birth control include Oral and other system contraceptives. Individuals must be on a stable use for 3 months prior to study enrollment. Individuals on oral contraceptives must not alter their use, including dose or regimen for the duration of the study Double barrier Bilateral tubal ligation Partner vasectomy Abstinence | | |
| | Is willing to follow study requirements and report any changes in health status or medications, adverse event symptoms, or reactions immediately. | | |
| 14. | Must be stable on any medication they are taking for at least 30 days | | |
| *If any | v criterion is answered no*. <b>DO NOT</b> enroll the subject. | | |

Visit 1 –Baseline (Day 1)

| ſ | Source Documents | | | | | | |
|---|---|---|---|---|---|---|---|
| Ī | | | | | Subject Ir | nitials | |
| | | Galderma | Study # C16-CD020 | INVESTIGTOR NAME | | | |
| | | | | To be added per site | | | |
| | | | | | Subject N | lumber | |
| | | | | | | Yes* | No |
| | 1. | Has been diagnose | ed with allergies to topica | Lacne products. | | | |
| | 2. | | • | hat the Investigator deems | | | |
| | | inappropriate for | | 0 | | | |
| | 3. | Is nursing, pregna | nt, or planning to become | pregnant during the study. | | | |
| | 4. | Have pre-existing | or dormant dermatologic | conditions on the face (e.g. | , | | |
| | | psoriasis, rosacea, eczema, seborrheic dermatitis, severe excoriations etc.) | | etc.) | | | |
| | | which in the opini | on of the Investigator cou | ıld interfere with the outcor | ne of the | | |
| | | study. | | | | | |
| | 5. | Has a history of im | nmunosuppression/immu | ne deficiency disorders (incl | uding | | |
| | | • | | munosuppressive medication | ons (e.g., | | |
| | | • | | le, Enbrel, Imuran, Humira, | | " | |
| | | | | dnisone, Remicade, Stelara. | ). | | |
| | 6. | | | a, diabetes, hypertension, | | | |
| | | • • | | duals having multiple health | | | |
| | | | | ion even if the conditions a | re | | _ |
| | | • | , medication, etc. at the Ir | | | | |
| | 7. | | | sage study or has participate | | _ | |
| | | | | rch facility or doctor's office | e within | | |
| | | • | nclusion into the study. | _ | | | |
| | 8. | • | in cancer within the past | | | | |
| | 9. | | _ | medical procedures during t | ne | | |
| | 40 | course of the stud | • | . (UDT) | ı.l. | | |
| | 10. | | · | s (HRT) or hormones for bir | | | |
| | | | | ntry or plans on starting, sto | pping, or | | |
| | 11 | | | th control during the study. I skin or is not willing to avo | منط طمناب | | |
| | 11. | | | nning beds or sunless tannin | • | | |
| | | • | uration of the study. | ining beas of suffices tailinin | Б | | |
| | 12 | | | nodules or cysts (more than | <br>1 2) | | |
| | | | | testosterone blocker (e.g. sa | | | |
| | 13. | , , | · · | berry, spironolactone, dros | | | |
| | | progestins). | moon, chaste tree, chaste | Serry, spiroriolactoric, arosp | c | | |
| | 14. | | estosterone booster or pr | escription testosterone (e.g | . DHFA. | | |
| | ± ··• | • | one cypionate, testostero | | , | | |
| | | | • • | nylpropriate, Omnadren etc | .). | _ | _ |
| | | (CONTINUED ON | • | 7 p p | <i>r</i> - | † | |
| | | , | - , | | | 1 | |

| | Source D | ocuments | Subject Ir | nitials | |
|---|---|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME | Judgetti | Treats | |
| | | To be added per site | Subject N | umber | |
| Visit 1 –Baseline | | | | | |
| VISIC 1 DUSCHIIC | | | | | |
| EXCLUSION CRITERIA (CON | NTINUED) | | | 1 | |
| | | | | Yes* | No |
| prescription med<br>Clindamycin, Bac<br>tretinoin.(Retin A | dications for acne suctrim, Tetracycline, Eryth | nromycin, Vibramycin an<br>Tazarotene), Azelaic acid | nocycline,<br>d topical | | |
| | retinoin (Accutane) within | | | | |
| 17. Is routinely using (3x a week or more) topical OTC acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 30 days of the study entry. | | | | | |
| 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. | | | | | |
| 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. | | | | | |
| | · | <b>OT</b> enroll the subject. | 1 | ı | |
| Visit 1 – Baseline INCLUSION/EXCLUSION | | | | | |
| Is the subject eligible per I | | a? | | | |
| ☐ Yes ☐ No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: | | | | | |
| Inclusion # Exclusion # | | | | | |
| Investigators review | | | | | |
| • | | wed by me, deemed accuration and is eligible to be enr | | • | and |

DD

MMM

YYYY

Investigator's Signature

| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME Barry T. Reece | Subject Initials |
| | | (RCTS, Inc.) | Screening Number |

# Visit 1 –Screening/Baseline (Day 1)

| INCLUS | SION CRITERIA | | |
|---|---|---|---|
| | | Yes | No* |
| 1. | Is a man or woman between the ages of 21 and 45 years of age at the | | |
| | time of enrollment. | | |
| 2. | Has mild to moderate acne (score of 2-3 on FDA Investigator's Global Assessment Scale) on the face. | | |
| 3. | Have at least 5 inflammatory lesions. | | |
| 4. | Have 10 – 100 non-inflammatory lesions. | | |
| 5. | Is willing to use the test products as instructed for 24 weeks. | | |
| 6. | Has a Fitzpatrick skin type I-VI | | |
| | · | | Ш |
| 7. | Is willing and able to comply with all of the time commitments and | | |
| 0 | procedural requirements of the clinical trial protocol. | | |
| 8. | Is willing to provide written informed consent including photo release, | | |
| | Health Insurance Portability and Accountability Act (HIPAA), and is able to | | |
| | read, speak, write, understand English and is willing to share personal | | |
| | information and data, as verified by signing a written authorization at the | | |
| 0 | screening | | |
| 9. | Is willing to withhold all facial treatments during the course of the study | | |
| | including botulinum toxin, injectable fillers, microdermabrasion, IPL, | | |
| | peels, facials, laser treatments and tightening treatments. Waxing and | | |
| 10 | threading is allowed but not facial laser hair removal. | | |
| 10 | . If male, who is a regular shaver and willing to shave on the day of the study visits (prior to clinic visits). | | |
| 11 | . If a woman of child bearing potential, is willing to take a urine pregnancy | | |
| 11. | test prior to study enrollment, at week 24, and when deemed appropriate | | |
| | by the Investigator and/or Sponsor. | | |
| 12 | . Is of child bearing potential who uses an acceptable method of | - | |
| 12. | contraception throughout the study. Acceptable methods of birth control | | |
| | include | | |
| | Oral and other system contraceptives. Individuals must be on a | | |
| | stable use for 3 months prior to study enrollment. Individuals on | | |
| | oral contraceptives must not alter their use, including dose or | | |
| | regimen for the duration of the study | | |
| | Double barrier | | |
| | Bilateral tubal ligation | | |
| | Partner vasectomy | | |
| | Abstinence | | |
| 12 | . Is willing to follow study requirements and report any changes in health | | |
| 13 | status or medications, adverse event symptoms, or reactions immediately. | | |
| 1.4 | . Must be stable on any medication they are taking for at least 30 days | | П |
| | · | | |
| ı "ıt an | y criterion is answered no*, <b>DO NOT</b> enroll the subject. | | |

| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME Barry T. Reece | Subject Initials |
| | | (RCTS, Inc.) | Screening Number |

# Visit 1 –Screening/Baseline (Day 1)

| EXCLUSION CRITERIA | | |
|---|---|---|
| | Yes* | No |
| <ol> <li>Has been diagnosed with allergies to topical acne products.</li> </ol> | | |
| 2. Has a condition and/or disease of the skin that the Investigator deems | | |
| inappropriate for participation. | | |
| 3. Is nursing, pregnant, or planning to become pregnant during the study. | | |
| 4. Have pre-existing or dormant dermatologic conditions on the face (e.g., | | |
| psoriasis, rosacea, eczema, seborrheic dermatitis, severe excoriations etc.) | | l 🗖 |
| which in the opinion of the Investigator could interfere with the outcome of th | e $\Box$ | |
| study. | | |
| 5. Has a history of immunosuppression/immune deficiency disorders (including | | |
| (HIV infection or AIDS) or currently using immunosuppressive medications (e.g. | , l 🗆 | |
| azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, | | |
| mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.). | | |
| 6. Has an uncontrolled disease such as asthma, diabetes, hypertension, | | |
| hyperthyroidism, or hypothyroidism. Individuals having multiple health | | |
| conditions may be excluded from participation even if the conditions are | | |
| controlled by diet, medication, etc. at the Investigator's discretion. | _ | |
| 7. Is currently participating in another facial usage study or has participated in a | | П |
| clinical trial at this or at another research facility or doctor's office within 4 weeks prior to inclusion into the study. | | |
| | <del> </del> | П |
| <ul><li>8. Has a history of skin cancer within the past 5 years.</li><li>9. Has any planned surgeries and/or invasive medical procedures during the</li></ul> | <del> </del> | Ш |
| course of the study. | | |
| 10. Has started hormone replacement therapies (HRT) or hormones for birth | | |
| control less than 3 months prior to study entry or plans on starting, stopping, o | r 🗆 | П |
| changing doses of HRT or hormones for birth control during the study. | ' " | |
| 11. Has facial sunburn or excessive tanned facial skin or is not willing to avoid daily | | |
| sun exposure on the face and the use of tanning beds or sunless tanning | | |
| products for the duration of the study. | | |
| 12. Has severe acne, acne conglobata, multiple nodules or cysts (more than 2). | | |
| 13. Is currently taking a natural or prescription testosterone blocker (e.g. saw | | |
| palmetto, blask cohosh, chaste tree, chasteberry, spironolactone, drospirenone | e, 🗆 | |
| progestins). | | |
| 14. Is currently on a testosterone booster or prescription testosterone (e.g. DHEA, | | |
| tribulus, testosterone cypionate, testosterone enanthate, Sustanon, | | |
| testosterone propionate, testosterone phenylpropriate, Omnadren etc.). | | |
| (CONTINUED ON NEXT PAGE) | | |
| Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | | Source D | ocuments | | | | |
|---|---|---|---|---|---|---|--|
| Study # C16-CD020 | | Source D | ocuments | Subject In | nitials | | |
| Screening Number Screening N | Galderma | Study # C16-CD020 | INVESTIGTOR NAME | Jubject II | iitiais | | |
| Screening Number | | | | | | | |
| SEXCLUSION CRITERIA (CONTINUED) Yes* No | | | · · | Screening | Number | | |
| SEXCLUSION CRITERIA (CONTINUED) Yes* No | | | | | | | |
| SEXCLUSION CRITERIA (CONTINUED) Yes* No | | | | | | | |
| Yes* No 15. Is currently taking or has taken within the last 30 days oral or topical prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin.(Retin A Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo. 16. Has used oral isotretinoin (Accutane) within the past 6-months. 17. Is routinely using (3x a week or more) topical OTC acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 30 days of the study entry. 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | Visit 1 –Screening/Baselin | <u>1e</u> | | | | | |
| 15. Is currently taking or has taken within the last 30 days oral or topical prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin. (Retin A Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo. 16. Has used oral isotretinoin (Accutane) within the past 6-months. 17. Is routinely using (3x a week or more) topical OTC acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 30 days of the study entry. 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Wisit 1 - Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete and of Study page: Inclusion # | EXCLUSION CRITERIA (CON | NTINUED) | | | | | |
| prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin.(Retin A Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo. 16. Has used oral isotretinoin (Accutane) within the past 6-months. 17. Is routinely using (3x a week or more) topical OTC acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 30 days of the study entry. 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | | | | | Yes* | No | |
| prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin.(Retin A Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo. 16. Has used oral isotretinoin (Accutane) within the past 6-months. 17. Is routinely using (3x a week or more) topical OTC acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 30 days of the study entry. 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | 15 Is currently takin | g or has taken within | the last 20 days oral of | or tonical | | | |
| Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin.(Retin A Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo. 16. Has used oral isotretinoin (Accutane) within the past 6-months. 17. Is routinely using (3x a week or more) topical OTC acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 30 days of the study entry. 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | | ~ | · | • | | | |
| tretinoin. (Retin A Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo. 16. Has used oral isotretinoin (Accutane) within the past 6-months. 17. Is routinely using (3x a week or more) topical OTC acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 30 days of the study entry. 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | · | | • • | • | | | |
| 16. Has used oral isotretinoin (Accutane) within the past 6-months. 17. Is routinely using (3x a week or more) topical OTC acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 30 days of the study entry. 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | • | | | • | | | |
| 17. Is routinely using (3x a week or more) topical OTC acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 30 days of the study entry. 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | peroxide, Dapsone | e, Sodium sulfacetamide, I | Differin, Epiduo. | | | | |
| peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 30 days of the study entry. 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | 16. Has used oral isot | retinoin (Accutane) within | the past 6-months. | | | | |
| products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 30 days of the study entry. 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | , , | • | • | • | | | |
| 30 days of the study entry. 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # Inclusion # Exclusion # | • • • • | | | • | | | |
| 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | · | · | isks, scrubs, gels and cream | is) within | | | |
| acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | | • | n considered to affect the | course of | | | |
| days prior to entry into the study. 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | | · · | | | П | | |
| 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. *If any criterion is answered Yes*, DO NOT enroll the subject. Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | | | | | | | |
| *If any criterion is answered Yes*, DO NOT enroll the subject. *Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | | | | | | | |
| Visit 1 – Screening/Baseline INCLUSION/EXCLUSION Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # | could interfere wi | th evaluations by Investiga | ator or designee. | | | Ш | |
| Investigators review Inclusion/Exclusion Exclusion criteria? Investigators review Infirm that all required information has been reviewed by me, deemed accurate and complete and | *If any criterion is an | nswered <b>Yes*, <u>DO N</u>O</b> | <u>OT</u> enroll the subject. | | | | |
| Investigators review Inclusion/Exclusion Exclusion criteria? Investigators review Infirm that all required information has been reviewed by me, deemed accurate and complete and | | | | | | | |
| Investigators review Inclusion/Exclusion Inclusion/Exclusion criteria? Inclusion # Exclusion # Investigators review Infirm that all required information has been reviewed by me, deemed accurate and complete and | Visit 1 — Scrooning/Basoli | no | | | | | |
| Is the subject eligible per Inclusion/Exclusion criteria? Yes No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # Investigators review Infirm that all required information has been reviewed by me, deemed accurate and complete and | VISIC 1 — Screening/ basein | <u>iie</u> | | | | | |
| ☐ Yes ☐ No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # Investigators review I affirm that all required information has been reviewed by me, deemed accurate and complete and | INCLUSION/EXCLUSION | | | | | | |
| □ No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # Investigators review I affirm that all required information has been reviewed by me, deemed accurate and complete and | Is the subject eligible per I | nclusion/Exclusion criteria | a? | | | | |
| □ No If no, please indicate which Inclusion/Exclusion criteria the subject did not meet and complete End of Study page: Inclusion # Exclusion # Investigators review I affirm that all required information has been reviewed by me, deemed accurate and complete and | _ | | | | | | |
| Inclusion # Exclusion # Investigators review Infirm that all required information has been reviewed by me, deemed accurate and complete and | □ Yes | | | | | | |
| Inclusion # Exclusion # Investigators review Infirm that all required information has been reviewed by me, deemed accurate and complete and | □ No. If no. please indica | to which Inclusion/Evolusi | on critoria the subject did : | not meet a | nd com | nloto | |
| Inclusion # Exclusion # Investigators review I affirm that all required information has been reviewed by me, deemed accurate and complete and | - | te willen inclusion, exclusi | on criteria the subject did i | not meet a | na com | piete | |
| Investigators review I affirm that all required information has been reviewed by me, deemed accurate and complete and | zna or otaay pager | | | | | | |
| affirm that all required information has been reviewed by me, deemed accurate and complete and | Inclusion # | Exclusion # | | | | | |
| affirm that all required information has been reviewed by me, deemed accurate and complete and | | | | | | | |
| affirm that all required information has been reviewed by me, deemed accurate and complete and | | | | | | | |
| affirm that all required information has been reviewed by me, deemed accurate and complete and | | | | | | | |
| affirm that all required information has been reviewed by me, deemed accurate and complete and | Investigators review | | | | | | |
| that the subject meets the inclusion/exclusion criteria, and is eligible to be enrolled in the study. | | nformation has been revie | wed by me, deemed accura | ate and cor | nplete a | and | |
| | that the subject meets the inclusion/exclusion criteria, and is eligible to be enrolled in the study. | | | | | | |

DD

MMM

YYYY

Investigator's Signature


| Source Documents | | | | | | |
|---|---|---|---|---|---|---|
| | | | | Su | bject Initials | ; |
| Galderma | Study # C16-CD020 | INV | ESTIGTOR NAM | E | | |
| | | To I | be added per sit | e L | | |
| | | | | Su | bject Numb | er |
| | | SITE | E NUMBER | | | |
| | | Tol | be added per sit | e L | | |
| Visit 1 –Screening | | ١ | /isit Date: | | | |
| | | | DI | O-MMM-Y | /YYY | |
| Check In Procedures | | | | | | |
| Has the subject cleansed t | | | - | - | | |
| ☐ Yes ☐ No | (If no, subject needs to re | emove | e residual makeu | ip and acc | dimate 20 m | ninutes) |
| Acclimation | | | | | | |
| *Reminder: Subject must | acclimate for at least 15 n | minuta | os in tomporatu | o of 69.7 | E°E and rola | tivo |
| humidity range 35-65% be | | | • | | | live |
| | _ | | | | | |
| Acclimation start time : | :AM/PM | Accl | imation end tim | e : | _: | AM/PM |
| Technician initials: | Date(D | D-MM | M-YYYY): | | | |
| | , | | - | | | |
| Informed Consent/HIPAA | /Photo Release | | | | | |
| Date & Time Consent | | | | | | |
| Obtained | DD MMM YYYY | | Time::: | AM / PM | | |
| Date of HIPAA | I I I I I I I I I I I I I I I I I I I | | | | | |
| Authorization | | | | | | |
| | DD MMM YYYY | | | | YES | NO |
| Was consent obtained price | or to any study related nr | ocedu | ıre? | | | |
| Was the consent reviewed | | occuu | | | | |
| Was the subject allowed to | | them | answered? | | | |
| Did the subject receive a f | | | | | | |
| Was the photo release sign | , , | - | | | | |
| , | | | | | | 1 |
| Demographics | | | | | | |
| Sex: ☐ Male ☐ Female | Date of Birth: | | / | | tween 21 and 4 | 5 years of age. |
| | DD | MN | | Age ( | Years): | |
| Race: | | | Ethnicity: | | | |
| □ American Indian/Alaskan Native □ Hispanic or Latino □ | | | | | | |
| □ Asian □ Not Hispanic or Latino | | | | | | |
| □Black/African American | | | | | | |
| □Native Hawaiian/ other Pacific Islander | | | | | | |
| □White | | | | | | |
| □Other: (specify) | | | | | | |
| Fitzpatrick Skin Type (Mark one): | | | | | | |


Subject Initials

| | | | | | | | | | Suk | oject Num | ber | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | _ | NUMBE | | | | | | |
| | All > 0 | | | | To b | e added | per s | ite | <u> </u> | | | |
| | All Visits | | | | | | | | | | | |
| Medical His | tory Pag | je 🗆 1 🗆 2 | □3 □4 | □5 [ | | | Last | Page | | | | |
| ☐ Check thi | is box only if there is <b>NO</b> | recent ar | nd relevar | <u>nt</u> med | dical histo | ory and le | eave 1 | the forr | n bla | ank | | |
| | ent/relevant past and/one condition or surgery | | | | | • | _ | | | | • | _ |
| | on and one line for the s | - | | _ | | | _ | - | | | | |
| medication | | argery. En | ter an me | arcatic | JIIJ takei | · wiciiii c | , ,,,, | iciis pii | 01 10 | , serceilli | g on the cont | Jonnana |
| | quired for Date of Diag | nosis/Surg | ery and R | Resolv | ed. Ente | r UN for | any u | ınknow | n DI | or MMN | Л. | |
| | <u>, , </u> | | | | | | - | | | | | Physician |
| Condition/D | Diagnosis/Surgery | | of Diagnos<br>DD-MMM | | • . | | | te Resc<br>-MMM | | | Ongoing | 's initials |
| | | (1 | ואוואוואו-טכ | -1111, | <u> </u> | | (00 | -101101101 | -111 | 1) | | and date |
| | | | | | | | | 40.40.4 | - | | | |
| | | DD - | MMM | - | YYYY | DD | - N | ИММ | - | YYYY | | |
| | | _ | | _ | | | _ | | _ | | | |
| | | DD - | MMM | | YYYY | DD | - N | 1MM | _ | YYYY | | |
| | | | | | | | | | - | | | |
| | | DD - | MMM | - | YYYY | DD | - N | MM | - | YYYY | | |
| | | <br>DD - | MMM | · | YYYY | DD | | 1MM | _ | YYYY | | |
| | | | 171171171 | | | | .,, | | | | | |
| | | | | - | | | | | - | | | |
| | | DD - | MMM | - | YYYY | DD | - N | <b>ИММ</b> | - | YYYY | | |
| | | | | · | | | | | - | | | |
| | | DD - | MMM | - | YYYY | DD | - N | 1MM | - | YYYY | | |
| | | <br>DD - | MMM | · | YYYY | DD | - N | <br>1MM | _ | YYYY | | |
| | | | ********** | | | 55 | ., | | | | <del> _</del> | |
| | | | | <b>.</b> | | | | | - | | | |
| | | DD - | MMM | | YYYY | DD | - N | 1MM | _ | YYYY | | |
| | Enter all medications ta | ken withir | n 6 month | s prio | r to Scree | ening on | the c | oncomi | itant | medicati | on page. | |

**Source Documents** 

INVESTIGTOR NAME
To be added per site

Study # C16-CD020

Galderma

| Source Documents | | | |
|---|---|---|---|
| | | | Subject Initials |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME | |
| | | To be added per site | |
| | | | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |

## **All Visits**

| <b>MEDICATIONS</b> | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| RECORD ANY MEDICA | ATIONS INCLUDING | PRESCRIPTION | ON AND | OTC DRUGS | TAKEN REG | GURARLY, IN | TERMITTITENTLY OR ONE TIM | E ONLY TAKEN WITH | N 6 MONTHS |
| PRIOR TO SIGING THE | ICF UNTIL THE EN | D OF THE STU | JDY. A j | ear is requi | red for Stai | t Date. Ente | er UN for any unknown DD o | MMM. | |
| | | | | | | | Page | □ 1 □ 2 □3 □4 □! | 5 🗆 |
| Review for prohibite | d medications use | e for the last ( | 6 month | ıs | | | | ☐ Last Page | <u> </u> |
| □ NONE USED/TAKEN (leave | e rest of the page blank ) | | | | | | | | |
| Drug name (Generic or | | Used to | | | | | Start Date | | Physician's |
| Brand name) | Indication | treat an AE? | Dose | Frequency | Route* | | Stop Date<br>(DD-MMM-YYYY) | Ongoing | initials and date |
| | | | | | | Start | | | |
| | | ☐ Yes | | | | | _ | | |
| | | □ Yes | | | | | | | |
| | | l live | | | | Stop | | | |
| | | | | | | Start | | | |
| | | ☐ Yes | | | | | _ | | |
| | | □ Yes | | | | | | | |
| | | | | | | Stop | | | |
| | | | | | | | <del></del> | | |
| | | | | | | Start | | | |
| | | ☐ Yes | | | | | _ | | |
| | | □ No | | | | Ston | | | |
| | | | | | | Stop | | | |

<sup>\*1=</sup>oral, 2=topical, 3=subcutaneous, 4=transdermal, 5=Intraocular,6=Intramuscular, 7=Inhalation, 8= Intralesion, 9=Intraperitoneal, 10=Intravenous, 11=Nasal, 12=Vaginal, 13=Rectal,14= Ophthalmic, 15=Unknown, 16=Other

| | | | | | | Page <b>4</b> of | 3 |
|---|---|---|---|---|---|---|---|
| | Source [ | Documents | | | | | |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site SITE NUMBER To be added per site | | | Subject<br>Subject | Number | _<br>]<br>] |
| Visit 1 – Screening | | 10000000 | - 1 | | | | |
| Qualification Criteria Subject must have mild to Assessment Scale, at least | | | | _ | | | |
| Does the subject have mile | • | | | l Yes Scor | • | □No | |
| Does the subject have at le | east 5 inflammatory lesio | ns? | | l Yes (>5) | | □No | |
| Does the subject have 10 - | - 100 non-inflammatory I | lesions? | Е | ☐ Yes (10-100) * ☐ No | | | |
| Technician initials: | Date(I | DD-MMM-YYYY): | | | | _ | |
| *Tolerability Instructions:<br>symptoms of erythema, di<br>stinging/burning on the gla<br>more accurately describe to<br>Parameter | ryness, and scaling, and book obal face (treatment area the skin condition): 0 = no | y subject repo<br>a). (Half-point<br>one, 1 = mild,<br><b>Glob</b> | orti<br>sco<br>2 =<br><b>cal</b> | ng of the de<br>ores may be<br>moderate,<br>Face | gree of<br>used as<br>3 = seve | necessary to | |
| | Ent | ter 2 digits for al | I SC | ores (le 0.5, 1.0 | , 2.0) | | |
| Erythema | | | • | | | | |
| Dryness | | | • | | | | |
| Scaling | | | • | | | | |
| Burning/Stinging | | | • | | | | |
| Evaluator's initials: | Date(DD-MM | M-Y | YYY): | | | | |

| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |
| | | SITE NUMBER To be added per site | |

# Visit 1 –Screening

| INCLU | JSION CRITERIA | Yes | No* |
|---|---|---|---|
| 1. Is | s a man or woman between the ages of 21 and 45 years of age at the | Ι | |
| ti | me of enrollment. | | Ш |
| 2. H | las mild to moderate acne (score of 2-3 on FDA Investigator's Global | | П |
| А | ssessment Scale) on the face. | | |
| 3. H | lave at least 5 inflammatory lesions. | | |
| 4. H | lave 10 – 100 non-inflammatory lesions. | | |
| 5. Is | s willing to use the test products as instructed for 24 weeks. | | |
| 6. H | las a Fitzpatrick skin type I-VI | | |
| 7. Is | s willing and able to comply with all of the time commitments and | | |
| р | rocedural requirements of the clinical trial protocol. | ] | ] |
| 8. Is | s willing to provide written informed consent including photo release, | | |
| Н | lealth Insurance Portability and Accountability Act (HIPAA), and is able | | |
| to | o read, speak, write, understand English and is willing to share | | |
| р | ersonal information and data, as verified by signing a written | | |
| а | uthorization at the screening | | |
| | s willing to withhold all facial treatments during the course of the | | |
| st | tudy including botulinum toxin, injectable fillers, microdermabrasion, | П | |
| | PL, peels, facials, laser treatments and tightening treatments. Waxing | | |
| a | nd threading is allowed but not facial laser hair removal. | | |
| | male, who is a regular shaver and willing to shave on the day of the | | П |
| | tudy visits (prior to clinic visits). | ] | ] |
| | a woman of child bearing potential, is willing to take a urine | | |
| - | regnancy test prior to study enrollment, at week 24, and when | | |
| | eemed appropriate by the Investigator and/or Sponsor. | | |
| | of child bearing potential who uses an acceptable method of | | |
| | ontraception throughout the study. Acceptable methods of birth | | |
| | ontrol include | | |
| ' | Oral and other system contraceptives. Individuals must be on a | | |
| | stable use for 3 months prior to study enrollment. Individuals on | | |
| | oral contraceptives must not alter their use, including dose or | | |
| | regimen for the duration of the study | | |
| | Double barrier | | |
| | Bilateral tubal ligation | | |
| | Partner vasectomy | | |
| | Abstinence | | |
| | s willing to follow study requirements and report any changes in | | |
| | ealth status or medications, adverse event symptoms, or reactions | | |
| | nmediately. | | |
| | Must be stable on any medication they are taking for at least 30 days | | |
| *If a | *If any criterion is answered no*, <b>DO NOT</b> enroll the subject. | | |

| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |
| | | SITE NUMBER To be added per site | |

# Visit 1 –Screening

| EXCLU | SION CRITERIA | Yes* | No |
|---|---|---|---|
| 1. Ha | s been diagnosed with allergies to topical acne products. | | |
| | s a condition and/or disease of the skin that the Investigator deems | | |
| | appropriate for participation. | | |
| | nursing, pregnant, or planning to become pregnant during the study. | Ш | Ш |
| pso<br>wh | ove pre-existing or dormant dermatologic conditions on the face (e.g., oriasis, rosacea, eczema, seborrheic dermatitis, severe excoriations etc.) nich in the opinion of the Investigator could interfere with the outcome the study. | | |
| (in<br>me<br>Im | is a history of immunosuppression/immune deficiency disorders cluding (HIV infection or AIDS) or currently using immunosuppressive edications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, uran, Humira, mycophenolate mofetil, methotrexate, prednisone, emicade, Stelara.). | | |
| hy <sub>l</sub><br>coi<br>coi | is an uncontrolled disease such as asthma, diabetes, hypertension, perthyroidism, or hypothyroidism. Individuals having multiple health nditions may be excluded from participation even if the conditions are ntrolled by diet, medication, etc. at the Investigator's discretion. | | |
| in a | currently participating in another facial usage study or has participated a clinical trial at Stephens or at another research facility or doctor's fice within 4 weeks prior to inclusion into the study. | | |
| 8. Ha | s a history of skin cancer within the past 5 years. | | |
| | is any planned surgeries and/or invasive medical procedures during the urse of the study. | | |
| 10. Ha | os started hormone replacement therapies (HRT) or hormones for birth ntrol less than 3 months prior to study entry or plans on starting, opping, or changing doses of HRT or hormones for birth control during e study. | | |
| dai | is facial sunburn or excessive tanned facial skin or is not willing to avoid ily sun exposure on the face and the use of tanning beds or sunless nning products for the duration of the study. | | |
| 12. Ha | s severe acne, acne conglobata, multiple nodules or cysts (more than 2). | | |
| ра | currently taking a natural or prescription testosterone blocker (e.g. saw Imetto, blask cohosh, chaste tree, chasteberry, spironolactone, ospirenone, progestins). | | |
| DH | currently on a testosterone booster or prescription testosterone (e.g. HEA, tribulus, testosterone cypionate, testosterone enanthate, Sustanon, stosterone propionate, testosterone phenylpropriate, Omnadren etc.). | | |
| | (CONTINUED ON NEXT PAGE) | | |


| | Source Documents | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |


| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |

# Visit 1 –Screening

| EXCLUSION CRITERIA CONTINUED | Yes* | No |
|---|---|---|
| 15. Is currently taking or has taken within the last 30 days oral or topical prescription medications for acne such as Doxycycline, Minocycline, Clindamycin, Bactrim, Tetracycline, Erythromycin, Vibramycin and topical tretinoin.(Retin A Renova, Adapalene, Tazarotene), Azelaic acid, benzoyl peroxide, Dapsone, Sodium sulfacetamide, Differin, Epiduo. | | |
| 16. Has used oral isotretinoin (Accutane) within the past 6-months. | | |
| 17. Is routinely using (3x a week or more) topical OTC acne product (e.g. benzoyl peroxide, salicylic acid, alpha hydroxyl, beta hydroxyl and/or polyhydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) within 30 days of the study entry. | | |
| 18. Is using or has used any systemic medication considered to affect the course of acne, specifically, but not exclusively antibiotics or steroids within the last 30 days prior to entry into the study. | | |
| 19. Has excessive facial hair, including beard, mustache or goatee, or scars, which could interfere with evaluations by Investigator or designee. | | |
| *If any criterion is answered <b>Yes*</b> , <b>DO NOT</b> enroll the subject. | | |

| Urine Pregnancy Test | | | |
|---|---|---|---|
| If the candidate subject qualifies and is female of child-bearing potential, conduct a urine pregnancy test. Candidate female subjects with negative results, females of non-child-bearing potential, or candidate males that qualify will proceed to the next step. | | | |
| Test Results | Reason Not Applicable | Kit Lot # | Kit Expiration date |
| □ Neg □ Pos □N/A | | | |
| Technician initials: | Time::AN | //PM Date(DD-MMM-Y | YYY): |

YYYY

| | | | Page <b>9</b> of <b>3</b> |
|---|---|---|---|
| | Source | Documents | |
| | | | Subject Initials |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME | |
| | | To be added per site | |
| | | | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |
| Visit 1 –Screening | | | |
| 111011101011/57011101011 | _ | | |
| INCLUSION/EXCLUSION | | . • | |
| Is the subject eligible per | Inclusion/Exclusion crite | ria? | |
| <b></b> | | | |
| ☐ Yes | | | |
| □ No. of an alamatada. | ata di Nahata di Ata de Ate | ata a sa atra da atra a lata a lata a | |
| • | ate which inclusion/Exclu | sion criteria the subject did | not meet and complete |
| End of Study page: | | | |
| In aluaio a # | Evaluation # | | |
| inclusion # | Exclusion #_ | | |
| Investigators review | | | |
| | nformation has been revi | iewed by me, deemed accu | rate and complete and |
| | | eria, and is eligible to be er | |

DD

MMM

Investigator's Signature


| | Source D | Documents | | | 1 450 10 011 |
|---|---|---|---|---|---|
| | | | | Subject | nitials |
| Galderma | Study # C16-CD020 | INVESTIGTO | R NAME | | |
| | , | To be added | d per site | | |
| | | | | Subject I | Number |
| | | SITE NUMB | ER | | |
| | | To be added | d per site | | |
| Visit 2 –Baseline | | Visit Date | e: | | |
| | | | DD-MM | 1M-YYYY | |
| Check In Procedures | | | | | |
| Has the subject cleansed t | heir face and removed all | l makeup at le | ast 30 minute | es prior? | |
| ☐ Yes ☐ No | (If no, subject needs to re | emove residua | I makeup and | d acclimate | e 20 minutes) |
| Review of Adverse Events | | | | | |
| Has the subject experience | | nedical proble | ms since thei | ir last visit | ? |
| ☐ Yes (If yes, record on Al | E page) 🔲 No | | | | |
| Has the subject started or | | | ion since the | ir last visit | , |
| $\square$ Yes (If yes, record on M | ledications page) | No | | | |
| Has the subject had any p | | | visit? | | |
| ☐ Yes (If yes, record on M | ledications page) □ | No | | | |
| Acclimation | | | | | |
| *Reminder: Subject must | acclimate for at least 15 r | minutos in tom | porature of 6 | 50 7E°E an | d rolativo |
| humidity range 35-65% be | | | | | u relative |
| | | s, and photog | гарпу ргосец | ures. | |
| Acclimation start time : | :AM/PM | Acclimation | end time : | <b>:</b> | AM/PM |
| Technician initials: | Date( | DD-MMM-YYYY):_ | | | _ |
| Qualification Criteria (cor | nfirm that subject still me | eets eligibility | criteria) | | |
| Subject must have mild to | o moderate facial acne (se | core of 2-3 on | FDA Investig | ator's Glo | bal |
| Assessment Scale, at least | t 5 inflammatory lesions, | and 10-100 n | on-inflamma | tory lesio | ns |
| Does the subject have mile | • | | | ore: | □No |
| Does the subject have at l | | | ☐ Yes (>5) * | * | □No |
| Does the subject have 10 − 100 non-inflammatory lesions? ☐ Yes (10-100) * ☐ No | | | | | |
| *If yes, please fill out lesion | | | - | | |
| Evaluator's initials: | Date( | DD-MMM-YYYY): | | | |

| Source Documents | | |
|---|---|---|
| Galderma Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | Subject Number |
| | SITE NUMBER | |
| | To be added per site | |

#### Visit 2 -Baseline

| Lesion | Count |
|--------|-------|
|--------|-------|

A trained grader will count and record the number of open comedones, closed comedones, papules, and pustules on each subject's face. Note that papules and pustules are classified as inflammatory acne lesions while open and closed comedones are classified as non-inflammatory lesions.

\*Lesions on the nose, under the jaw line or along the hairline (including eye brows) will not be included in the counts.

| Parameter | Forehead<br>Enter 2 digits<br>for all scores (ie<br>05, 10, 20) | | Enter 2 digits for all scores (ie for all scores | | Chin<br>Enter 2 digits for<br>all scores (ie 05,<br>10, 20) | | Enter 2 digits for all scores (ie 05, | | Enter 2 digits for all scores (ie 05, | | Right (<br>Enter 2 d<br>all score<br>10, | ligits for<br>s (ie 05, | Total<br>3 digits<br>s (ie 050<br>100) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Open Comedones | | | | | | | | | | | | | |
| Closed<br>Comedones | | | | | | | | | | | | | |
| Papules | | | | | | | | | | | | | |
| Pustules | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | |
| Evaluator's initials:_ | | 1 | | Date( | DD-MMM- | -YYYY): | | 1 | | I | | | |

| Investigator <sup>,</sup> | 's Global | Assessment | (IGA) |
|---------------------------|-----------|------------|-------|
| investigator | SCHODAL | Assessment | UGAL |

A trained grader will evaluate each subject's global face for Investigator's Global Improvement Assessment.

#### Scale:

| 0 | Clear | No inflammatory or non-inflammatory lesions |
|---|---|---|
| 1 | Almost Clear | Rare non-inflammatory lesions with no more than one small inflammatory |
| | | lesion |
| 2 | Mild | Greater than Grade 1, some non-inflammatory lesions with no more than a |
| | | few inflammatory lesion (papules/pustules only, no nodular lesions) |
| 3 | Moderate | Greater than Grade 2, up to many non-inflammatory lesions and may have |
| | | some inflammatory lesions, but no more than one small nodular lesion |
| 4 | Severe | Greater than Grade 3, up to many non-inflammatory and inflammatory |
| | | lesions, but no more than a few nodular lesions |

| Parameter | Global Face Enter 1 digit for all scores (ie 1, 2, 3) |
|---|---|
| IGA | |
| Evaluator's initials:_ | Date(DD-MMM-YYYY): |


| | | Sourc | n Do | cuments | | | | rage | 12 01 3 |
|---|---|---|---|---|---|---|---|---|---|
| | | 30010 | .6 00 | Cuments | | | Subject | Initials | |
| Galderma | Study | # C16-CD020 | | INVESTIGT | ΩR | ΝΔΜΕ | Jubject | IIIItiais | |
| - Caracinia | Study | | | To be adde | | | | | |
| | | | | | - C | - | Subject | Number | |
| | | | | SITE NUMBER | | | | | |
| | | | | To be added per site | | er site | | | |
| Visit 2 –Baseline | | | • | | | | | | |
| *Tolerability Instructions: | Local c | utaneous tolera | abilit | ty will be ev | alu | ated by asse | essing the | e signs a | nd |
| symptoms of erythema, dr | | | | | | | | _ | |
| stinging/burning on the glo | obal fac | e (treatment ai | rea). | (Half-point | sco | ores may be | used as | necessa | ry to |
| more accurately describe t | he skin | condition): 0 = | non | e, 1 = mild, | 2 = | moderate, | 3 = seve | re | |
| Parameter | | | | | | Face | | | |
| | Enter 2 digits for all scores (ie 0.5, 1.0, 2.0) | | | | | | | | |
| Erythema | | | | | • | | | | |
| Dryness | | | | | • | | | | |
| Scaling | | | | | • | | | | |
| Burning/Stinging | | | | | • | | | | |
| Evaluator's initials: | | Dat | te(DD | D-MMM-YYYY) | ): | | | | |
| VISIA Imaging – 1 2 3 St | ephens | TX site only, d | elete | e if not nee | ded | | | | |
| *Reminder: Subject must | have a d | clean face (no n | nake | up) and all | jew | elry remove | d. Subje | ct must | be |
| wearing a black or gray ma | atte hea | dband to keep | hair | away from | the | e face. Subje | ct must | be wear | ing a |
| black matte shirt or drape | | | | | | | bjects m | ust have | e a |
| neutral, non-smiling expre | ssion w | ith their eyes g | ently | y closed in a | all p | ictures. | | | |
| Please mark the box for ea | ch phot | to that was take | en. Ij | lf one was n | ot | taken, leave | box unn | narked. | |
| <u>Left View:</u> | | | ter V | | | | Right V | | |
| ☐ Standard Lighting 1 (vis | | ☐ Standard Li | _ | _ | | ☐ Standa | _ | _ | |
| ☐ Standard Lighting 2 (visi | ible) | ☐ Standard Lighting 2 (visible) | | | ☐ Standa | _ | ng 2 (vis | ible) | |
| □Cross Polarized | | □Cross Polari | | _ | | □Cross P | | | |
| □Parallel Polarized | | □Parallel Pola | | | | □Parallel | | | |
| ☐ UV Fluorescence | | ☐ UV Fluorescence | | | □UV Fluc | | e | | |
| Seat height: cm | | | | adrest: 1 | 2 | 3 (circle | one) | | |

Technician initials:\_\_\_\_\_ Time: \_\_\_\_:\_\_AM/PM Date(DD-MMM-YYYY):\_\_\_\_\_


| | Source Documents | | | | | | |
|---|---|---|---|---|---|---|---|
| Galderma | Studv | # C16-CD020 | INVEST | IGTOR NAME | Subject | Initials | |
| | 3.5.5.7 | ==0 0=0=0 | _ | dded per site | | | |
| | | | | | Subject | Number | |
| | | | SITE NU | | | | |
| | | | L . | dded per site | | | |
| Visible Light Imaging (Bea | _ | | | | | | |
| For subjects completing at | | | | | | _ | will |
| be taken of each subject's | | | | | | • | |
| center view. Subjects will | | | | | chinrest. | Subjects | will |
| be instructed to adopt neu | | | | | | | |
| Please mark the box for ed | ich phot | to that was taken. | If one w | as not taken, leave | e box unn | narked. | |
| <u>Center View:</u> | | Coat boig | h+. | Camar | o bolabti | | |
| ☐ Visible light | | Seat heig | nt: | _ Camer | nera height: | | |
| Technician initials: | т | ime:: <i>F</i> | AM/PM | Date(DD-MMM-YY | YY): | | |
| Product Distribution | | | | | | | |
| 1 Todact Distribution | | | | | | | |
| Randomization Group: A | B (circl | le one) | | | | | |
| Was the subject provided | | • | perly us | e the study produ | cts? | ☐ Yes | □ No |
| Was the subject provided | | • | · · · | | | ☐ Yes | □ No |
| Was the subject instructed visit? | Was the subject instructed to bring back the dispensed study products at the next visit? ☐ Yes ☐ No | | | | | | |
| Technician initials: | T | ime:: | AM/PM | Date(DD-MMM-YY | YY): | | |

| | | | Page <b>14</b> of <b>3</b> |
|---|---|---|---|
| | Source D | ocuments | |
| | | | Subject Initials |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME | |
| | , | To be added per site | |
| | | · | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |
| Visit 3 – Week 1 | <u>I</u> | Visit Date: - | - |
| | | | <br>1M-YYYY |
| | | 22 1111 | |
| Check In Procedures | | | |
| Has the subject cleansed t | heir face and removed all | makeup at least 30 minute | es prior? |
| _ | | move residual makeup and | - |
| | , , | · | , |
| Have the subject's test ma | nterials been visually inspe | ected and weighed? Record w | veights in Test Material Sheet |
| ☐ Yes ☐ No | | J | |
| Has the subject's diary bee | en reviewed for compliand | ce? | |
| ☐ Yes ☐ No | · | | |
| Has the subject been instr | ucted to bring back the di | spensed study products at | the next visit? |
| ☐ Yes ☐ No | _ | spensed stady products at | the field viole. |
| 2.163 | | | |
| Review of Adverse Events | | | |
| | | nedical problems since thei | ir last visit? |
| ☐ Yes (If yes, record on Al | | ilculcul problems since the | ii last visit: |
| Tes (ii yes, record on Ai | - page) — No | | |
| Has the subject started or | discontinued any concorr | nitant medication since the | ir lact vicit? |
| ☐ Yes (If yes, record on M | • | | וו ומגנ עוגונ: |
| Tes (ii yes, record oii ivi | edications page) | NO | |
| Has the subject had any p | racaduras ar traatmants s | inco thoir last visit? | |
| ☐ Yes (If yes, record on Medications page) ☐ No | | | |
| Acclimation | | | |
| | acclimate for at least 15 :- | ninutas in tananaraturs =£ ( | CO 75°5 and relative |
| _ | | ninutes in temperature of 6 | |
| number of the following from the | nore starting assessments | s, and photography proced | iures. |

Technician initials:\_\_\_\_\_\_ Date(DD-MMM-YYYY):\_\_\_\_\_

Acclimation end time :\_\_\_\_\_:\_\_AM/PM

Acclimation start time :\_\_\_\_\_:\_\_AM/PM

| | | | | | | | | | | | Pa | age <b>15</b> | of <b>38</b> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | S | ource [ | Oocumer | nts | | | | | |
| | | | | | | | | | | Subjec | ct Initia | ls | |
| Galderma | | Study # C16-CD020 | | INVES | TIGTOR | NAME | | | | | | | |
| | | | | | | | To be | added p | er site | | | | |
| | | | | | | | | | | Subjec | ct Num | ber | |
| | | | | | | | SITE N | IUMBER | | | | | |
| | | | | | | | | added p | | | | | |
| <u>Visit 3 –</u> | <u>Visit 3 – Week 1</u> Visit Date: | | | | | | | | | | | | |
| | DD-MMM-YYYY | | | | | | | | | | | | |
| Lesion C | Count | | | | | | | | | | | | |
| A traine | d grade | er wil | l count | and reco | rd the n | umber | of open | comedoi | nes, close | d comed | ones, p | apules | , and |
| pustules | s on eac | ch su | bject's | face. Not | e that pa | apules a | and pust | ules are | classified | as inflan | nmator | y acne | |
| lesions v | while o | pen a | nd clos | sed come | dones ar | re class | ified as r | non-infla | mmatory | lesions. | | | |
| *Lesions | s on the | nose | e, unde | r the jaw | line or a | long th | e hairlin | e (includ | ing eye br | ows) wil | l not | | |
| be includ | ded in t | he co | ounts. | - | | | | • | | • | | | |
| | | | For | ehead | Left C | heek | Ch | nin | Right ( | Cheek | | Total | |
| Para | ameter | | | 2 digits | Enter 2 | - | | digits for | Enter 2 c | • | Enter 3 digits for al | | |
| | | | | scores (ie | for all s | | | es (ie 05, | all score | - | score | (ie 050 | , 099, |
| | | | 05, | 10, 20) | (ie 05, 1 | 10, 20) | 10, | 20) | 10, | 20)<br> | | 100) | |
| Open C | | nes | | | | | | | | | | | |
| | osed | | | | | | | | | | | | |
| Com | edones | 5 | | | | | | | | | | | |
| Pa | pules | | | | | | | | | | | | |
| Pu | stules | | | | | | | | | | | | |
| Т | otal | | | | | | | | | | | | |
| Evaluato | or's init | ials:_ | | | | Date( | DD-MMM- | -YYYY): | | | | • | |
| Investig | ator's ( | Globa | al Asses | ssment (I | GA) | | | | | | | | |
| | | | | - | | glohal | face for | Investiga | ator's Glo | hal Impr | ovemer | nt | |
| Assessm | _ | <b></b> | CVara | ate edem | oubject 5 | Biobai | race ror | iii v estigi | 2001 3 010 | our impri | Overrier | | |
| Scale: | 10110. | | | | | | | | | | | | |
| Scare. | 0 | Clea | ır | No ir | ıflammatı | orv or n | on-inflam | matory le | esions | | | | $\overline{}$ |
| | 1 | | ost Clea | | | | | | nore than | one smal | l inflamı | natorv | |
| | | | | lesio | | | , | | | | | , | |
| | 2 | Milo | t | Grea | ter than ( | Grade 1, | some no | n-inflamr | natory lesi | ons with | no more | than a | 3 |
| | | | | few inflammatory lesion | | | | les/pustu | les only, n | o nodular | lesions) | ) | |
| | 3 | Mod | loderate Greater than Grade 2, up to many non-inflammatory lesions and may | | | | | | • | | | | |
| | | | some inflammatory lesions, but no more than one small nodular lesion were Greater than Grade 3, up to many non-inflammatory and inflammatory | | | | | | | | | | |
| | 4 | Seve | ere | l l | | | | | | ry and inf | flammat | ory | |
| | | | | lesio | ns, but no | more | nan a iev | v nodular | lesions | | | | |
| Para | meter | | | | | | | obal Fac | | | | | |
| | | | | | | Ente | er 1 digit f | or all score | es (ie 1, 2, 3 | ) | | | |
| IGA | | | | | | | | | | | | | |
| Evaluato | Evaluator's initials: Date(DD-MMM-YYYY): | | | | | | | | | | | | |


| | | | | Page . | 10 01 3 |
|---|---|---|---|---|---|
| | Source I | Documents | | | |
| | | Subject Initials | | | |
| Galderma | Study # C16-CD020 | INVESTIGTO | R NAME | | |
| | • | To be added | per site | | |
| | | | | Subject Number | |
| | | SITE NUMBE | R | | |
| | | To be added | per site | | |
| Visit 3 – Week 1 | 1 | | p = 1 = 1 = 1 | <u>. l</u> | |
| *Tolerability Instructions: | Local cutaneous tolerab | ility will be eval | uated by as | sessing the signs an | ıd |
| symptoms of erythema, d | ryness, and scaling, and b | y subject repor | ting of the | degree of | |
| stinging/burning on the gl | obal face (treatment area | a). (Half-point s | cores may b | e used as necessary | / to |
| more accurately describe | the skin condition): 0 = no | one, 1 = mild, 2 | = moderate | e, 3 = severe | |
| D | Global Face | | | | |
| Parameter | Enter 2 digits for all scores (ie 0.5, 1.0, 2.0) | | | | |
| Erythema | | . | , | | |
| Dryness | | | , | | |
| Scaling | | | | | |
| Burning/Stinging | | | , | | |
| Francisco de la | Data | (55.44.44.40.44) | | | |
| Evaluator's initials: | Date( | [DD-MMM-YYYY):_ | | | |
| Self-Assessment Question | naire | | | | |
| Has the subject completed | the self-assessment que | estionnaire? | | ☐ Yes ☐ N | lo |
| • | · | | | <u> </u> | |
| Technician initials: | nician initials: Date(DD-MMM-YYYY): | | | | |

|---|---|---|---|
| | Source D | ocuments | |
| | | | Subject Initials |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME | |
| | | To be added per site | |
| | | | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |
| Visit 4 – Week 2 | | Visit Date: | |
| | | DD-MMN | 1-YYYY |
| Check In Procedures | | | |
| Has the subject cleansed t | heir face and removed all | makeup at least 30 minute | es prior? |
| ☐ Yes ☐ No | (If no, subject needs to re | move residual makeup and | d acclimate 20 minutes) |
| Have the subject's test ma | aterials been visually inspe | ected and weighed? Record v | veights in Test Material Sheet |
| ☐ Yes ☐ No | | | |
| Has the subject's diary be | • | ce? | |
| ☐ Yes ☐ No | | | |
| • | _ | spensed study products at | the next visit? |
| ☐ Yes ☐ No | | | |
| Review of Adverse Events | • | | _ |
| | | nedical problems since the | ir last visit? |
| ☐ Yes (If yes, record on Al | | realear problems since the | ii idst visit: |
| = 1e3 (ii ye3, 1ecord oii 7ii | L puge/ — 110 | | |
| Has the subject started or | discontinued any concom | nitant medication since the | ir last visit? |
| ☐ Yes (If yes, record on M | • | No | |
| ( | | | |
| Has the subject had any procedures or treatments since their last visit? | | | |
| ☐ Yes (If yes, record on M | ledications page) | No | |
| , , . | , , | | |
| Acclimation | | | |
| *Reminder: Subject must | acclimate for at least 15 n | ninutes in temperature of | 68-75°F and relative |
| humidity range 35-65% be | efore starting assessments | s, and photography proced | lures. |
| Acclimation start time : | :AM/PM | Acclimation end time : | :AM/PM |
| | I | | |

Date(DD-MMM-YYYY):\_

Technician initials:\_\_\_\_

| | | | 1 agc 10 01 30 |
|---|---|---|---|
| | Source | Documents | |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | SITE NUMBER | Subject Number |
| Visit 4 – Week 2 | | To be added per site | |

#### **Lesion Count**

A trained grader will count and record the number of open comedones, closed comedones, papules, and pustules on each subject's face. Note that papules and pustules are classified as inflammatory acne lesions while open and closed comedones are classified as non-inflammatory lesions.

\*Lesions on the nose, under the jaw line or along the hairline (including eye brows) will not be included in the counts.

| Parameter | Enter 2 digits Er for all scores (ie fo | | Left Cheek<br>Enter 2 digits<br>for all scores<br>(ie 05, 10, 20) | | Enter 2 o | Chin<br>Enter 2 digits for<br>all scores (ie 05,<br>10, 20) | Enter 2 digits for Enter 3 | Total<br>3 digits<br>s (ie 050<br>100) | |
|---|---|---|---|---|---|---|---|---|---|
| Open Comedones | | | | | | | | | |
| Closed<br>Comedones | | | | | | | | | |
| Papules | | | | | | | | | |
| Pustules | | | | | | | | | |
| Total | | | | | | | | | |
| Evaluator's initials:_ | | 1 | | Date( | DD-MMM- | -YYYY): | 1 | | 1 |

| Investigator's Global Asse | ssment (IGA) |
|----------------------------|--------------|
|----------------------------|--------------|

A trained grader will evaluate each subject's global face for Investigator's Global Improvement Assessment.

### Scale:

| 0 | Clear | No inflammatory or non-inflammatory lesions |
|---|---|---|
| 1 | Almost Clear | Rare non-inflammatory lesions with no more than one small inflammatory |
| | | lesion |
| 2 | Mild | Greater than Grade 1, some non-inflammatory lesions with no more than a |
| | | few inflammatory lesion (papules/pustules only, no nodular lesions) |
| 3 | Moderate | Greater than Grade 2, up to many non-inflammatory lesions and may have |
| | | some inflammatory lesions, but no more than one small nodular lesion |
| 4 | Severe | Greater than Grade 3, up to many non-inflammatory and inflammatory |
| | | lesions, but no more than a few nodular lesions |

| Parameter | Global Face Enter 1 digit for all scores (ie 1, 2, 3) |
|---|---|
| IGA | |
| Evaluator's initials:_ | Date(DD-MMM-YYYY): |

|---|---|---|---|---|---|---|---|---|
| | Source D | Documents | | | | | | |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME | | | Subject | Init | ials | |
| | | To be adde | a b | er site | <u> </u> | <u>—</u> | | |
| | | SITE NUME | יבט | 1 | Subject | Nur | mber | , |
| | | To be adde | | - | <b> </b> | | | |
| Visit 4 – Week 2 | | To be adde | ։ս բ | Jei site | | | | |
| VISIL 4 - VVCCK Z | | | | | | | | |
| *Tolerability Instructions:<br>symptoms of erythema, dry<br>stinging/burning on the glo<br>more accurately describe the | yness, and scaling, and bobbal face (treatment area | y subject repo<br>a). (Half-point | orti<br>scc | ing of the dores may be | egree of e used as | nec | - | |
| Parameter | Global Face | | | | | | | |
| raiailletei | Enter 2 digits for all scores (ie 0.5, 1.0, 2.0) | | | | | | | |
| Erythema | | | • | | | | | |
| Dryness | | | • | | | | | |
| Scaling | | | • | | | | | |
| Burning/Stinging | | | • | | | | | |
| Evaluator's initials: | Date( | DD-MMM-YYYY) | : | | | | | |
| Self-Assessment Question | naire | | | | | | | |
| Has the subject completed | the self-assessment que | stionnaire? | | | ☐ Yes | ; | | No |
| Technician initials: Date(DD-МММ-YYYY): | | | | | | | | |

| | | | Page <b>20</b> of <b>3</b> |
|---|---|---|---|
| Source Documents | | | |
| | | Subject Initials | |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME | |
| | | To be added per site | |
| | | | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |
| Visit 5 – Week 6 | | Visit Date: - | - |
| | | DD-MMN | <del></del> |
| Check In Procedures | | | |
| | heir face and removed al | l makeup at least 30 minut | es prior? |
| _ | | emove residual makeup an | - |
| | (ii iio) subject fields to re | and the residual makeup and | a dominate 20 minutes; |
| Have the subject's test ma | aterials heen visually inso | ected and weighed? Record v | voights in Tost Material Shoot |
| ☐ Yes ☐ No | · · · | ected and weighted: Record | veignts in Test Material Sheet |
| Lifes Lino | | | |
| Has the subject's diary be | on ravioused for complian | co2 | |
| ☐ Yes ☐ No | | ce: | |
| Li res Li No | | | |
| Harris I de la | | | |
| Has the subject been give | - | | |
| ☐ Yes ☐ No | | | |
| | | ispensed study products at | the next visit? |
| ☐ Yes ☐ No | | | |
| Review of Adverse Events | <b>;</b> | | |
| Has the subject experience | ed an Adverse Events or r | nedical problems since the | ir last visit? |
| ☐ Yes (If yes, record on Al | E page) □ No | | |
| Has the subject started or | discontinued any concon | nitant medication since the | ir last visit? |
| ☐ Yes (If yes, record on M | ledications page) $\Box$ | No | |
| | , . | | |
| Has the subject had any procedures or treatments since their last visit? | | | |
| ☐ Yes (If yes, record on M | | No | |
| Li 163 (ii yes, record oii Medications page) | | | |
| Acclimation | | | |
| | acclimate for at least 15 r | minutes in temperature of | 68-75°E and relative |
| • | | • | |
| humidity range 35-65% before starting assessments, and photography procedures. | | | |
| Acclimation start time : | :AM/PM | Acclimation end time : | :AM/PM |

Date(DD-MMM-YYYY):\_

Technician initials:\_


| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |

### Visit 5 – Week 6

| <u></u> | | |
|---|---|---|
| VISIA Imaging | | |
| *Reminder: Subject must have a | clean face (no makeup) and all jewe | elry removed. Subject must be |
| wearing a black or gray matte hea | dband to keep hair away from the | face. Subject must be wearing a |
| black matte shirt or draped with a | a black or gray matte cloth to hide o | lothing. Subjects must have a |
| neutral, non-smiling expression w | ith their eyes gently closed in all pi | ctures. |
| Please mark the box for each pho | to that was taken. If one was not to | aken, leave box unmarked. |
| <u>Left View:</u> | Center View: | Right View: |
| ☐ Standard Lighting 1 (visible) | ☐ Standard Lighting 1 (visible) | ☐ Standard Lighting 1 (visible) |
| ☐ Standard Lighting 2 (visible) | ☐ Standard Lighting 2 (visible) | ☐ Standard Lighting 2 (visible) |
| □Cross Polarized | □Cross Polarized | □Cross Polarized |
| □Parallel Polarized | □Parallel Polarized | □Parallel Polarized |
| ☐ UV Fluorescence | ☐ UV Fluorescence | ☐ UV Fluorescence |
| Seat height: cm | Headrest: 1 2 | 3 (circle one) |
| Technician initials: T | ime::AM/PM | D-MMM-YYYY): |

| | | | . ugc == 0. <b>00</b> |
|---|---|---|---|
| | Source | Documents | |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |
| Visit 5 – Week 6 | | | |

#### **Lesion Count**

A trained grader will count and record the number of open comedones, closed comedones, papules, and pustules on each subject's face. Note that papules and pustules are classified as inflammatory acne lesions while open and closed comedones are classified as non-inflammatory lesions.

\*Lesions on the nose, under the jaw line or along the hairline (including eye brows) will not be included in the counts.

| Parameter | Forehead<br>Enter 2 digits<br>for all scores (ie<br>05, 10, 20) | Left Cheek Enter 2 digits for all scores (ie 05, 10, 20) | | Chin<br>Enter 2 digits for<br>all scores (ie 05,<br>10, 20) | | Right Cheek<br>Enter 2 digits for<br>all scores (ie 05,<br>10, 20) | Total<br>Enter 3 digits for<br>scores (ie 050, 09<br>100) |
|---|---|---|---|---|---|---|---|
| Open Comedones | | | | | | | |
| Closed<br>Comedones | | | | | | | |
| Papules | | | | | | | |
| Pustules | | | | | | | |
| Total | | | | | | | |
| Evaluator's initials: | | | Date( | DD-MMM- | -YYYY): | | |

| Investigator's Global Assessment | (IGA) |
|----------------------------------|-------|
|----------------------------------|-------|

A trained grader will evaluate each subject's global face for Investigator's Global Improvement Assessment.

### Scale:

| 0 | Clear | No inflammatory or non-inflammatory lesions |
|---|---|---|
| 1 | Almost Clear | Rare non-inflammatory lesions with no more than one small inflammatory |
| | | lesion |
| 2 | Mild | Greater than Grade 1, some non-inflammatory lesions with no more than a |
| | | few inflammatory lesion (papules/pustules only, no nodular lesions) |
| 3 | Moderate | Greater than Grade 2, up to many non-inflammatory lesions and may have |
| | | some inflammatory lesions, but no more than one small nodular lesion |
| 4 | Severe | Greater than Grade 3, up to many non-inflammatory and inflammatory |
| | | lesions, but no more than a few nodular lesions |

| Parameter | | Global Face Enter 1 digit for all scores (ie 1, 2, 3) |
|---|---|---|
| IGA | | |
| Evaluator's initials:_ | D | Oate(DD-MMM-YYYY): |

| | | | | | | Page 2 | : <b>3</b> of 3 |
|---|---|---|---|---|---|---|---|
| | Source [ | Documents | | | | | |
| Galderma | Study # C16-CD020 | | INVESTIGTOR NAME To be added per site | | | tials | |
| | | | Ċ | | Subject Nu | mber | |
| | | SITE NUMB | ER | | | | |
| | | To be adde | d p | er site | | | |
| Visit 5 – Week 6 | | | | | | | |
| *Tolerability Instructions:<br>symptoms of erythema, dr<br>stinging/burning on the glo<br>more accurately describe t | yness, and scaling, and bobal face (treatment area | y subject repo<br>a). (Half-point | orti<br>scc | ng of the dores may be | egree of<br>e used as ned | | |
| Parameter | Ent | Global Face Enter 2 digits for all scores (ie 0.5, 1.0, 2.0) | | | | | |
| Erythema | | | • | | | | |
| Dryness | | | • | | | | |
| Scaling | | | • | | | | |
| Burning/Stinging | | | • | | | | |
| Technician initials: | Date (DD-MMM-YYYY | ·): | | | | | |
| <b>Self-Assessment Question</b> | naire | | | | | | |
| Has the subject completed | the self-assessment que | estionnaire? | | | ☐ Yes | | כ |
| Technician initials: | Date(I | DD-MMM-YYYY): | | | | | |


| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site SITE NUMBER To be added per site | Subject Initials Subject Number |
| Follow-up Phone Call (bet | ween Week 6 and Week | • | |
| Review of Adverse Events | | - | |
| Has the subject experienced an Adverse Events or medical problems since their last visit? ☐ Yes (If yes, record on AE page) ☐ No Has the subject started or discontinued any concomitant medication since their last visit? ☐ Yes (If yes, record on Medications page) ☐ No | | | |
| • | Has the subject had any procedures or treatments since their last visit? ☐ Yes (If yes, record on Medications page) ☐ No | | |
| Does the subject have end ☐ Yes ☐ No | Does the subject have enough study product to until the next study visit? ☐ Yes ☐ No | | |
| Technician initials: | Date(D | D-MMM-YYYY): | |

| | | | Page <b>25</b> of <b>3</b> |
|---|---|---|---|
| | Source D | ocuments | |
| | | | Subject Initials |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME | |
| | | To be added per site | |
| | | | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |
| Visit 6 – Week 12 | | Visit Date: | <u>-</u> |
| | | DD-MMM | 1-YYYY |
| Check In Procedures | | | |
| Has the subject cleansed t | heir face and removed all | makeup at least 30 minute | es prior? |
| ☐ Yes ☐ No | (If no, subject needs to re | move residual makeup and | d acclimate 20 minutes) |
| Have the subject's test ma | aterials been visually inspe | cted and weighed? Record w | veights in Test Material Sheet |
| ☐ Yes ☐ No | | _ | |
| Has the subject's diary bee | en reviewed for complianc | e? | |
| □ Yes □ No | | | |
| Has the subject been given | n a new diary? | | |
| ☐ Yes ☐ No | | | |
| Lifes Lino | | | |
| Has the subject been instr | usted to bring back the div | spansod study products at | the next visit? |
| ☐ Yes ☐ No | _ | spensed study products at | the next visit: |
| □ Yes □ NO | | | |
| Davies of Advance France | | | |
| Review of Adverse Events | | | |
| Has the subject experience | | iedical problems since the | ir last visit? |
| ☐ Yes (If yes, record on Al | E page) 🔲 No | | |
| Has the subject started or | - | | ir last visit? |
| ☐ Yes (If yes, record on M | ledications page) 🗆 🗆 I | No | |
| Has the subject had any p | rocedures or treatments si | ince their last visit? | |
| ☐ Yes (If yes, record on M | ledications page) □ [ | No | |
| · · · · · · | | | |
| Acclimation | | | |
| *Reminder: Subject must | acclimate for at least 15 m | ninutes in temperature of 6 | 68-75°F and relative |
| humidity range 35-65% be | | | |
| | _ | | |
| Acclimation start time : | :AM/PM | Acclimation end time : | :AM/PM |

Date(DD-MMM-YYYY):\_

Technician initials:\_


| | | Source Do | ocuments | | | | |
|---|---|---|---|---|---|---|---|
| | | | | | Subject | Initials | |
| Galderma | Study | # C16-CD020 | INVESTIGTOR N | IAME | | | |
| | | | To be added pe | er site | | | |
| | | | | - | Subject | Number | • |
| | | | SITE NUMBER | | | | |
| | | | To be added pe | er site | | | |
| Visit 6 – Week 12 | | | | | | | |
| VISIA Imaging | | | | | | | |
| *Reminder: Subject must | have a d | clean face (no make | eup) and all jewe | lry remove | ed. Subje | ct must | be |
| wearing a black or gray ma | atte hea | dband to keep hair | r away from the | face. Subje | ect must l | be wear | ing a |
| black matte shirt or drape | d with a | black or gray matt | te cloth to hide c | lothing. Su | ıbjects m | ust have | e a |
| neutral, non-smiling expre | ssion w | ith their eyes gentl | y closed in all pion | ctures. | | | |
| Please mark the box for ed | ich phot | to that was taken. | If one was not to | aken, leave | box unn | narked. | |
| Left View: | | <u>Center \</u> | | Right View: | | | |
| $\square$ Standard Lighting 1 (vis | ible) | ☐ Standard Light | ☐ Standard Lighting 1 (visible) | | | ible) | |
| ☐ Standard Lighting 2 (vis | ible) | ☐ Standard Light | ☐ Standard Lighting 2 (visible) | | | ible) | |
| □Cross Polarized | | □Cross Polarized | □Cross Polarized | | | | |
| ☐Parallel Polarized | | □Parallel Polarize | □Parallel Polarized | | | | |
| ☐ UV Fluorescence | | ☐ UV Fluorescend | ☐ UV Fluorescence | | | | |
| Seat height: cm | | He | adrest: 1 2 | 3 (circle | e one) | | |
| Technician initials: | т | ime: : A | AM/PM Date(D | D-MMM-YYY | w). | | |
| Tecinician iniciais | | | AIVI/PIVI Date(D | D-IVIIVIIVI-Y Y | (1) | | |
| Visible Light Imaging (Bea | uty sho | t) <mark>Stephens sites o</mark> | nly, delete if no | t needed | | | |
| For subjects completing at | sites 1 | and 2 (Stephens' T | exas and Colorad | do location | ns), digita | l images | will |
| be taken of each subject's | face us | ing visible light. Ful | II-face images wi | ll be taken | of each | subject's | 5 |
| center view. Subjects will | not be v | vearing any headba | and or using any | headrest/ | chinrest. | Subject | s will |
| be instructed to adopt neu | utral, no | n-smiling expression | ons with their ey | es open. | | | |
| Please mark the box for ed | ich phot | to that was taken. | If one was not to | aken, leave | box unn | narked. | |
| <b>Center View:</b> | | 6 | | | | | |
| ☐ Visible light | | Seat heig | nt: | Camer | a height: | | |

Time: \_\_\_\_:\_\_AM/PM Date(DD-MMM-YYYY):\_

Technician initials:\_

| | | | 1 450 =7 01 50 |
|---|---|---|---|
| | Source | Documents | |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | SITE NUMBER To be added per site | Subject Number |
| Visit 6 – Week 12 | | <u> </u> | • |

#### **Lesion Count**

A trained grader will count and record the number of open comedones, closed comedones, papules, and pustules on each subject's face. Note that papules and pustules are classified as inflammatory acne lesions while open and closed comedones are classified as non-inflammatory lesions.

\*Lesions on the nose, under the jaw line or along the hairline (including eye brows) will not be included in the counts.

| Parameter | Forehead<br>Enter 2 digits<br>for all scores (ie<br>05, 10, 20) | Left Cheek Enter 2 digits for all scores (ie 05, 10, 20) | | Chin<br>Enter 2 digits for<br>all scores (ie 05,<br>10, 20) | | Right Cheek<br>Enter 2 digits for<br>all scores (ie 05,<br>10, 20) | Total<br>Enter 3 digits for<br>scores (ie 050, 09<br>100) | |
|---|---|---|---|---|---|---|---|---|
| Open Comedones | | | | | | | | |
| Closed<br>Comedones | | | | | | | | |
| Papules | | | | | | | | |
| Pustules | | | | | | | | |
| Total | | | | | | | | |
| Evaluator's initials: | | | Date( | DD-MMM- | -YYYY): | | | • |

| Investigator's Global Asse | ssment (IGA) |
|----------------------------|--------------|
|----------------------------|--------------|

A trained grader will evaluate each subject's global face for Investigator's Global Improvement Assessment.

### Scale:

| 0 | Clear | No inflammatory or non-inflammatory lesions |
|---|---|---|
| 1 | Almost Clear | Rare non-inflammatory lesions with no more than one small inflammatory |
| | | lesion |
| 2 | Mild | Greater than Grade 1, some non-inflammatory lesions with no more than a |
| | | few inflammatory lesion (papules/pustules only, no nodular lesions) |
| 3 | Moderate | Greater than Grade 2, up to many non-inflammatory lesions and may have |
| | | some inflammatory lesions, but no more than one small nodular lesion |
| 4 | Severe | Greater than Grade 3, up to many non-inflammatory and inflammatory |
| | | lesions, but no more than a few nodular lesions |

| Parameter | | Global Face<br>Enter 1 digit for all scores (ie 1, 2, | 3) |
|---|---|---|---|
| IGA | | | |
| Evaluator's initials:_ | D | Oate(DD-MMM-YYYY): | |

| | | | | | Page <b>28</b> of <b>3</b> |
|---|---|---|---|---|---|
| | Source D | ocuments | | | |
| | | | | Subject Init | ials |
| Galderma Study # C16-CD020 INVESTIGTOR | | | RNAME | | |
| | • | To be added | per site | | |
| | | | | Subject Nu | mber |
| | | SITE NUMBER | ₹ | | |
| | | To be added | per site | | |
| Visit 6 – Week 12 | | | | | |
| *Tolerability Instructions: | Local cutaneous tolerabil | ity will be evalu | uated by asse | essing the sig | gns and |
| symptoms of erythema, dry | | • | • | • | • |
| stinging/burning on the glo | bal face (treatment area | ). (Half-point sc | ores may be | used as nec | essary to |
| more accurately describe the | ne skin condition): 0 = no | ne, 1 = mild, 2 | = moderate, | 3 = severe | |
| Parameter | Global Face | | | | |
| Parameter | Ento | Enter 2 digits for all scores (ie 0.5, 1.0, 2.0) | | | |
| Erythema | | • | | | |
| Dryness | | | | | |
| Scaling | | | | | |
| Burning/Stinging | | | | | |
| Evaluator's initials: | Date(t | DD-MMM-YYYY): | | | |
| | | · — | | | |
| Self-Assessment Question | naire | | | | |
| Has the subject completed | the self-assessment ques | stionnaire? | | ☐ Yes | □No |
| Technician initials: | Date(D | D-MMM-YYYY): | | | |


| | | | rage 23 01 3 |
|---|---|---|---|
| | Source Do | ocuments | 6 1 1 1 1 1 1 |
| Galderma | Ct. 1 # 64 C 6D020 | INIVESTICATOR ALABAS | Subject Initials |
| Galdellia | Study # C16-CD020 | INVESTIGTOR NAME | |
| | | To be added per site | |
| | | CITE AU INABED | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |
| <u>Visit 7 – Week 18</u> | | Visit Date: | |
| | | DD-MM | M-YYYY |
| Check In Procedures | | | |
| | | makeup at least 30 minute | • |
| ☐ Yes ☐ No | (If no, subject needs to rea | move residual makeup and | l acclimate 20 minutes) |
| Have the subject's test ma | aterials been visually inspe | cted and weighed? Record w | eights in Test Material Sheet |
| ☐ Yes ☐ No | | | |
| Has the subject's diary be | en reviewed for complianc | e? | |
| ☐ Yes ☐ No | | | |
| Has the subject been give | n a new diary? | | |
| ☐ Yes ☐ No | | | |
| Has the subject been instr | ucted to bring back the dis | spensed study products at | the next visit? |
| ☐ Yes ☐ No | | | |
| Review of Adverse Events | <del></del> | | |
| Has the subject experience | ed an Adverse Events or m | edical problems since thei | r last visit? |
| ☐ Yes (If yes, record on Al | E page) □ No | | |
| Has the subject started or | discontinued any concom | itant medication since thei | r last visit? |
| ☐ Yes (If yes, record on M | ledications page) □ I | No | |
| Has the subject had any p | rocedures or treatments si | ince their last visit? | |
| ☐ Yes (If yes, record on M | ledications page) 🗆 🛭 I | No | |
| | . • | | |
| Technician initials: | Date(D | D-MMM-YYYY): | |


| | Carrage D | | 1 486 30 013 |
|---|---|---|---|
| ļ | Source D | ocuments | T C 1 : |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | · | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |
| Visit 8 – Week 24 | | Visit Date: | |
| | | DD-MM | IM-YYYY |
| Check In Procedures | | | |
| Has the subject cleansed th | neir face and removed all | makeup at least 30 minut | es prior? |
| ☐ Yes ☐ No ( | (If no, subject needs to re | move residual makeup an | d acclimate 20 minutes) |
| Have the subject's test ma | terials been visually inspe | cted and weighed? Record | weights in Test Material Sheet |
| ☐ Yes ☐ No | | | |
| The the chief of the | to a difference of the co | 2 | |
| Has the subject's diary bee | n reviewed for compliand | ce? | |
| ☐ Yes ☐ No | | | |
| Review of Adverse Events | | | |
| Has the subject experience | <br>•d an Adverse Events or m | nedical problems since the | <br>Pir last visit? |
| ☐ Yes (If yes, record on AE | | roundar producting annual time | |
| , , | 1 0 7 | | |
| Has the subject started or o | discontinued any concom | itant medication since the | eir last visit? |
| ☐ Yes (If yes, record on Me | edications page) | No | |
| Has the subject had any pr | | ince their last visit? | |
| ☐ Yes (If yes, record on Me | edications page) | No | |
| Acclimation | l: | | |
| *Reminder: Subject must a | | · | |
| humidity range 35-65% bet | fore starting assessments | , and photography proced | aures. |
| Acclimation start time : | :AM/PM | Acclimation end time : | :AM/PM |
| Technician initials: | Date(D | D-MMM-YYYY): | |
| | | , | |
| Urine Pregnancy Test | | | <del></del> |
| If the subject is a female of | | | |
| Test Results | Reason Not Applicable | e Kit Lot # | Kit Expiration date |
| □ Neg □ Pos □N/A | | | |
| Technician initials: | :: | AM/PM Date(DD-MMM-Y | YYY): |


| | | Source D | ocuments | | 1 460 02 0 | |
|---|---|---|---|---|---|---|
| | | 30dree B | | | Subject Initials | |
| Galderma | Study | # C16-CD020 | INVESTIGTOR N | IVVIE | Subject illitials | |
| Caldellia | Study | # C10-CD020 | To be added pe | | | |
| | | | To be added pe | i site | Subject Number | _ |
| | | | SITE NUMBER | | Subject Number | |
| | | | To be added pe | r site | | |
| Visit 8 – Week 24 | | | To be added pe | .i site | | |
| VISICO VVCCK 24 | | | | | | |
| VISIA Imaging | | | | | | |
| *Reminder: Subject must | have a | clean face (no mak | eup) and all jewe | lry remov | ed. Subject must be | |
| wearing a black or gray ma | atte hea | dband to keep hai | r away from the | face. Subje | ect must be wearing a | |
| black matte shirt or drape | d with a | black or gray mat | te cloth to hide c | lothing. Sι | ıbjects must have a | |
| neutral, non-smiling expre | ssion w | ith their eyes gent | ly closed in all pi | ctures. | | |
| Please mark the box for ed | ich phot | to that was taken. | If one was not to | aken, leave | box unmarked. | |
| Left View: | | <u>Center</u> | View: | | Right View: | |
| ☐ Standard Lighting 1 (vis | ible) | ☐ Standard Lighting 1 (visible) | | ☐ Standard Lighting 1 (visible) | | |
| ☐ Standard Lighting 2 (vis | ible) | ☐ Standard Lighting 2 (visible) | | ☐ Standard Lighting 2 (visible) | | |
| □Cross Polarized | | □Cross Polarized | | □Cross Polarized | | |
| ☐Parallel Polarized | | □Parallel Polarized | | □Parallel Polarized | | |
| ☐ UV Fluorescence | | ☐ UV Fluorescence | | ☐ UV Fluorescence | | |
| Seat height: cm | | He | eadrest: 1 2 | 3 (circle | e one) | |
| Technician initials: | т | ime::/ | AM/PM Date(D | D-MMM-YY | YY): | _ |
| Visible Light Imaging (Bea | | | | | | |
| For subjects completing at | | The state of the s | | | | |
| be taken of each subject's | | - | | | | |
| center view. Subjects will | not be v | vearing any headb | and or using any | headrest/ | chinrest. Subjects will | |
| be instructed to adopt neu | ıtral, no | n-smiling expressi | ons with their ey | es open. | | |
| Please mark the box for ed | ich phot | to that was taken. | If one was not to | aken, leave | e box unmarked. | |
| <u>Center View:</u> ☐ Visible light | | Seat heig | ht: | Camer | a height: | |

Time: \_\_\_\_:\_\_AM/PM Date(DD-MMM-YYYY):\_

Technician initials:\_\_\_\_\_

| | Source D | ocuments | |
|----------|-------------------|----------------------|------------------|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME | Subject Initials |
| | | To be added per site | Subject Number |
| | | | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |

#### Visit 8 – Week 24

#### **Lesion Count**

A trained grader will count and record the number of open comedones, closed comedones, papules, and pustules on each subject's face. Note that papules and pustules are classified as inflammatory acne lesions while open and closed comedones are classified as non-inflammatory lesions.

\*Lesions on the nose, under the jaw line or along the hairline (including eye brows) will not be included in the counts.

| Parameter | Fore<br>Enter 2<br>for all so<br>05, 10 | 2 digits<br>cores (ie | Left Cl<br>Enter 2<br>for all s<br>(ie 05, 1 | digits<br>cores | Enter 2 d | nin<br>digits for<br>es (ie 05,<br>20) | Right (<br>Enter 2 d<br>all score<br>10, | ligits for<br>s (ie 05, | Total<br>3 digits<br>s (ie 050<br>100) |
|---|---|---|---|---|---|---|---|---|---|
| Open Comedones | | | | | | | | | |
| Closed<br>Comedones | | | | | | | | | |
| Papules | | | | | | | | | |
| Pustules | | | | | | | | | |
| Total | | | | | | | | | |
| Evaluator's initials:_ | | | | Date( | DD-MMM- | -YYYY): | | | |

| Investigator's Global Assessment (IG | iΑ | ) |
|--------------------------------------|----|---|
|--------------------------------------|----|---|

A trained grader will evaluate each subject's global face for Investigator's Global Improvement Assessment.

### Scale:

| 0 | Clear | No inflammatory or non-inflammatory lesions |
|---|---|---|
| 1 | Almost Clear | Rare non-inflammatory lesions with no more than one small inflammatory |
| | | lesion |
| 2 | Mild | Greater than Grade 1, some non-inflammatory lesions with no more than a |
| | | few inflammatory lesion (papules/pustules only, no nodular lesions) |
| 3 | Moderate | Greater than Grade 2, up to many non-inflammatory lesions and may have |
| | | some inflammatory lesions, but no more than one small nodular lesion |
| 4 | Severe | Greater than Grade 3, up to many non-inflammatory and inflammatory |
| | | lesions, but no more than a few nodular lesions |

| Parameter | Global Face Enter 1 digit for all scores (ie 1, 2, 3) |
|---|---|
| IGA | |
| Evaluator's initials:_ | Date (DD-MMM-YYYY): |

| | | | | | | | Page <b>33</b> c | )† <b>3</b> |
|---|---|---|---|---|---|---|---|---|
| | Source [ | Documents | | | | | | |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | | | Subject I | niti | als | |
| | | 10 50 4440 | . G P | ici sicc | Subject I | Mur | nher | |
| | | SITE NUME | 3ER | | Jubject . | Va. | TIDE! | $\neg$ |
| | | To be adde | ed p | er site | | | | |
| Visit 8 – Week 24 | | | | | | | | |
| *Tolerability Instructions:<br>symptoms of erythema, dry<br>stinging/burning on the glo<br>more accurately describe the | yness, and scaling, and bobal face (treatment area | oy subject repo<br>a). (Half-point | orti<br>scc | ng of the de<br>ores may be | egree of<br>e used as r | nece | | |
| Parameter | Ent | Global Face Enter 2 digits for all scores (ie 0.5, 1.0, 2.0) | | | | | | |
| Erythema | | | • | , | | | | |
| Dryness | | | • | | | | | |
| Scaling | | | • | | | | | |
| Burning/Stinging | | | • | | | | | |
| Evaluator's initials: Date (DD-MMM-YYYY): | | | | | | | | |
| Self-Assessment Question | naire | | | | | | | |
| Has the subject completed | the self-assessment que | estionnaire? | | | ☐ Yes | | □ No | |
| Technician initials: Date(DD-MMM-YYYY): | | | | | | | | |

| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |

## **Test Material Sheet**

| Kit #:<br>Date Dispensed:<br>Date Returned: | Pre-<br>Weight | Week 1 | Week 2 | Week 6 |
|---|---|---|---|---|
| Product: □A □B (check one) | g | g | g | g |
| Facial Cleanser | g | g | g | g |
| <b>Moisturizing Lotion</b> | g | g | g | g |
| Facial Moisturizer SPF 30 | g | g | g | g |
| Staff Initials / Date | | | | |

| Kit #: Date Dispensed: Date Returned: | Pre-<br>Weight | Week 12 |
|---------------------------------------|----------------|---------|
| Product: □A □B (check one) | g | g |
| Facial Cleanser | g | g |
| Moisturizing Lotion | g | g |
| Facial Moisturizer SPF 30 | g | g |
| Staff Initials / Date | | |

| Kit #:<br>Date Dispensed:<br>Date Returned: | Pre-<br>Weight | Week 18 |
|---------------------------------------------|----------------|---------|
| Product: □A □B (check one) | g | g |
| Facial Cleanser | g | g |
| Moisturizing Lotion | g | g |
| Facial Moisturizer SPF 30 | g | g |
| Staff Initials / Date | | |

| Kit #: Date Dispensed: Date Returned: | Pre-<br>Weight | Week 24 |
|---------------------------------------|----------------|---------|
| Product: □A □B (check one) | g | g |
| Facial Cleanser | g | g |
| Moisturizing Lotion | g | g |
| Facial Moisturizer SPF 30 | g | g |
| Staff Initials / Date | | |

| Kit #:<br>Date Dispensed:<br>Date Returned: | Pre-<br>Weight | Unschedul<br>ed |
|---|---|---|
| Product: □A □B (check one) | g | g |
| Facial Cleanser | g | g |
| Moisturizing Lotion | g | g |
| Facial Moisturizer SPF 30 | g | g |
| Staff Initials / Date | | |


| | Galderm | Galderma Study # C16-CD020 INVESTIGTOR NAME | | ΔΝΕ | Subject Initials | | ٦ ا | | |
|---|---|---|---|---|---|---|---|---|---|
| | Galaciiii | | Study # CIC | F-CD020 | To be added per site | | | | |
| | | | | | | | Subject | Number | |
| | | | | | SITE NUMBER | | | | |
| | | | | Adverse | To be added pe | rsite | | | <u>-</u> |
| Adverse Events FROM TIME CONSENTED UNTIL STUDY EXIT | | | | | | | | | |
| | | | | | 3 □4 □5 □_ | | | | |
| | | | | | | | | | ☐ Last Page |
| Did the sul | oject report any a | adverse ev | ents? □Yes | (complete for | m) □No (if r | o, leave t | he rest o | f the form blar | ık) |
| Adverse Even | t Onset Date DD-MMM-YYY | Cessation D | Serious | Severity | Relation to<br>Investigational<br>product | Action Ta<br>Investig<br>Prod | gational | Treatment Taken If yes, complete Concomitant medication form | Outcome |
| 1. | | | □No<br>□Yes* | □Mild □Moderate □Severe | □Reasonable possibility □No Reasonable possibility | □None □Modifi □Interru □Discon □Not Ap | pted<br>tinued | □No<br>□Yes | □Resolved □Ongoing □Fatal □Unknown |
| 2. | | | □No<br>□Yes* | □Mild □Moderate □Severe | □Reasonable possibility □No Reasonable possibility | □None □Modifi □Interru □Discon □Not Ap | ipted<br>tinued | □No<br>□Yes | □Resolved □Ongoing □Fatal □Unknown |
| 3. | | | □No<br>□Yes* | □Mild □Moderate □Severe | □Reasonable possibility □No Reasonable possibility | □None □Modifi □Interru □Discon □Not Ap | ipted<br>tinued | □No<br>□Yes | □Resolved □Ongoing □Fatal □Unknown |
| 4. | | | □No<br>□Yes* | □Mild<br>□Moderate<br>□Severe | ☐Reasonable possibility ☐No Reasonable possibility | □None □Modifi □Interru □Discon □Not Ap | ipted<br>tinued | □No<br>□Yes | □Resolved □Ongoing □Fatal □Unknown |
| | · | • | • | • | • | • | | • | |
| *Serious AEs only (must notify Sponsor within 24 hours): | | | | | | | | | |
| □Prolonge<br>□Persisten | atening<br>Hospitalization<br>d Hospitalization<br>t or Significant disa | | pacity | | | | | | |

Source Documents

□Other Medically Important Event
| | | | Page <b>36</b> of <b>38</b> |
|---|---|---|---|
| | Source | Documents | |
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | SITE NUMBER To be added per site | Subject Number |
| <b>END OF STUDY</b> | | | |
| Date of Completion or D | iscontinuation (DD-МММ-YYYY) | ) | |
| Did the subject complete | e through Visit 7? 🔲 Ye | es 🗆 No | |
| If NO, mark primary reas | on for premature withdra | awal: | |
| ☐ Voluntary Withdrawa | | | |
| ☐ Death | | | |
| ☐ Pregnancy | | | |
| ☐ Investigator decision the investigation | hat it is not the best med | ical interest of the subject | to continue participation in |
| ☐ Adverse/ Serious Adve | erse Event # | | |
| ☐ Subject not following | required study procedure | es | |
| ☐ Requires disallowed T | herapy | | |
| ☐ Lost to Follow-up | | | |
| ☐ Occurrence of relevan | t exclusion Criteria | | |


| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |
| | | SITE NUMBER | |
| | | To be added per site | |

| Contact Log | | |
|------------------------|---------------|---------------------------------|
| Initials of person | Date of | Decree for each 100 Hz 110 Hz |
| contacting the subject | contact | Reason for contact with subject |
| | (DD-MMM-YYYY) | |
| | l | |


| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site SITE NUMBER To be added per site | Subject Initials Subject Number |
| Notes Page | | To be added per site | |

| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |

| Questions | 1=Strongly<br>Agree | 2 | 3 | 4 | 5=Strongly<br>Disagree |
|---|---|---|---|---|---|
| This treatment works faster than my | | | | | |
| previous acne treatment. | | | | | |
| I feel that this treatment deep cleans and | | | | | |
| unblocks my pores. | | | | | |
| I noticed an improvement in my acne. | | | | | |
| I have noticed I had fewer breakouts than | | | | | |
| my previous treatments. | | | | | |
| I saw improvement in the overall health of | | | | | |
| my skin since starting the regimen | | | | | |
| This regimen is easy to use every day. | | | | | |
| I liked the feel of this product. | | | | | |

| Subject Initials and Date |
|---------------------------|

| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |

| Questions | 1=Strongly<br>Agree | 2 | 3 | 4 | 5=Strongly<br>Disagree |
|---|---|---|---|---|---|
| My skin is clearer skin using this treatment | | | | | |
| This treatment works faster than my | | | | | |
| previous acne treatment. | | | | | |
| I feel that this treatment deep cleans and | | | | | |
| unblocks my pores. | | | | | |
| I noticed an improvement in my acne. | | | | | |
| Strongly agree to Strongly disagree | | | | | |
| I have noticed I had fewer breakouts than | | | | | |
| my previous treatments. | | | | | |
| The areas of my skin where I used to have | | | | | |
| acne is now clear and radiant after daily | | | | | |
| treatment. | | | | | |

| Subject Initials and Date |
|---------------------------|

| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |

| Questions | 1=Strongly<br>Agree | 2 | 3 | 4 | 5=Strongly<br>Disagree |
|---|---|---|---|---|---|
| My skin is clearer skin using this treatment | | | | | |
| I feel my skin is now clear | | | | | |
| The treatment helped to reduce redness and inflammation caused by my acne. | | | | | |
| I feel that this treatment deep cleans and unblocks my pores. | | | | | |
| This treatment visually minimized my pore size. | | | | | |
| This treatment reduces my acne without leaving behind dry, flakey skin. | | | | | |
| I have noticed I had fewer breakouts than my previous treatments. | | | | | |
| My skin looks better than before | | | | | |
| I saw improvement in the overall health of my skin since starting the regimen | | | | | |
| My skin looks noticeably smoother and healthier | | | | | |
| The areas of my skin where I used to have acne is now clear and radiant after daily treatment. | | | | | |
| I feel better about my skin since I've started the treatment regimen | | | | | |
| I feel more confident since I've started the treatment | | | | | |
| What is your overall satisfaction with the regimen? | | | | | |
| I have noticed a positive difference in the appearance of my skin with this regimen. | | | | | |
| This regimen is easy to use every day. | | | | | |

| Subject Initials and Date |
|---------------------------|

| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |

| Questions | 1=Strongly<br>Agree | 2 | 3 | 4 | 5=Strongly<br>Disagree |
|---|---|---|---|---|---|
| I experienced noticeable improvement in my skin tone | | | | | |
| I experienced noticeable improvement in my skin texture | | | | | |
| I experienced noticeable improvement in my skin radiance | | | | | |
| My skin has a more youthful appearance | | | | | |
| My skin is clearer skin using this treatment | | | | | |
| I feel my skin is now clear | | | | | |
| This treatment is strong enough to give me clear, acne free skin. | | | | | |
| The treatment helped to reduce redness and inflammation caused by my acne. | | | | | |
| This treatment visually minimized my pore size. | | | | | |
| This treatment reduces my acne without leaving behind dry, flakey skin. | | | | | |
| I have noticed I had fewer breakouts than my previous treatments. | | | | | |
| My skin looks better than before | | | | | |
| This treatment breaks my cycle of acne and keeps my skin clear | | | | | |
| I saw improvement in the overall health of my skin since starting the regimen | | | | | |
| My skin looks noticeably smoother and healthier | | | | | |
| The areas of my skin where I used to have acne is now clear and radiant after daily | | | | | |
| treatment. | | | | | |
| I feel better about my skin since I've started | | | | | |
| the treatment regimen | | | | | |
| I feel more confident since I've started the treatment | | | | | |

| Subject Initials and Date |
|---------------------------|

| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |

# Week 12 (cont.)

| Questions | 1=Strongly<br>Agree | 2 | 3 | 4 | 5=Strongly<br>Disagree |
|---|---|---|---|---|---|
| Has your quality of life improved now that you have started using this product? | | | | | |
| What is your overall satisfaction with the regimen? | | | | | |
| I have noticed a positive difference in the appearance of my skin with this regimen. | | | | | |
| I would recommend this product to others. | | | | | |
| My acne is as clear as if I went to a doctor or received a prescription. | | | | | |
| I don't feel the need for a prescription after using this product. | | | | | |
| Do you feel this treatment is designed for you? | | | | | |
| Do you feel more positive and less frustrated about your acne and your skin since starting this treatment? | | | | | |
| Do you feel this treatment meets the needs of your skin? | | | | | |

| Subject Initials and Date |
|---------------------------|

| | Source D | ocuments | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |

| Questions | 1=Strongly<br>Agree | 2 | 3 | 4 | 5=Strongly<br>Disagree |
|---|---|---|---|---|---|
| I experienced noticeable improvement in my skin tone | | | | | |
| I experienced noticeable improvement in my skin texture | | | | | |
| I experienced noticeable improvement in my skin radiance | | | | | |
| My skin has a more youthful appearance | | | | | |
| My skin is clearer skin using this treatment | | | | | |
| I feel my skin is now clear | | | | | |
| This treatment is strong enough to give me clear, acne free skin. | | | | | |
| The treatment helped to reduce redness and inflammation caused by my acne. | | | | | |
| This treatment visually minimized my pore size. | | | | | |
| I noticed an improvement in my acne. Strongly agree to Strongly disagree | | | | | |
| This treatment reduces my acne without leaving behind dry, flakey skin. | | | | | |
| I have noticed I had fewer breakouts than my previous treatments. | | | | | |
| My skin looks better than before | | | | | |
| This treatment breaks my cycle of acne and keeps my skin clear | | | | | |
| I saw improvement in the overall health of my skin since starting the regimen | | | | | |
| The areas of my skin where I used to have acne is now clear and radiant after daily | | | | | |
| treatment. | | | | _ | |
| I feel better about my skin since I've started the treatment regimen | | | | | |

| Subject Ir | itials and | Date |
|------------|------------|------|

| Source Documents | | | |
|---|---|---|---|
| Galderma | Study # C16-CD020 | INVESTIGTOR NAME To be added per site | Subject Initials |
| | | | Subject Number |

# Week 24 (cont.)

| Questions | 1=Strongly<br>Agree | 2 | 3 | 4 | 5=Strongly<br>Disagree |
|---|---|---|---|---|---|
| I feel more confident since I've started the treatment | | | | | |
| Has your quality of life improved now that you have started using this product? | | | | | |
| I would continue using this treatment beyond 24 weeks as a regular part of my skincare routine. | | | | | |
| What is your overall satisfaction with the regimen? | | | | | |
| I have noticed a positive difference in the appearance of my skin with this regimen. | | | | | |
| I would recommend this product to others. | | | | | |
| My acne is as clear as if I went to a doctor or received a prescription. | | | | | |
| I don't feel the need for a prescription after using this product. | | | | | |
| Do you feel this treatment is designed for you? | | | | | |
| Do you feel more positive and less frustrated about your acne and your skin since starting this treatment? | | | | | |
| Do you feel this treatment meets the needs of your skin? | | | | | |

| Subje | ct Initials | and Da | te |
|-------|-------------|--------|----|

| Subject Initials: | Subject Number: |
|-------------------|-----------------|

#### Sample Diary 1

Please record daily (in BLACK INK) the time you applied the product. DO NOT use pencil or white out, or draw arrows  $\downarrow$  or quotation marks (" "). If you have any problems, please contact Miguel at (972) 852-5880 immediately!

#### **USAGE INSTRUCTIONS:**

- Facial cleanser: Massage a small amount onto wet skin. Rinse
- Dispense a nickel size amount of product and apply as a thin layer to the entire face or any other affected areas of the skin once daily, after washing gently with a mild soap-less cleanser and drying the area.
- Moisturizing Lotion: After applying the product, use moisturizer on the entire face. Apply daily to dry skin as needed or as directed by physician.
- Facial Moisturizer SPF 30: Apply lilberally 15 minutes before sun exposure. Use a water resistant sunscreen if swimming or sweating. Reapply at least every 2 hours.

| Date | Day | Cleanser (✓) | Application Time | Moisturizer (✓) | SPF (✓) | Comments |
|---|---|---|---|---|---|---|
| 5/6/2016<br>Visit 1 | Friday | | | | | |
| 5/7/2016 | Saturday | | | | | |
| 5/8/2016 | Sunday | | | | | |
| 5/9/2016 | Monday | | | | | |
| 5/10/2016 | Tuesday | | | | | |
| 5/11/2016 | Wednesday | | | | | |
| 5/12/2016 | Thursday | | | | | |
| 5/13/2016<br>Visit 2 | Friday | | | | | |
| 5/14/2016 | Saturday | | | | | |
| 5/15/2016 | Sunday | | | | | |
| 5/16/2016 | Monday | | | | | |
| 5/17/2016 | Tuesday | | | | | |
| 5/18/2016 | Wednesday | | | | | |
| 5/19/2016 | Thursday | | | | | |
| 5/20/2016<br>Visit 3 | Friday | | | _ | | |

| Subject Initials: | Subject Number: |
|-------------------|-----------------|
|-------------------|-----------------|

### Sample Diary 2

Please record daily (in BLACK INK) the time you applied the product. DO NOT use pencil or white out, or draw arrows  $\downarrow$  or quotation marks (" "). If you have any problems, please contact Miguel at (972) 852-5880 immediately!

#### **USAGE INSTRUCTIONS:**

- Facial cleanser: Massage a small amount onto wet skin. Rinse
- Clean the skin thoroughly before applying this product. Cover the entire affected area with a thin layer one to three times daily. Because excessive drying of the skin may occur, start with one application daily, then gradually increase to two or three daily if needed or as directed by a doctor. If bothersome dryness or peeling occurs, reduce application to once a day or every other day.
- Moisturizing Lotion: After applying the product, use moisturizer on the entire face. Apply daily to dry skin as needed or as directed by physician.
- Facial Moisturizer SPF 30: Apply lilberally 15 minutes before sun exposure. Use a water resistant sunscreen if swimming or sweating. Reapply at least every 2 hours.

| Date | Day | Cleanser (✓) | Application Time | | | 277.6 | | |
|---|---|---|---|---|---|---|---|---|
| | | | 1 | 2 | 3 | Moisturizer (✓) | SPF (✓) | Comments |
| 5/6/2016<br>Visit 1 | Friday | | | | | | | |
| 5/7/2016 | Saturday | | | | | | | |
| 5/8/2016 | Sunday | | | | | | | |
| 5/9/2016 | Monday | | | | | | | |
| 5/10/2016 | Tuesday | | | | | | | |
| 5/11/2016 | Wednesday | | | | | | | |
| 5/12/2016 | Thursday | | | | | | | |
| 5/13/2016<br>Visit 2 | Friday | | | | | | | |
| 5/14/2016 | Saturday | | | | | | | |
| 5/15/2016 | Sunday | | | | | | | |
| 5/16/2016 | Monday | | | | | | | |
| 5/17/2016 | Tuesday | | | | | | | |
| 5/18/2016 | Wednesday | | | | | | | |
| 5/19/2016 | Thursday | | | | | | | |
| 5/20/2016<br>Visit 3 | Friday | | | | | | | |